
#### The GlaxoSmithKline group of companies

204851

| Division | : | Worldwide Development |
|-------------------------|---|-----------------------------------|
| <b>Information Type</b> | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a multi-centre Phase IIa double-blind, placebo-controlled study to investigate the efficacy and safety of GSK3196165 in subjects with inflammatory hand osteoarthritis.

Compound Number : GSK3196165

Effective Date : 09-FEB-2018

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204851.
- This RAP is intended to describe the planned efficacy, safety, pharmacokinetic (PK), PK/PD and Biomarker analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Interim Analyses and Statistical Analysis Complete (SAC) deliverables.

#### **Author's Name and Functional Area:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Statistician (Immuno-Inflammation, Clinical Statistics) | NA | NA |
| Director Clinical Pharmacology (Immuno-<br>Inflammation, Clinical Pharmacology<br>Modelling and Simulation) | 07-Feb-2018 | eSignature |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Director, Statistics (Immuno-Inflammation, Clinical Statistics) | 09-Feb-2018 | eSignature |
| Manager, Programming (Immuno-<br>Inflammation, Clinical Programming) | 08-Feb-2018 | eSignature |

# **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | | |
| Manager, Programming (Immuno-<br>Inflammation, Clinical Programming) | 08-Feb-2018 | eSignature |
| PPD | | |
| Clinical Development Director (Immuno-<br>Inflammation, Clinical Development) | 08-Feb-2018 | eSignature |
| PPD | | |
| Clinical Development Manager (Immuno-<br>Inflammation, Clinical Pharmacology Sciences<br>and Study Operations) | 08-Feb-2018 | eSignature |
| PPD | | |
| Safety Development Lead (Global Clinical Safety and Pharmacovigilance) | 07-Feb-2018 | Email |
| PPD | | |
| Data Quality Lead (Immuno-inflammation Global Clinical Sciences and Operations) | 07-Feb-2018 | eSignature |

Copyright 2016 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING 8 | ANALYSIS | S PLAN SYNPOSIS | 6 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | Change<br>Study C<br>Study D | s to the Pro<br>bjectives ar<br>esign | TOCOL INFORMATIONotocol Defined Statistical Analysis Plannd Endpoints | |
| 3. | PLANI<br>3.1.<br>3.2. | Interim A | Analyses | | 13 |
| 4. | ANAL`<br>4.1. | | | S | |
| 5. | | ENTION | S | DATA ANALYSES AND DATA HANDLING | |
| 6. | STUD<br>6.1. | | w of Planne | ALYSESed Analysescomitant OA Medication | 18 |
| 7. | PRIM/<br>7.1. | | Analyses<br>Overview | ANALYSESof Planned Primary Efficacy Analyses<br>Primary Efficacy Statistical Analyses | 19<br>19 |
| 8. | SECO<br>8.1. | | Analyses<br>Overview<br>Planned S<br>8.1.2.1. | AL ANALYSES of Planned Secondary Efficacy Analyses Secondary Efficacy Statistical Analyses Continuous Endpoints Binary Endpoints | 21<br>21<br>22 |
| | 8.2. | 8.2.1. | Overview 8.2.1.1. | of Planned Adverse Event Analyses | 25<br>25 |
| | | 8.2.2.<br>8.2.3. | 8.2.2.1. | of Planned Clinical Laboratory Analyses Laboratory Values | 27<br>28<br>29<br>29 |
| | 8.3. | Pharma<br>8.3.1.<br>8.3.2.<br>8.3.3. | cokinetic Ar<br>Overview<br>Drug Con | nalysesof Planned Pharmacokinetic Analysesocentration Measuresnnnnnnnnnnnnnnnnnnnnnnnnnnnnnnnn | 31<br>31<br>31 |


| 9. | OTHE | R EXPLO | RATORY ST | TATISTICAL ANALYSES | 32 |
|---|---|---|---|---|---|
| | 9.1. | Imaging | analyses | | 32 |
| | | 9.1.1. | | f planned Imaging analyses | |
| | | 9.1.2. | Planned Im | aging Statistical Analyses | 32 |
| | 9.2. | Pharmad | okinetic / Ph | narmacodynamic Analyses | 33 |
| | 9.3. | | | | |
| | | 9.3.1. | Pharmacod | lynamic Biomarker Analyses | 34 |
| | | | | Overview of Planned Pharmacodynamic | |
| | | | | Biomarker Analyses | 34 |
| | | 9.3.2. | | narker Analyses | 35 |
| | | | | Overview of Planned Safety Biomarker | |
| | | | | Analyses | |
| | 9.4. | Analyses | | amol Data | |
| | | 9.4.1. | Overview o | f Planned Analyses on Paracetamol Data | 36 |
| 10. | INTER | RIM ANAL | YSES | | 37 |
| | 10.1. | Overviev | v of planned | Week 6 Interim Analysis | 37 |
| | | 10.1.1. | Overview o | f Study Population Analysis at Week 6 Interim | 37 |
| | | 10.1.2. | Overview o | f Safety Analysis at Week 6 Interim | 38 |
| | | 10.1.3. | Overview o | f Planned Efficacy Analysis at Week 6 Interim | 38 |
| | 10.2. | Overviev | v of planned | Pharmacokinetic Interim Analysis | 39 |
| | 10.3. | Overviev | v of Adminis | trative Interim Data Review | 40 |
| 11. | REFE | RENCES. | | | 42 |
| 40 | | NDIOEC | | | 40 |
| 12. | 12.1. | | | Deviation Management and Definitions for Per | 43 |
| | 12.1. | | | Deviation Management and Definitions for Fer | 11 |
| | 12.2. | | • | Events | |
| | 12.2. | 12.2.1. | | efined Time & Events | |
| | | 12.2.1. | | Screening period Time and Events table | |
| | | | | Treatment period Time and Events table | |
| | | | | Follow up visit and early withdrawal* | 40 |
| | | | | procedures list | 47 |
| | 12.3. | | | nent Windows | |
| | | 12.3.1. | Definitions | of Assessment Windows for Analyses | 48 |
| | 12.4. | | | ent States and Phases | |
| | | 12.4.1. | Study Phas | ses | 49 |
| | | 12.4.2. | | States | |
| | | | | Treatment States for AE Data | |
| | 12.5. | | | splay Standards & Handling Conventions | |
| | | 12.5.1. | | tment & Sub-group Display Descriptors | |
| | | 12.5.2. | | efinition & Derivations | |
| | | | | Baseline Definitions | 50 |
| | | | | Derivations and Handling of Missing Baseline Data | 51 |
| | | 12.5.3. | | Process & Standards | |
| | 12.6. | | | and Transformed Data | |
| | 12.0. | 12.6.1. | | and mansionned Data | |
| | | 12.6.1. | | ulation | |
| | | 12.6.3. | | | |
| | | 12.6.4. | • | | |
| | | | oaoy | | 55 |


| | 12.6.5. | Imaging | | 50 |
|---|---|---|---|---|
| | 12.6.6. | | Dhawsa and was win Dismontons | |
| | | | Pharmacodynamic Biomarkers | |
| | | | Safety Biomarkers | |
| 40.7 | ۸ ما ا | | Biomarker Derivations | |
| 12.7. | | | ure Withdrawals & Handling of Missing Data | |
| | 12.7.1. | | Withdrawals | |
| | 12.7.2. | | f Missing Data | |
| | | | Handling of Missing and Partial Dates | ხგ |
| | | | Handling of Missing Data for Statistical | 00 |
| | | | Analysis | |
| 40.0 | Δ !' | | Handling of Endpoint Specific Missing Data | |
| 12.8. | | | of Potential Clinical Importance | |
| | 12.8.1. | • | Values | |
| 400 | | | | |
| 12.9. | | | ter Studies | |
| 12.10. | | | e Comparisons & Multiplicity | |
| | | | f Multiple Comparisons & Multiplicity | 74 |
| 12.11. | | | Checking and Diagnostics for Statistical | |
| | 12.11.1. | | Analysis Assumptions | |
| | | | Continuous Endpoints | |
| | | | Binary Endpoints | |
| 12.12. | Appendix | (12: Definiti | ons of some Parameters of Interest | 76 |
| | | • | Parameters of Interest | |
| 12.13. | | | unistic Infections: MedDRA Preferred Terms | |
| | | | tic Infections: MedDRA Preferred Terms | |
| 12.14. | | | eviations & Trade Marks | |
| | | | ns | |
| | | | S | |
| 12.15. | | | Data Displays | |
| | | | ay Numbering | |
| | | | nple Shell Referencing | |
| | | | Priority] | |
| | | | ılation Tables | |
| | | | bles | |
| | | | gures | |
| | | | les | |
| | | | ıres | |
| | 12.15.9. | Pharmacol | kinetic Tables | 116 |
| | | | kinetic Figures | |
| | 12.15.11 | .Pharmacoo | dynamic and / or Biomarker Tables | 118 |
| | 12.15.12 | .Pharmacoo | dynamic and / or Biomarker Figures | 121 |
| | | | kinetic / Pharmacodynamic Figures | |
| | | | S | |
| | | | istings | |
| 12.16. | Appendix | : 17: Examp | le Mock Shells for Data Displays | 135 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for the final Clinical Study Report (CSR) of study 204851. |
| Protocol | This RAP is based on the protocol amendment 2(Dated:03Jan2017) of study 204851 (GSK Document No. : 2015N242468_02) |
| Primary<br>Objective | To assess the efficacy potential of GSK3196165 on pain in inflammatory Hand Osteoarthritis (HOA). |
| Primary<br>Endpoint | Change from baseline in 24h average hand pain intensity at Week 6, as measured by daily pain Numerical Rating Scale (NRS) averaged over the 7 days prior to assessment visit. |
| Study<br>Design | Randomised Phase IIa, multicentre, double-blind (sponsor unblind), placebo-<br>controlled parallel group study in patients with active inflammatory HOA. |
| | At least 40 subjects will be randomised to either placebo or GSK3196165 in a 1:1 ratio (n=20 per arm). |
| | <ul> <li>4 week screening period will be followed by a 12 week treatment period<br/>(dosing with GSK3196165 or placebo), then a follow up period completing on<br/>week 22.</li> </ul> |
| | <ul> <li>Treatment with GSK3196165 or placebo will be given as a single subcutaneous injection (shielded to subjects) to the abdomen or thigh, by an unblinded administrator weekly for 5 injections, from Week 0 to Week 4 (Days 1, 8, 15, 22, 29), then every other week for 3 further injections, from Week 6 until Week 10 (Days 43, 57 and 71).</li> </ul> |
| Planned | Efficacy (Primary Analysis) |
| Analyses | Safety, PK, PK/PD, Biomarkers, Imaging (Secondary/Exploratory analyses) |
| Analysis<br>Populations | Screened population: all subjects who were screened including those who are classified as screen failures. |
| | Enrolled population: all subjects who passed screening and entered the study. |
| | Intent to Treat (ITT) population: all subjects who were randomised to treatment and who received at least one dose of study treatment. This population will be based on randomised treatment group. |
| | Safety population: all subjects who received at least one dose of study treatment (GSK3196165 or placebo). This population will be based on the treatment actually received. |
| | Pharmacokinetic (PK) population: all subjects in the 'Safety' population who have at least one valid PK assessment. |


| Overview | Key Elements of the RAP |
|---|---|
| Hypothesis | H <sub>0</sub> : there is no difference between GSK3196165 and placebo in the change from baseline in the average Pain NRS Scale at Week 6. |
| | H <sub>A</sub> : there is a difference between GSK3196165 and placebo in the change from baseline in the average Pain NRS Scale at Week 6. |
| Primary<br>Analyses | The primary endpoint will be analysed using a repeated measures model (MMRM). |
| Secondary<br>Analyses | Continuous endpoints will be analysed using the same methods as the primary endpoint. For some endpoints this may be after transformation, if applicable. |
| | Binary endpoints will be summarised using counts and proportions and analysed using a Generalised Estimating Equations (GEE) model. |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Any changes from the originally planned statistical analysis specified in the protocol (GSK Document No. 2015N242468 02, Dated:03JAN2017) are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan Rationale for Char | |
| Endpoint is defined as 'Change from Baseline in patient global assessment (PtGA) and physician global assessment (PhGA) of disease activity at Week 6, 12 and 22'. | Endpoint is defined as<br>'Change from Baseline in<br>patient global assessment<br>(PtGA) and physician global<br>assessment (PhGA) of<br>disease activity at Weeks 2,<br>4, 8 12 and 22'. | PtGA and PhGA timepoints were incorrectly specified in the endpoints list on pages 11 and 16 of protocol, but correct in the time and events table and elsewhere |
| Endpoint is defined as 'Change from baseline in structural and inflammatory HOA features in the affected hand (including synovitis, bone erosions, joint space width, and bone marrow edema) as assesses by the RAMRIQ scoring system. | Endpoint is defined as 'Change from baseline in structural and inflammatory HOA features in the affected hand (including synovitis, bone erosions, joint space width, and bone marrow edema) as assesses by the HOAMRIQ scoring system. | Incorrect scoring<br>system is specified in<br>the protocol. |
| Administrative Interim Review not specified | Addition of Administrative<br>Interim Review | Administrative Interim Review was requested by II TA Head. This was requested after the protocol amendment was created and therefore is being documented in the RAP. The administrative interim review was approved by the MDL on 18May2017. The timing of this interim was after unblinding of the study at the protocol defined PK interim. |

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Protocol specifies 'The primary endpoint will be analysed using a repeated measures model (MMRM) adjusted for baseline pain score, treatment group, visit and the visit by treatment group interaction as fixed effects, patient as a random effect and day within patient as a repeated effect, using an unstructured covariance matrix.' | The MMRM model will also be investigated with the addition of the baseline*visit interaction term and the most appropriate model selected. | Error from protocol specified analyses |

# 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the efficacy potential of<br>GSK3196165 on pain in<br>inflammatory HOA. | <ul> <li>Change from baseline in 24h average hand pain<br/>intensity at week 6, as measured by daily pain<br/>Numerical Rating Scale (NRS) averaged over the<br/>7 days prior to assessment visit.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate impact of<br>GSK3196165 on average and<br>worst HOA pain, over time. | <ul> <li>Change from baseline in 24h average hand pain intensity at each visit, measured by daily pain NRS and averaged over the 7 days prior to each assessment visit.</li> <li>Change from baseline of worst hand pain intensity</li> </ul> |
| | over 24h at each visit, measured by daily NRS and averaged over the 7 days prior to each assessment visit. |
| | <ul> <li>Proportion of subjects in each treatment group<br/>achieving a 30% reduction in 24h average hand<br/>pain intensity at each visit, measured by daily NRS<br/>averaged over the 7 days prior to assessment visit.</li> </ul> |
| | <ul> <li>Proportion of subjects in each treatment group<br/>achieving a 50% reduction in 24h average hand<br/>pain intensity at each visit, measured by daily NRS<br/>averaged over the 7 days prior to assessment visit.</li> </ul> |
| | Proportion of subjects in each treatment group<br>achieving a 30% reduction in 24h worst hand pain<br>intensity at each visit, measured by daily NRS<br>averaged over the 7 days prior to assessment visit. |

| Objectives | Endpoints |
|---|---|
| | Proportion of subjects in each treatment group achieving a 50% reduction in 24h worst hand pain intensity at each visit, measured by daily NRS averaged over the 7 days prior to assessment visit. |
| <ul> <li>To assess the impact of<br/>GSK3196165 on hand pain (on<br/>use), stiffness and function, over<br/>time.</li> </ul> | <ul> <li>Change from baseline in Australian Canadian<br/>Hand Osteoarthritis Index (AUSCAN) 3.1 NRS,<br/>total and domains (pain, morning stiffness,<br/>function) scores at each visit.</li> </ul> |
| To assess the impact of<br>GSK3196165 on HOA<br>inflammation. | Change in number of swollen and tender hand joints at each visit. |
| To assess potential impact of<br>GSK3196165 on disease activity<br>in HOA. | <ul> <li>Change from baseline in patient global<br/>assessment (PtGA) and physician global<br/>assessment (PhGA) of disease activity at Weeks<br/>2, 4, 8 12 and 22.</li> </ul> |
| To assess safety of GSK3196165 in HOA patients, over the study duration. | <ul> <li>Incidence of adverse events and serious adverse events.</li> <li>Incidence of infections.</li> <li>Incidence of pulmonary events (cough/dyspnea, PAP and D<sub>LCO</sub>).</li> <li>Immunogenicty.</li> </ul> |
| To assess population pharmacokinetics of GSK3196165 in HOA. | Population pharmacokinetics endpoints such as CL/F, Vss/F, Ka. |
| Exploratory Objectives | Exploratory Endpoints |
| To explore the potential impact of<br>GSK3196165 on disease<br>progression/modification in HOA,<br>using MRI imaging. | <ul> <li>Change from baseline in synovitis in the affected hand*, as measured by DCE-MRI including the exchange rate (K<sup>trans</sup>), interstitial volume (v<sub>e</sub>), plasma volume (v<sub>p</sub>), volume of synovitis, initial rate of enhancement (IRE), and maximum signal intensity enhancement (ME).</li> <li>Change from baseline in structural and</li> </ul> |
| | inflammatory HOA features in the affected hand* (including synovitis, erosive damage, cysts, osteophytes, cartilage space loss, malalignment, and bone marrow lesions) as assessed by the OMERACT HOAMRIS scoring system |
| | <ul> <li>Change from baseline in structural and inflammatory HOA features in the affected hand* (including synovitis, bone erosions, joint space width, and bone marrow edema) as assesses by the HOAMRIQ scoring system.</li> <li>Change from baseline in bone shape as assessed by structural MRI of the affected hand*.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| The exploration of the relationship<br>between GSK3196165 PK and PD<br>effects and/or efficacy. | <ul> <li>Relationship between concentration or PK<br/>parameters and PD endpoint(s).</li> </ul> |
| To evaluate the potential of<br>GSK3196165 to affect biomarkers<br>of HOA. | Change in blood biomarkers from baseline at each visit. |

<sup>\*</sup> If only one hand is affected by HOA and meets the inclusion criteria, the affected hand will be documented at screening and used for all assessments. In cases where both hands are affected by HOA and both meet the inclusion criteria, then the dominant hand will be documented at screening and this hand will be used for the MRI assessments throughout the study.

## 2.3. Study Design



## 2.4. Statistical Hypotheses

The primary endpoint of the study is to evaluate the change from baseline in the average Pain NRS following 6 weeks of treatment with GSK3196165 or placebo in adult subjects with HOA.

The study will test the null hypothesis that there is no difference between GSK3196165 and placebo in the change from baseline in the 24h average Pain NRS Scale at Week 6. The alternative hypothesis is that there is a difference between GSK3196165 and placebo in the change from baseline in the 24h Pain NRS Scale at Week 6 using a two-sided test  $(\alpha=0.05)$ .

#### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

An interim analysis will be performed during the study to review the available PK data and target engagement biomarkers. The timing of this analysis will coincide with other internal decision making across the GSK3196165 project.

Another formal interim analysis may be conducted on the key safety, primary efficacy and key secondary endpoints in this study. The purpose of this interim will be to help with decision-making regarding the subsequent clinical development of GSK3196165 for OA. The timing of this analysis will be once a minimum of 30 subjects have completed day 43 (Week 6). It is likely that by the time 30 subjects have completed week 6 the study would have fully recruited and the interim would not lead to early stopping of this study for efficacy.

In addition to the formal planned interim analyses, further data reviews may be carried out by senior managers not involved in the study conduct to aid in portfolio and budget decisions. These administrative reviews will have no impact on the ongoing study.

Full details can be found in Section 10.

# 3.2. Final Analyses

The final planned end of study analyses on all endpoints will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprise of all subjects who were screened including those subjects who were classified as Screen Failures | Study Population |
| Enrolled | <ul> <li>All participants who passed screening and entered the study. Included are: Run-in Failures; Randomized Participants; in non-randomized study and participants who were assigned a treatment in a non-randomised study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| Intent-To-Treat | Comprise of all randomised subjects who | Study Population |
| (ITT) | receive at least one dose of study treatment (GSK3196165 or placebo). | Efficacy |
| | This population will be based on the treatment to which the subject was randomised. | |
| | Any subject who receives a treatment randomisation number will be considered to have been randomised. | |
| Safety | Comprise of all subjects who receive at least | Safety |
| | one dose of study treatment (GSK3196165 or placebo). | PD/Biomarker |
| | This population will be based on the treatment the subject actually received. | |
| | If a subject consistently received the same wrong treatment arm, then this will be considered as the actual treatment arm. The handling of subjects receiving a wrong treatment only for some applications will be decided on a case by case basis. | |
| Pharmacokinetic | Subjects in the 'Safety' population for whom a | • PK |
| (PK) | pharmacokinetic sample was obtained and analysed. | PK/PD |

#### NOTES:

• Please refer to Appendix 15: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

Please refer to the Protocol Deviation Management Plan (PDMP): Dated: 30Nov2017 (Version 3) for full details.

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---|---|
| 12.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 12.2 | Appendix 2: Time & Events |
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Treatment States and Phases |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |
| 12.9 | Appendix 9: Multicentre Studies |
| 12.10 | Appendix 10: Multiple Comparisons & Multiplicity |
| 12.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses. |
| 12.12 | Appendix 12: Definition of some Parameters of Interest |
| 12.13 | Appendix 13: Opportunistic Infections: MedDRA Preferred Terms |
| 12.14 | Appendix 14: Abbreviations & Trade Marks |
| 12.1512<br>.15 | Appendix 15: List of Data Displays |
| 12.16 | Appendix 16: Example Mock Shells for Data Displays |

#### 5.1. General Considerations

- This is a multi-centre study and there are no planned adjustments for multiple centres or regions.
- There are no planned adjustments for multiple comparisons or multiplicity.

#### Unless otherwise stated, the following rules will apply:

- Summaries and displays will present data by treatment group.
- Listings will be sorted by treatment group.
- The following statistics will be used to summarise the data, unless otherwise specified:

- Continuous Variables: number of observations (n), mean, standard deviation (SD), median, minimum and maximum.
- Categorical Variables: number of observations (n), frequency counts and percentages.
- Summaries by Visit: Only scheduled visits will be presented, unless otherwise stated. Scheduled visits will be slotted as shown in section 12.3.1.
- Unscheduled visits will be listed but will not contribute towards any summary statistics/analyses, unless otherwise stated.
- For continuous endpoints, no imputation for missing values across visits will be done, individual missing item scores contributing to PRO domain scores may be imputed as per the rules given within each PRO (see section 12.7.2.3 for full details)..
- For binary endpoints, subjects with missing values will be considered as non-responders.

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The Study Population analyses will be based on the Screened, Enrolled or Intent-to-Treat (ITT) population, as appropriate unless otherwise specified.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 17: List of Data Displays.

Table 3 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Randomisation | | |
| Randomised and Actual Treatments | | Y |
| Subject Disposition | | |
| Subject Disposition | Υ | |
| Screening Status and Reasons for Screening Failures | Υ | Υ |
| Subjects by Country and Site ID | Υ | |
| Reasons for Subject Withdrawals | | Υ |
| Subjects for Whom the Treatment Blind was Broken | | Υ |
| Protocol Deviations | | |
| Important protocol deviations | Υ | Υ |
| Subjects with Inclusion/Exclusion Criteria Deviations | | <b>Y</b> [1] |
| Populations Analysed | | |
| Study Populations | Υ | |
| Subjects Excluded from Any Population | | Υ |
| <b>Demographic and Baseline Characteristics</b> | | |
| Demographics Characteristics | Υ | Υ |
| Baseline Efficacy Parameters | Υ | |
| Race and Racial Combinations | Υ | <b>Y</b> [2] |
| OA Disease History | Υ | Υ |
| Medical Condition & Concomitant Medications | | |
| Current Medical Conditions | Υ | Υ |
| Concomitant medication | Υ | Υ |
| Concomitant OA medication | Υ | |
| Prior Medication | Υ | Υ |
| Prior OA medication | Υ | |
| Exposure &Treatment Compliance | | |
| Exposure to Study Treatment | Υ | Y |
| NOTES · | | |

#### NOTES:

- Y = Yes display generated.
- [1] Listing also includes analysis population exclusions.
- [2] Listing of race.

#### 6.1.1. Prior/Concomitant OA Medication

OA medications will be identified by the Medical Monitor through review of unique terms and indications prior to unblinding.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Efficacy Analyses

## 7.1.1. Overview of Planned Primary Efficacy Analyses

The Primary Endpoint is defined as the change from baseline in 24h average hand pain intensity at week 6, as measured by the daily pain Numerical Rating Scale (NRS) averaged over the 7 days prior to assessment visit.

The primary efficacy analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

Table 4 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Section 12.15: List of Data Displays.

Table 4 Overview of Planned Primary Efficacy Analyses

| Endpoint | Absolute | | | | | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Stats Analysis S | | Summary Individual | | Stats Analysis | | | Summary | | Individual | | | |
| | Т | F | Г | ٦ | F | F | L | Т | F | L | Т | F | F | L |
| Pain | Pain | | | | | | | | | | | | | |
| 24h <b>average</b> hand<br>pain NRS score<br>averaged over 7 days<br>prior to assessment | Υ[2] | | Y<br>[1,2] | <b>Y</b> [2] | <b>Y</b> [2] | Y | Y | Y | Y | Y<br>[1] | Y | Y | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Raw SAS log output from analysis
- [2] Absolute values will be displayed in the same outputs as the change from baseline.

## 7.1.2. Planned Primary Efficacy Statistical Analyses

#### **Primary Statistical Analyses**

#### Endpoint(s)

• Change from baseline in 24h average hand pain intensity at week 6, as measured by daily pain Numerical Rating Scale (NRS) averaged over the 7 days prior to assessment visit.

#### **Model Specification**

- Endpoints will be statistically analysed using a mixed model repeated measures (MMRM) model.
- The model will be fitted using an unstructured covariance matrix.
- Terms fitted in the MMRM model will include:

Fixed Categorical : Treatment group, Visit, Treatment group \* Visit Interaction

Fixed Continuous Covariates : Baseline pain score #

Random Covariates : Subject Repeated : Visit

# A model will also be explored fitting Baseline\*Visit & the most appropriate model selected.

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Point estimates and corresponding 95% confidence intervals will be constructed for the treatment differences (GSK3196165-Placebo) at each visit, using the least squared (LS) means obtained from the repeated measures mixed-effects model.
- Plots of LS means and 95% confidence intervals from the model will be generated for each treatment group by time.

#### **Sensitivity and Supportive Statistical Analyses**

- Following review of the data, additional analyses maybe conducted to further support the primary statistical analyses, if deemed appropriate.
- Non-parametric analyses may be conducted if the normality assumption does not hold.
- Analyses using different covariance structures may be explored if the unstructured covariance matrix does not converge. The first covariance structures to be tested will be compound symmetry (CS) and then first order autoregressive (AR(1)).
- Sensitivity analyses maybe conducted to assess the impact of missing data.
- Further sensitivity analyses may be conducted to assess the impact of rescue medication use:
- E.g. The impact of imputing all 24h average pain scores to be the 24h worst pain score on days in which paracetamol was used (any dose) may be assessed.
- Further sensitivity analyses may be conducted excluding any subjects taking prohibited medications throughout the study.

•

## 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Efficacy Analyses

## 8.1.1. Overview of Planned Secondary Efficacy Analyses

The secondary efficacy analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

Table 5 provides an overview of the planned efficacy analyses, with further details of data displays being presented in Appendix 17: List of Data Displays.

Table 5 Overview of Planned Efficacy Analyses

| Endpoint | Abs | olute | | | | | | Chan | ge fror | n Base | eline | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | | nmary | | vidual | | Analy | sis | | mary | | idual |
| | Т | F | L | Τ | F | F | L | Τ | F | L | Т | F | F | L |
| 24h average hand pai | | Ssco | | 1 | 1 | | | 1 | 1 | 1 | 1 | 1 | 1 | |
| Proportion of<br>subjects achieving a<br>30% reduction in 24h<br>average hand pain<br>NRS score averaged<br>over 7 days prior to<br>assessment | Y<br>[2] | | Y<br>[1] | Y<br>[2] | Υ | | Y | | | | | | | |
| Proportion of<br>subjects achieving a<br>50% reduction in 24h<br>average hand pain<br>NRS score averaged<br>over 7 days prior to<br>assessment | Y<br>[2] | | Y<br>[1] | Y<br>[2] | Υ | | Y | | | | | | | |
| Daily 24h average hand pain NRS | | | | | | | Υ | | | | | | | |
| 24h worst hand pain l | | score | | | 1 | | 1 | | | • | 1 | 1 | 1 | |
| 24h worst pain NRS<br>score averaged over<br>7 days prior to<br>assessment | <b>Y</b> [<br>3] | | <b>Y</b><br>[1,3] | Y<br>[3] | Y<br>[3] | Y | Y | Y | Y | <b>Y</b> [1] | Y | Y | | Υ |
| Daily 24h worst hand pain NRS | | | | | | | Υ | | | | | | | |
| Proportion of<br>subjects achieving a<br>30% reduction in 24h<br>worst pain NRS<br>score averaged over<br>7 days prior to<br>assessment | Y<br>[2] | | Y<br>[1] | Y<br>[2] | Υ | | Y | | | | | | | |
| Proportion of<br>subjects achieving a<br>50% reduction in 24h<br>worst pain NRS | Y<br>[2] | | Y<br>[1] | Y<br>[2] | Υ | | Y | | | | | | | |

| Endpoint | Abs | Absolute | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis S | | Sun | Summary Individual | | Stats Analysis | | | Summary | | Individual | | |
| | Τ | F | Ĺ | Τ | F | F | L | T | F | L | Τ | F | F | L |
| score averaged over | | | | | | | | | | | | | | |
| 7 days prior to | | | | | | | | | | | | | | |
| assessment | | | | | | | | | | | | | | |
| AUSCAN | | | | | | | | | | | | | | |
| AUSCAN 3.1 NRS | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | | Υ |
| Components | [3] | | [1,3] | [3] | [3] | | | | | [1] | | | | |
| Joint Assessments | l | ı | l | | | | | ı | | | | | | |
| Swollen hand joints | Υ | | <b>Y</b> [1,3] | Υ | Υ | | Υ | Υ | Υ | <b>Y</b> [1] | Υ | Υ | | Υ |
| | [3] | | | [3] | [3] | | | | | | | | | |
| Tender hand joints | Y[ | | <b>Y</b> [1,3] | Υ | Υ | | Υ | Υ | Υ | <b>Y</b> [1] | Υ | Υ | | Υ |
| | 3] | | | [3] | [3] | | | | | | | | | |
| Pain/Tenderness | | | | | | | Υ | | | | | | | |
| Hand Joint | | | | | | | | | | | | | | |
| Assessment | | | | | | | | | | | | | | |
| Disease Global Asses | sme | nt | | | | | | | | | | | | |
| PhGA | Υ | | <b>Y</b> [1,3] | Υ | Υ | | Υ | Υ | Υ | Y[1] | Υ | Υ | | Υ |
| | [3] | | | [3] | [3] | | | | | | | | | |
| PtGA | Y[ | | <b>Y</b> [1,3] | Υ | Υ | | Υ | Υ | Υ | <b>Y</b> [1] | Υ | Υ | | Υ |
| | 3] | | | [3] | [3] | | | | | | | | | |

#### NOTES:

T = Table, F = Figure, L = Listing, Y = Yes display generated.

Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.

Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.

Individual = Represents FL related to any displays of individual subject observed raw data.

- [1] Raw SAS log output from analysis.
- [2] Summaries and analysis will be presented together in one output.
- [3] Absolute values will be displayed in the same outputs as the change from baseline.

#### 8.1.2. Planned Secondary Efficacy Statistical Analyses

#### 8.1.2.1. Continuous Endpoints

# **Secondary Statistical Analyses**

#### Endpoint(s)

- Change from baseline in 24h average hand pain intensity at each visit, measured by daily pain NRS and averaged over the 7 days prior to each assessment visit.
- Change from baseline of **worst** hand pain intensity over 24h at each visit, measured by daily NRS and averaged over the 7 days prior to each assessment visit.
- Change from baseline in Australian Canadian Hand Osteoarthritis Index (AUSCAN) 3.1 NRS, total and domains (pain, morning stiffness, function) scores at each visit.
- Change from baseline in number of swollen and tender hand joints at each visit.
- Change from baseline in patient global assessment (PtGA) and physician global assessment (PhGA) of disease activity at Weeks 2, 4, 8, 12 and 22.

#### **Model Specification**

#### **Secondary Statistical Analyses**

• Continuous endpoints will be statistically analysed using the same methods as the primary endpoint (MMRM). See Section 7.1.2 for full details.

## **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Continuous endpoints will be presented using the same methods as the primary endpoint.

#### **Sensitivity and Supportive Statistical Analyses**

- Non-parametric analyses may be conducted if the normality assumption does not hold.
- Analyses using different covariance structures may be explored if the unstructured covariance matrix does not converge. The first covariance structures to be tested will be compound symmetry and then first order autoregressive (AR(1)).
- Further sensitivity analyses may be conducted to assess the impact of missing data.
- Further sensitivity analyses may be conducted to assess the impact of rescue medication use:
  - E.g. The impact of imputing all 24h average pain scores to be the 24h worst pain score on days in which paracetamol was used (any dose) may be assessed.
- Further sensitivity analyses may be conducted excluding any subjects taking prohibited medications throughout the study.

## 8.1.2.2. Binary Endpoints

#### Secondary Statistical Analyses

#### Endpoint(s)

- Proportion of subjects in each treatment group achieving a 30% reduction in 24h average hand pain intensity at each visit, measured by daily NRS averaged over the 7 days prior to assessment visit.
- Proportion of subjects in each treatment group achieving a 50% reduction in 24h average hand pain intensity at each visit, measured by daily NRS averaged over the 7 days prior to assessment visit.
- Proportion of subjects in each treatment group achieving a 30% reduction in 24h worst hand pain intensity at each visit, measured by daily NRS averaged over the 7 days prior to assessment visit.
- Proportion of subjects in each treatment group achieving a 50% reduction in 24h worst hand pain intensity at each visit, measured by daily NRS averaged over the 7 days prior to assessment visit.

#### **Model Specification**

Binary efficacy endpoints will be statistically analysed using a Generalised Estimating
Equations (GEE) model, which will be used to test the treatment comparison of GSK3196165
versus placebo, accounting for the within-subject correlation of outcomes across the multiple
visits.

#### **Secondary Statistical Analyses**

• The model will be fitted using an unstructured covariance structure of the correlated responses.

Terms fitted in the GEE model will include:

Fixed Categorical : Treatment group, Visit, Treatment group \* Visit Interaction,

Respective Baseline NRS score

Repeated : Visit

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- The Binary endpoints will be summarised using counts and proportions of subjects achieving a response by treatment group.
- Differences in the proportions of subjects achieving response between active and placebo will be summarised at each visit. 95% CI for the differences will be constructed using their asymptotic standard errors (asymptotic Wald confidence limits) without continuity correction.
- Point estimates and corresponding 95% confidence intervals will be constructed using contrasts for the treatment by day interactions.
- Plots of the point estimates and 95% confidence intervals from the model will be generated for each treatment group by time.

#### **Sensitivity and Supportive Statistical Analyses**

- Analyses using different covariance structures may be explored if considered appropriate.
- Further sensitivity analyses may be conducted excluding any subjects taking prohibited medications throughout the study.

## 8.2. Safety Analyses

#### 8.2.1. Overview of Planned Adverse Event Analyses

The Adverse Event analyses will be based on the "Safety" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 16: List of Data Displays.

Table 6 Overview of Planned Safety Analyses

| Endpoint | Absolute | | | |
|---|---|---|---|---|
| | Sum | nmary | Individual | |
| | T | F | F | L |
| Adverse Events (AEs) | | | | |
| AE's (Overview) | Υ | | | |
| All AE's | Υ | | | Υ |
| Common (>=5%) AE's | Υ | Υ[1] | | |
| All Drug-Related AE's | Υ | | | |
| Subjects & No. Of Occurrences of Common (>=5%) | Υ | | | |
| Non-Serious AE's | | | | |
| Subject Numbers for Individual AE's | | | | Υ |
| Relationship between AE SOC, PT and Verbatim | | | | Υ |
| Text | | | | ī |
| Serious and Other Significant AE's | | | | |
| Serious AE's | Υ | | | |
| Fatal Serious AE's | | | | Υ |
| Non-Fatal Serious AE's | | | | Υ |
| Reasons for Considering as a Serious AE | | | | Υ |
| AE's leading to permanent discontinuation of study | Υ | | | Υ |
| treatment/ withdrawal | ī | | | |
| AESI's | Υ | | | Υ |
| AESI's – Injection site reactions | Υ | | | |
| AESI's – Systemic Hypersensitivity Reactions | Υ | | | |

#### NOTES:

- T=Table, F=Figure, L=Listing, Y=Yes display generated.
- Summary= Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual= Represents FL related to any displays of individual subject observed raw data.
  [1] Plot of common AEs and Relative Risk will be generated.

#### 8.2.1.1. Adverse Events

- Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) in the latest available version.
- Adverse events of special interest (AESI) will be derived using Common Terminology Criteria for Adverse Events, 2009 v4.0 (CTCAE) and will include:

| AESI | Programmatical Derivation |
|---|---|
| Serious infections, including serious respiratory infections. | SAEs, Filter on infections SOC. Also include HLT Respiratory Infections which will be derived from the Respiratory SOC. |
| Opportunistic infections including TB reactivation | Opportunistic infections will be adjudicated by the SRT, using the preferred terms list given in Section 12.13. Final adjudication conducted by SRT. |
| Neutropenia | Based on Grade 3 or 4 absolute neutrophil count |
| PAP (Pulmonary alveolar proteinosis) | Derived using PAP PT. |
| Hypersensitivity reactions, including anaphylaxis | Hypersensitivity reactions will be adjudicated by the SRT, using AE data and data from hypersensitivity reactions eCRF page. Final adjudication conducted by SRT. |
| Injection site reactions | Derived from PT. |

- AEs with missing intensity will be considered severe.
- Common AEs will be defined as those reported by  $\geq 5\%$  of the subjects in either treatment group, with the threshold applied before any rounding.
- AEs with partial or missing start and/or stop dates will be assumed to be treatmentemergent unless there is evidence through comparison of partial dates to suggest otherwise.
- AEs will be summarised and sorted by system organ class (SOC) and preferred term (PT), unless otherwise specified. Tables will be sorted by overall decreasing frequency of the SOC and then decreasing frequency of PT within the AE.
- Summaries will provide the number and percentage of subjects reporting at least one AE and the total number of events reported.

#### 8.2.2. Overview of Planned Clinical Laboratory Analyses

The Clinical Laboratory analyses will be based on the "Safety" population, unless otherwise specified.

Table 7 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 16: List of Data Displays.

Table 7 Overview of Planned Clinical Laboratory Analyses

| Endpoint / Parameter/ Display Type | | Absol | ute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sun | nmary | Individual | Sur | nmary | Individual |
| | T | F | L | Т | F | L |
| Labs | | | | | | |
| Clinical Chemistry | | | | Υ | | |
| Haematology | | | | Υ | | |
| Urinalysis | | | | Υ | | |
| Proportion of Subjects with Urinalysis findings | | | | Υ | | |
| Lab Parameters of Interest by CTCAE Grade | | | | Υ | Υ | |
| Shift of Lab Parameters of Interest from Baseline to Worst CTCAE Grade | Υ | | | | | |
| All Lab Data for Subjects with any value of PCI | | | Υ | | | |
| Lab Values of PCI | | | Υ | | | |
| Lab Data with Character Results | | | Υ | | | |
| Urinalysis Data for Subjects with any value if PCI | | | Y | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.2.2.1. Laboratory Values

• Refer to Appendix 6 for handling of laboratory values that are above or below the lower limit of quantification.

## 8.2.3. Overview of Planned Other Safety Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 8 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 17: List of Data Displays.

Table 8 Overview of Planned Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | | Change from BL | | |
|---|---|---|---|---|---|---|---|
| | Sum | mary | Indiv | ridual | Sumr | nary | Individual |
| | Т | F | L | F | T | F | L |
| ECG | | | | | | | |
| ECG Findings | Υ | | | | | | |
| ECG Values | | | | | Υ | Υ | |
| Maximum QTc Values Post-Baseline | Υ | | | | | | |
| All ECG Values for Subjects with a Value of PCI | | | Υ | | | | |
| ECG Values of PCI | | | Υ | | | | |
| Abnormal ECG Findings | | | Υ | | | | |
| Subjects meeting QTc discontinuation criteria | | | Υ | | | | |
| Vital Signs | | | | | ı | | |
| Vital Signs | | | Υ | | Υ | | |
| Vital Signs of PCI | | | Υ | | | | |
| All Vital Signs for Subjects with Values of PCI | | | Υ | | | | |
| Immunogenicity | | • | • | | • | | |
| Immunogenicity Results | Υ | | Υ | | | | |
| Pulmonary Assessments | | | | | | | |
| Subjects with Pulmonary Findings | Υ | | | | | | |
| Persistent Cough, Dyspnea and D <sub>LCO</sub> Decrease | Υ | | | | | | |
| Pulse Oximetry | Y | | Υ | | Υ | | |
| D <sub>LCO</sub> | | | Υ | Υ | Υ | | |
| Proportion of Subjects with 15% Relative Decrease in | Υ | | | | | | |
| D <sub>LCO</sub> | | | | | | | |
| Spirometry (FEV1 and FVC) | | | Υ | | Υ | | |
| Cough | Y | | Υ | | | | |
| Borg CR10 | Y | | Υ | | Υ | | |
| Lung Auscultation | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.2.3.1. ECGs

• Triplicate 12-lead ECGs will be collected at the various time points throughout the study shown in Appendix 2. All ECG parameters will be calculated by taking the mean of the non-missing values obtained in the up to three 12-lead ECG evaluations at each visit.

#### 8.2.3.2. Vital Signs

- The following vital signs will be assessed at the various time points in the study shown in Appendix 2:
  - o Temperature (in °C)
  - Systolic and diastolic blood pressure (mmHg)
  - Heart rate (beats/min)
  - o Height (cm)
  - Weight(kg)
  - o Calculated BMI (kg/m²)
  - o Blood oxygen (%).

#### 8.2.3.3. Immunogenicity

- Serum samples for anti-drug antibody (ADA) measurements will be obtained from all randomized subjects after administration of study drug at the scheduled visits.
- Samples taken after dosing with GSK3196165 that have a value at or above the cutpoint will be considered potentially treatment-emergent ADA-positive. A Shift table from baseline to every assessment will be produced for the Immunogenicity population to assess the number of subjects going from:
  - 1) negative  $\rightarrow$  negative,
  - 2) negative  $\rightarrow$  positive,
  - 3) positive  $\rightarrow$  negative, and
  - 4) positive  $\rightarrow$  positive.
- Serum analysis will be performed under the management of Immunogenicity and Clinical Immunology (ICI), GlaxoSmithKline. Serum will be tested for the presence of anti- GSK3196165 antibodies using the currently approved analytical methodology incorporating screening, confirmation and titration steps.
  - Anti-GSK3196165 Binding AB Detection (positive/negative) will be listed together with titre value (mL)

#### 8.2.3.4. Pulmonary Assessments

- The following pulmonary assessments will be performed at the various time points in the study shown in Appendix 2:
  - o Cough (as defined by CTCAE)
  - o Borg CR10
  - Lung Auscultation
  - o Pulse Oximetry
  - o Pulmonary Function Tests (PFTs spirometry, gas transfer [D<sub>LCO</sub>])

Pulmonary findings are defined as follows:

o At least one 15% relative decrease from baseline in D<sub>LCO</sub>.

- $\circ$  At least one 15% relative decrease from baseline in D<sub>LCO</sub> to <70%.
- o Cough of any grade.
- o Any abnormal lung auscultation.

Respiratory Events are defined as follows:

| Event | Definition |
|---|---|
| Persistent cough | Cough CTCAE grade 2 or greater recorded for 3 consecutive weeks (15 or more days). |
| | Identified through Cough 'Yes' entered in the eCRF with Grade determined from AE reporting with the following definition: AESEV=Mild = Grade 1 AESEV=Moderate= Grade 2 AESEV=Severe= Grade 3 |
| Persistent dyspnea | Borg Scale grade 3 or greater recorded for 3 consecutive weeks (15 or more days) on the eCRF page. |
| Persistent decrease of D <sub>LCO</sub> by >15% | Relative decrease of D <sub>LCO</sub> of >15% compared to Baseline for 3 consecutive weeks (15 or more days) |

These definitions are provided for guidance to identify potential cases. Final adjudication will be conducted by the SRT.

#### 8.2.3.5. Cardiovascular Events

In the occurrence of a Cardiovascular Event, patient profiles will be produced using IDSL standard templates.

## 8.3. Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified. There are no planned statistical analyses.

GSK3196165 serum concentration data will be analysed using population approach as described in section 8.3.3.

#### 8.3.1. Overview of Planned Pharmacokinetic Analyses

#### 8.3.2. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Process & Standards) for details on how the concentration data will be derived.

#### 8.3.3. Population Pharmacokinetic (PopPK) Analyses

The primary goal of this analysis is to characterise the PK of GSK3196165 administered subcutaneously in subjects with HOA and compare it with other populations.

- The influence of subject demographics, baseline characteristics, and immunogenicity on the pharmacokinetics of GSK3196165 in this population will be investigated.
- The individual subject PK parameters will be estimated and documented for the purposes of any subsequent model based exposure-response (PK/PD) analyses.

PK analysis will be performed based on population PK approach. GSK3196165 serum concentration-time data will be subjected to nonlinear mixed effects modelling using the program NONMEM. To support this analysis a NONMEM file will be generated, which will be combined with already existing NONMEM file from pooled population PK analysis (Population Pharmacokinetic Analysis of GSK3196165 Following Intravenous and Subcutaneous Administration to Healthy Volunteers, Subjects with Rheumatoid Arthritis and Multiple Sclerosis (Date: 08-Jan-2016)). PK model from previous pooled analysis will be starting point this analysis. If the current PK model described the PK data from HOA subjects well (as per criteria set in TP-EP.BS-WW-001-01) no further base model development will be done. Effect of following covariates will be tested:

- Population type (HOA, healthy volunteers, rheumatoid arthritis and multiple sclerosis)
- Subject demographics (age, sex, and race)
- Baseline characteristics (body weight, free GM-CSF levels)
- Immunogenicity

Results of population PK analysis and PK/PD described in section 9.2 will be reported in detail in a standalone report which will go as an appendix/attachment to the CSR.

## 9. OTHER EXPLORATORY STATISTICAL ANALYSES

## 9.1. Imaging analyses

## 9.1.1. Overview of planned Imaging analyses

The Imaging analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

Table 10 provides an overview of the planned Imaging analyses, with further details of data displays being presented in Section 12.15: List of Data Displays.

Table 9 Overview of Planned Imaging Analyses

| Endpoint | Absolute | | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Stats Analysis 3 | | | mma | Indiv | /idual | Stats Analysis | | | Summary | | Individual | |
| | | | | | ry | | | | | | | | | |
| | Τ | F | L | Т | F | F | L | Т | F | L | Τ | F | F | L |
| Inflammatory Structural Joint Damage | | | | | | | | | | | | | | |
| HOAMRIS Individual | <b>Y</b> [2] | | Υ | Υ | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| Components | | | [1,2] | [2] | [2] | | | | | [1] | | | | |
| HOAMRIQ Individual | <b>Y</b> [2] | | Υ | Υ | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| Components | | | [1,2] | [2] | [2] | | | | | [1] | | | | |
| Joint Inflammation | | | | | | | | | | | | | | |
| DCE-MRI quantitative | <b>Y</b> [2] | | Υ | Υ | Υ | | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| parameters | | | [1,2] | [2] | [2] | | | | | [1] | | | | |
| Bone Shape Parameters | | | | | | | | | | | | | | |
| Bone Shape Parameters | | | | Υ | Υ | | Υ | | | | Υ | Υ | | Υ |
| | | | | [2] | [2] | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Raw SAS log output from analysis.
- [2] Absolute values will be displayed in the same outputs as the change from baseline.

#### 9.1.2. Planned Imaging Statistical Analyses

#### **Planned Statistical Analyses**

#### Endpoint(s)

- Change from baseline in structural and inflammatory HOA features in the affected hand\* (including synovitis, erosive damage, cysts, osteophytes, cartilage space loss, malalignment, and bone marrow lesions) as assessed by the OMERACT HOAMRIS scoring system
- Change from baseline in structural and inflammatory HOA features in the affected hand\* (including synovitis, bone erosions, joint space width, and bone marrow edema) as assessed by the HOAMRIQ scoring system.

#### **Planned Statistical Analyses**

- Change from baseline in synovitis in the affected hand\*, as measured by DCE-MRI including
  the exchange rate (K<sup>trans</sup>), interstitial volume (v<sub>e</sub>), plasma volume (v<sub>p</sub>), volume of synovitis,
  initial rate of enhancement (IRE), and maximum signal intensity enhancement (ME).
- Change from baseline in bone shape as assessed by structural MRI of the affected hand.

#### **Planned Analyses and Model Specification**

- Descriptive Statistics will be calculated for the change from baseline in each individual component of the HOAMRIS (i.e. synovitis, erosive damage, cysts, osteophytes, cartilage space loss, malalignment and bone marrow lesions), as a total for the affected/dominant (whichever is scanned) hand.
- Individual Components of Interest in the HOAMRIS will be statistically analysed using the same methods as the primary endpoint (MMRM).
- Descriptive statistics will be calculated for each individual component of the HOAMRIQ (i.e. synovitis, erosive damage, cysts, osteophytes, cartilage space loss, malalignment and bone marrow lesions), a total for the affected/dominant (whichever is scanned) hand.
- Individual Components of Interest in the HOAMRIQ will be statistically analysed using the same methods as the primary endpoint (MMRM).
- Individual components of the HOAMRIQ may be presented as measured, standardized or both (see section 12.6.5 for full details).
- Descriptive Statistics will be calculated for the change from baseline in DCE-MRI quantitative derived parameters (i.e. K<sup>trans</sup>, v<sub>e</sub>, v<sub>p</sub>, IRE, ME and volume of synovitis), as a total for the affected/dominant (whichever is scanned) hand.
- DCE-MRI Parameters of interest will be statistically analysed using the same methods as the primary endpoint (MMRM).
- Individual components of the DCE-MRI may be presented as measured and standardized (see section 12.6.5 for full details).
- Descriptive Statistics will be calculated for the change from baseline in bone shape parameters (i.e. Surface area of bone) as a total for the affected/dominant (whichever is scanned) hand.
- All parameters will be listed by subject and joint/bone.

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

Results will be presented using the same methods as the primary endpoint.

#### **Sensitivity and Supportive Statistical Analyses**

- Non-parametric analyses may be conducted if the normality assumption does not hold.
- Analyses using different covariance structures may be explored if the unstructured covariance matrix does not converge.

# 9.2. Pharmacokinetic / Pharmacodynamic Analyses

The pharmacokinetic / pharmacodynamic (PK/PD) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

The primary goal of this analysis is to characterize the PK/PD relationship of GSK3196165 administered subcutaneously in subjects with HOA.

The analysis will be a graphical analysis and if data permits model based analysis might be conducted on adhoc basis. Overall plots will be generated for response/biomarker data against GSK3196165 exposure parameter.

Examples of the PK/PD plots include:

- Scatter plot of change from baseline in 24h average hand pain intensity at week 4 versus pre-dose concentration values (C<sub>trough</sub>) at week 4.
- Scatter plot of change from baseline in 24h average hand pain intensity at week 6 versus C<sub>trough</sub> at week 6.

## 9.3. Biomarker Analyses

#### 9.3.1. Pharmacodynamic Biomarker Analyses

#### 9.3.1.1. Overview of Planned Pharmacodynamic Biomarker Analyses

The pharmacodynamic biomarker analyses will be based on the "Safety" population, unless otherwise specified.

See section 12.6.6.1 for a full list of Pharmacodynamic Biomarkers.

Table 10 provides an overview of the planned pharmacodynamic biomarker analyses, with full details of data displays being presented in Appendix 16: List of Data Displays.

All Biomarkers may require transformations; see Section 12.5.3 regarding the process of presenting log transformed data.

Prior to any data being analysed, the distributions and proportion of data falling within the quantification limits will be assessed to determine if analysis is appropriate.

Additional analysis assessing the relationship between biomarkers and clinical efficacy endpoints may be conducted if considered appropriate.

Table 10 Overview of Planned Pharmacodynamic Biomarker Analyses

| Endpoint | | Transformed/Untransformed | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - | | | A | Absolu | ıte | | Change from Baseline | | | | | | | |
| | Stat | s Ana | lysis | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Τ | F | L | Т | F | F | L | Τ | F | L | Т | F | F | L |
| Target Engagement Bi | omark | ers | | | | | | | | | | | | |
| Distribution | | | | | Υ | | | | | | | | | |
| By Treatment & Time | | | | <b>Y</b> [1] | Υ | | Υ | | | | Υ | Υ | | Υ |

| Endpoint | Transformed/Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Δ | bsolu | ıte | | Change from Baseline | | | | | | | |
| | Stat | s Ana | lysis | Sum | mary | Indiv | ridual | Stat | s Ana | lysis | Summary | | Indiv | ridual |
| | Т | F | L | Т | F | F | L | Т | F | L | T | F | F | L |
| Predictive Biomarkers | | | | | | | | | | | | | | |
| Distribution | | | | | Υ | | | | | | | | | |
| By Treatment & Time | Υ | Υ | Y<br>[1,2] | <b>Y</b> [1] | Υ | | Υ | Υ | Υ | <b>Y</b> [2] | Υ | Υ | | Υ |
| Cartilage Biomarkers | ı | ı | ı | ı | | ı | | ı | ı | ı | ı | ı | ı | |
| Distribution | | | | | Υ | | | | | | | | | |
| By Treatment & Time | | | | <b>Y</b> [1] | Υ | | Υ | | | | Υ | Υ | | Υ |
| Mechanistic Biomarker | s | | | | | | | | | | | | | |
| Distribution | | | | | Υ | | | | | | | | | |
| By Treatment & Time | | | | <b>Y</b> [1] | Υ | | Υ | | | | Υ | Υ | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Absolute values will be displayed in the same outputs as the change from baseline.
- [2] [1] Raw SAS log output from analysis.

## 9.3.2. Safety Biomarker Analyses

#### 9.3.2.1. Overview of Planned Safety Biomarker Analyses

The safety biomarker analyses will be based on the "Safety" population, unless otherwise specified. See section 12.6.6.2 for a full list of Safety Biomarkers.

Table 11 provides an overview of the planned safety biomarker analyses, with full details of data displays being presented in Appendix 16: List of Data Displays.

Table 11 Overview of Planned Safety Biomarker Analyses

| Endpoint | Transformed/Untransformed | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | A | bsolu | ite | | | Change from Baseline | | | | | | |
| | Stat | s Ana | lysis | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Safety Biomarkers | | | | | | | | | | | | | | |
| Distribution | | | | | Υ | | | | | | | | | |
| By Treatment & Time | | | | Y[1] | Υ | | Υ | | | | Υ | Υ | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - [1] Absolute values will be displayed in the same outputs as the change from baseline.

## 9.4. Analyses on Paracetamol Data

## 9.4.1. Overview of Planned Analyses on Paracetamol Data

The analyses on the paracetamol data will be based on the "Intent-to-Treat" population, unless otherwise specified.

Table 12 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Section 12.15: List of Data Displays.

Table 12 Overview of Planned Analyses on Paracetamol Data

| Endpoint | | | F | bsolu | te | | Change from Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | Sum | Summary | | Individual | | Stats Analysis | | | Summary | | idual | |
| | Т | F | Г | Т | F | F | L | Т | F | L | Т | F | F | Г |
| Paracetamol | | | | | | | | | | | | | | |
| 24h Dose of | | | | <b>Y</b> [1] | <b>Y</b> [1] | | Υ | | | | <b>Y</b> [1] | <b>Y</b> [1] | | |
| Paracetamol Averaged | | | | | | | | | | | | | | |
| over 7 Days Prior to | | | | | | | | | | | | | | |
| Assessment | | | | | | | | | | | | | | |
| Proportion of Subjects | | | | Υ | | | | | | | | | | |
| Using Paracetamol | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Absolute values will be displayed in the same outputs as the change from baseline.
#### 10. INTERIM ANALYSES

Two formal interim analyses are planned during the course of this study. In addition to the formal planned interim analyses, further data reviews may be carried out by senior managers not involved in the study conduct to aid in portfolio and budget decisions. These administrative reviews will have no impact on the ongoing study.

The timing and content of each Interim deliverable is summarised in Table 13.

**Table 13 Interim Deliveries** 

| Analysis | Timing | <b>Unblinded Team</b> | Main Objective |
|---|---|---|---|
| PK Interim | To coincide with other internal decision making across the GSK3196165 project | Study Pharmacokineticist, Statistics and Programming, Project Statistician, GSK3196165 MDT | To compare PK of GSK3196165 in subjects with HOA with other populations |
| Week 6<br>Interim | Once a minimum of 30 subjects have completed day 43 (week 6) | Study Statistician and<br>Programmer, Project<br>Statistician and<br>Programmer, TA<br>Head, Clinical<br>Statistics TA Head,<br>MDL | To assist with decision making regarding the subsequent clinical development of GSK3196165 for OA |
| Administrative<br>Interim Data<br>Review | At the discretion of<br>Senior Managers<br>not involved in the<br>study conduct | Study Statistician and<br>Programmer, Project<br>Statistician and<br>Programmer, TA<br>Head, Clinical<br>Statistics TA Head,<br>MDL | To aid with dynamic portfolio and budget decisions |

# 10.1. Overview of planned Week 6 Interim Analysis

#### 10.1.1. Overview of Study Population Analysis at Week 6 Interim

The Study Population analyses will be based on the Intent-to-Treat (ITT) population, unless otherwise specified.

Table 14 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 16: List of Data Displays.

Table 14 Overview of Planned Study Population Analyses at Week 6 Interim

| Display Type | Data Displays | s Generated |
|------------------------------------------|---------------|-------------|
| | Table | Listing |
| Demographic and Baseline Characteristics | | |
| Demographics Characteristics | Υ | |

#### NOTES:

• Y = Yes display generated.

#### 10.1.2. Overview of Safety Analysis at Week 6 Interim

The Adverse Event analyses will be based on the "Safety" population, unless otherwise specified.

Table 15 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 16: List of Data Displays.

Table 15 Overview of Planned Safety Analyses at Week 6 Interim

| Endpoint / Parameter/ Display Type | Absolute | | Cha | from BL | | | |
|---|---|---|---|---|---|---|---|
| | Summary Individual S | | Sumn | nary | Individual | | |
| | Т | F | F | L | Т | F | L |
| Adverse Events (AE's) | | | | | | | |
| All AE's | Υ | | | | | | |
| Serious and Other Significant AE's | | | | | | | |
| Serious AE's | Υ | | | | | | |
| Withdrawal AE's | Υ | | | | | | |
| Drug Related AE's | Υ | | | | | | |
| AE's leading to death | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 10.1.3. Overview of Planned Efficacy Analysis at Week 6 Interim

Table 17 provides an overview of the planned interim analyses, with full details of data displays being presented in Appendix 16: List of Data Displays

Table 16 Overview of Planned Efficacy Analysis at Week 6 Interim

| Endpoint | | Absolute | | | | | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Stats Analysis | | | Summary I | | Individual Sta | | Stats Analysis | | Summary | | Individual | |
| | Т | F | L | Τ | F | F | L | Т | F | L | Т | F | F | L |
| Pain | | | | | | | | | | | | | | |
| 24h average hand | | | | Υ | Y[2] | | | Υ | Υ | <b>Y</b> [1] | Y[2] | Y[2] | | |
| pain NRS score | | | | [2] | | | | | | | | | | |
| averaged over 7 | | | | | | | | | | | | | | |

| Endpoint | | | Α | bsol | ute | | | | Ch | ange | from E | Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Analysis | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | Т | F | F | L | T | F | L | Т | F | F | L |
| days prior to assessment | | | | | | | | | | | | | | |
| 24h worst hand pain<br>NRS score averaged<br>over 7 days prior to<br>assessment | | | | Y<br>[2] | <b>Y</b> [2] | | | Y | Y | <b>Y</b> [1] | <b>Y</b> [2] | <b>Y</b> [2] | | |
| AUSCAN | | | | | | | | | | | | | | |
| AUSCAN 3.1 NRS<br>Components | | | | | | Υ | | Y | Y | <b>Y</b> [1] | Y | Y | | |
| C-Reactive Protein | | | | | | | | | | | | | | |
| C-Reactive Protein | | | | Y<br>[2] | Υ[2] | | | Υ | Y | <b>Y</b> [1] | <b>Y</b> [2] | <b>Y</b> [2] | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - [1] Raw SAS log output from Analysis.
  - [2] Absolute value and change from baseline will be displayed on the same output

## Week 6 Interim Analysis

#### **Model Specification**

 Continuous endpoints will be statistically analysed using the same methods as described in Sections 7.1.2 and 8.1.2.1

#### **Model Checking & Diagnostics**

Refer to Appendix 11: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Continuous endpoints will be presented using the same methods as described in Sections 7.1.2 and 8.1.2.1

#### **Sensitivity and Supportive Statistical Analyses**

- Following review of the data, additional analyses maybe conducted to further support the primary statistical analyses, if deemed appropriate.
- Analyses using different covariance structures may be explored if considered appropriate.

# 10.2. Overview of planned Pharmacokinetic Interim Analysis

The pharmacokinetic (PK) analysis will be based on the "Pharmacokinetic" population, unless otherwise specified.

The primary objective of the interim PK analysis is to compare PK of GSK3196165 in subjects with HOA with other populations. Plot of GSK3196165 concentration with median value by visit will be produced and compared with similar plot from BAROQUE study including data only till week 12 and 180 mg dose group.

To derive PK parameters, GSK3196165 serum concentration-time data from HOA will be pooled with dataset generated for population PK meta analysis (Population Pharmacokinetic Analysis of GSK3196165 Following Intravenous and Subcutaneous Administration to Healthy Volunteers, Subjects with Rheumatoid Arthritis and Multiple Sclerosis (Date: 08-Jan-2016)) and subjected to nonlinear mixed effects modelling using the program NONMEM. Effect of following covariates will be tested:

- Population type (HOA, healthy volunteers, rheumatoid arthritis and multiple sclerosis)
- Subject demographics (age, sex, and race)
- Baseline characteristics (body weight, free GM-CSF levels)
- Immunogenicity

Individual PK parameters will be summarized by population type and distribution of the derived PK parameters will be plotted by population type.

#### 10.3. Overview of Administrative Interim Data Review

The purpose of the Administrative Interim Data Review is to aid with dynamic portfolio and budget decisions. The outcome of the Administrative Interim Data Review will have no direct impact on the ongoing study.

Table 17 provides an overview of the planned analyses, with full details of data displays being presented in Section 12.15: List of Data Displays.

Table 17 Overview of Analyses for Administrative Interim Data Review

| Endpoint | | | - | Absolu | te | | | | Cł | nange | from | Basel | ine | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Stats Analysis | | | mary | Indiv | Individual | | Stats Analysis | | | Summary | | Individual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Pain | | | | | | | | | | | | | | |
| 24h average hand | | | | | | | | Υ | Υ | | Υ | Υ | | |
| pain NRS score | | | | | | | | | | | | | | |
| averaged over 7 days | | | | | | | | | | | | | | |
| prior to assessment | | | | | | | | | | | | | | |
| 24h worst hand pain | | | | | | | | Υ | Υ | | Υ | Υ | | |
| NRS score averaged | | | | | | | | | | | | | | |
| over 7 days prior to | | | | | | | | | | | | | | |
| assessment | | | | | | | | | | | | | | |
| Paracetamol | | | | | | | | | | | | | | |
| 24h Dose of | | | | | | | | | | | | Υ | | |
| Paracetamol | | | | | | | | | | | | | | |
| Averaged over 7 | | | | | | | | | | | | | | |


204851

| Endpoint | | Absolute | | | | | | | | Change from Baseline | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Summary | | Individual | | Stats Analysis | | | Summary | | Individual | |
| | T | F | L | Т | F | F | L | Т | F | L | Т | F | F | Г |
| Days Prior to | | | | | | | | | | | | | | |
| Assessment | | | | | | | | | | | | | | |
| Proportion of | | | | Υ | | | | | | | | | | |
| Subjects Using | | | | | | | | | | | | | | |
| Paracetamol | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 11. REFERENCES

[1] Population Pharmacokinetic Analysis of GSK3196165 Following Intravenous and Subcutaneous Administration to Healthy Volunteers, Subjects with Rheumatoid Arthritis and Multiple Sclerosis (Date: 08-Jan-2016)

# 12. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 12.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 12.2 | Appendix 2: Time and Events |
| Section 12.3 | Appendix 3: Assessment Windows |
| Section 12.4 | Appendix 4: Treatment States & Phases |
| Section 12.5 | Appendix 5: Data Display Standards & Handling Conventions Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 12.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic and or Biomarkers |
| Section 12.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 12.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 12.9 | Appendix 9: Multicentre Studies |
| Section 12.10 | Appendix 10: Multiple Comparisons and Multiplicity |
| Section 12.11 | Appendix 11: Model Checking and Diagnostics for Statistical Analyses |
| Section 12.12 | Appendix 12: Definition of some Parameters of Interest |
| Section 12.13 | Appendix 13: Opportunistic Infections: MedDRA Preferred Terms |
| Other RAP App | endices |
| Section 12.14 | Appendix 14: Abbreviations & Trade Marks |
| Section 12.15 | Appendix 15: List of Data Displays |
| Section 12.16 | Appendix 16: Example Mock Shells for Data Displays |

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

There is no planned Per Protocol population in this phase IIa study.

# 12.2. Appendix 2: Time & Events

#### 12.2.1. Protocol Defined Time & Events

## 12.2.1.1. Screening period Time and Events table

| (must be c | Subject Screening<br>arried out ≤ 28 days prior to Day 1) | |
|---|---|---|
| Screening Day 1 | Screening Days 1-7, at home | Screening Day ≥8 |
| <b>\</b> | | 1 |
| Informed Consent | Daily Pain NRS questionnaire[2] | Pain NRS eligibility assessment <sup>[3]</sup> |
| Inclusion/exclusion criteria | | MRI <sup>[4]</sup> |
| Demographics | | |
| Medical/medication/alcohol history | | |
| Con. Med. Review | | |
| Vital signs | | |
| 12-lead ECG | | |
| Full Physical Exam | | |
| Swollen and tender joints <sup>[1]</sup> | | |
| Haem/Chem/Urinalysis | | |
| HIV, TB, Hepatitis B & Hepatitis C screen | | |
| RF, ACPA (anti-CCP) | | |
| Pregnancy test (serum) | | |
| Urine drug / alcohol screen | | |
| Spirometry (FEV1, FVC) & DLCO | | |
| Pain NRS training | J | |
| SAE assessment | | |

#### NOTES:

- [1] Where possible, the same individual should perform all disease assessments for an individual subject (with separate joint assessor).
- [2] Pain NRS questions should be completed at approximately the same time each day (recommended between 6pm and 10pm).
- [3] Eligibility assessment will be based on a 7 day average of the '24h average hand pain NRS' question.
- [4] Subjects must have passed all screening assessments, including laboratory tests and 7-day pain NRS assessment, prior to undertaking MRI scanning.

#### 12.2.1.2. Treatment period Time and Events table

| | δ | | | | | Treatm | ent peri | od | | | | = | 2 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | days | Wee | k 0 | Wk 1 | Wk 2 | Wk 3 | Wk 4 | Wk 6 | Wk 8 | Wk 10 | Wk 12 | <b>s ca</b> | ek 2<br>d) |
| Study events | Screening (≤28 on prior to Day 1 | Baseline & Day<br>1 treatment visit | Day 3 (± 1d)PK<br>biomarker visit | Day 8 (± 1d)<br>treatment visit | Day 15 (± 1d)<br>treatment visit | Day 22 (± 1d)<br>treatment visit | Day 29 (± 1d)<br>treatment visit | Day 43 (± 3d)<br>treatment visit | Day 57 (± 3d)<br>treatment visit | Day 71 (± 3d)<br>treatment visit | Day 85 (± 3d)<br>treatment visit | Week 20 phone call (Day 141 $\pm$ 5d) | <b>Follow up</b> (Week 22 (Day 155 ± 7d) |
| Borg CR10 Scale <sup>[1]</sup> | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | ~ ~: | |
| Patient <sup>[1]</sup> and physician global assessment <sup>[2]</sup> | | Χ | | | Χ | | Χ | | Χ | | Х | Site to contact subject by phone and remind them to begin completing the daily Pain NRS questionnaire starting 7 days before their Follow-up visit at Week 22 | |
| AUSCAN 3.1 NRS[1] | | Χ | | Χ | Х | | Χ | Χ | Χ | Х | Х | th<br>at W | |
| Brief Physical Exam | | Χ | | | Χ | | Χ | | Χ | | Χ | oletir<br>isit a | |
| Vital signs | See separate T&E table for screening procedures | Χ | | | Χ | | Χ | | Χ | | Χ | n dr<br>dwc | res |
| 12-lead ECG | Sedi | X <sup>4</sup> | | | | | | | | | Χ | in co<br>Jw-L | See separate table for follow-up visit procedures |
| Swollen and tender joints <sup>[2]</sup> | pro | Χ | | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | peg<br>-ollc | oroc |
| MRI <sup>[3]</sup> | ing | | | | | | | | | | X <sup>[3]</sup> | n to<br>eir F | isit |
| Haem/Chem/Urinalysis | eeu | Χ | | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | hen<br>e th | ^ dr |
| PK sampling <sup>[4]</sup> | SCI | Χ | Χ | Χ | | | Χ | Χ | | | Χ | nd t<br>efor | J-WC |
| Blood Biomarkers <sup>[4]</sup> | Į Į | Χ | Χ | Χ | Χ | | Χ | | Χ | | Χ | emi<br>/s b | 톟 |
| Urine drug/alcohol | table | Χ | | | | | | | | | Χ | nd r<br>day | fo |
| Study treatment dosing | Ä<br>T | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | ie a<br>ng 7 | aple |
| Cough, Auscultation, Pulse Oximetry | E — | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | ohor<br>:artii | Ite t |
| Spirometry (FEV1, FVC) & D <sub>LCO</sub> | arat | Χ | | | | | | | | | Χ | by p | oara |
| Immunogenicity blood sampling | sep | <b>X</b> [5] | | | Χ | | Χ | | | | Χ | ect<br>nair | seg |
| Pharmacogenetics <sup>[6]</sup> | )ee | Χ | | | | | | | | | | subj<br>tion | See |
| Pregnancy test (urine) | 0) | Χ | | | | | Χ | | Χ | | Χ | act s<br>lues | |
| Post-treatment Interview | | | | | | | | | | | Χ | onta<br>SS q | |
| Daily Pain NRS questions[7] | | < | | | | | - X | | | | > | to c<br>NR | |
| SAE/AE assessment | | <> | | | | | | Site to contact subject by phone Pain NRS questionnaire starting | | | | | |
| Con. medication review | | < | | | | | - X | | | | > | 1 | |

#### Treatment period T&E table notes

- [1] PROs are performed before any other assessments, or procedures, to avoid influencing subject.
- [2] Where possible, the same individual should perform all disease assessments for an individual subject (with separate joint assessor).
- [3] MRI scanning at week 12 may take place on a separate day from other assessments and may occur on Day 85 (± 5d).
- [4] Before dosing.
- [5] Day 1 immunogenicity sample includes anti-GM-CSF auto-antibody analysis
- [6] Consenting subjects only.
- [7] Pain NRS questions should be completed at approximately the same time each day (recommended between 6pm and 10pm).

# 12.2.1.3. Follow up visit and early withdrawal\* procedures list

| Subject Follow-up Visit<br>Task List |
|---------------------------------------------------------------------|
| Week 22 |
| (Day 155 $\pm$ 7d) |
| ↓ |
| Borg CR10 Scale[1] |
| Patient <sup>1</sup> and physician global assessment <sup>[3]</sup> |
| Pain NRS assessment <sup>[2]</sup> |
| Vital signs |
| Full Physical Exam |
| Swollen and tender joints <sup>[3]</sup> |
| SAE/AE assessment |
| Con. Med. Review |
| Pregnancy test (urine) |
| Haem/Chem/Urinalysis |
| Immunogenicity |
| MRI <sup>[4]</sup> |
| Blood Biomarkers |
| PK Sampling |
| Cough, Auscultation, Pulse Oximetry |
| Spirometry (FEV1, FVC) & D <sub>LCO</sub> |

#### NOTES:

- [1] PROs are performed before any other assessments, or procedures, to avoid influencing subject.
- [2] Assessment is based on a 7 day average of the Pain NRS questions.
- [3] Where possible, the same individual should perform all disease assessments for an individual subject (with separate joint assessor).
- [4] If scheduling MRI on the same day as the follow up visit is not possible, the MRI visit may take place on a separate day *before the Follow-up visit* but it must occur within the same Day 155 ±7day window.

<sup>\*</sup>for early withdrawal, Day 85 procedures are followed and a follow up visit scheduled.

# 12.3. Appendix 3: Assessment Windows

# 12.3.1. Definitions of Assessment Windows for Analyses

| Analysis Set | Parameter | Target | Analysis | Window | Analysis |
|---|---|---|---|---|---|
| / Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | Timepoint |
| All | All | Day -1 | Day -28 | Day -1 | Screening |
| MRI | MRI | Day -1 | Day -28 | Day 1 | Baseline |
| All | All | Day 1 | Day 1 | Day 1 | Baseline |
| PK/Biomarker | PK/Biomarker | Day 3 | Day 2 | Day 4 | Day 3 |
| All | All | Day 8 | Day 6 | Day 10 | Week 1 |
| All | All | Day 15 | Day 13 | Day 17 | Week 2 |
| All | All | Day 22 | Day 20 | Day 24 | Week 3 |
| All | All | Day 29 | Day 27 | Day 31 | Week 4 |
| All | All | Day 43 | Day 38 | Day 48 | Week 6 |
| All | All | Day 57 | Day 52 | Day 62 | Week 8 |
| All | All | Day 71 | Day 66 | Day 76 | Week 10 |
| All | All | Day 85 | Day 80 | Day 90 | Week 12 |
| MRI | MRI | Day 85 | Day 76 | Day 94 | Week 12 |
| All | All | Day 155 | Day 148 | Day 162 | 12 Week<br>Follow Up |
| All (subjects<br>withdrawn early<br>from treatment) | All (subjects<br>withdrawn early<br>from treatment) | 84 days after last treatment | 77 days after last treatment | 91 days after last treatment | 12 Week<br>Follow Up |

Note: All data will be listed, but 'out of window' data would not contribute towards any summary statistics or analyses.

Note: MRI rescan visits will be slotted to the nearest analysis time window and will contribute towards summary statistics and analyses.

## 12.4. Appendix 4: Treatment States and Phases

# 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment start date, unless otherwise specified.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date + 14 Days |
| Safety Follow-Up | Date > Study Treatment Stop Date + 14 Days |

#### 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before first dose of study treatment. |
| Concomitant | Any medication that is not a prior |

#### NOTES:

Please refer to Appendix 7 for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### 12.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 12.4.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 14 Days |
| Safety Follow-Up | AE Start Date > Study Treatment Stop Date + 14 Days |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

AE's with partial start and/stop dates will be assumed to have occurred on treatment unless there is
evidence through comparison of partial dates to suggest otherwise.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

## 12.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code Description | | Description | Order [1] |
| Α | GSK3196165 180mg | GSK3196165 180mg | 2 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

#### 12.5.2. Baseline Definition & Derivations

#### 12.5.2.1. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in<br>Data Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Primary | | | |
| 24h average hand pain NRS score averaged over 7 days prior to assessment <sup>[1]</sup> | X | X | Day 1 (Pre-Dose) |
| Secondary | | | |
| 24h worst pain NRS score<br>averaged over 7 days prior to<br>assessment <sup>[1]</sup> | X | X | Day 1 (Pre-Dose) |
| AUSCAN 3.1 NRS | | X | Day 1 (Pre-Dose) |
| Swollen/Tender hand joints | | X | Day 1 (Pre-Dose) |
| PtGA/PhGA | | X | Day 1 (Pre-Dose) |
| PK parameters | | Χ | Day 1 (Pre-Dose) |
| Safety | Safety | | |
| Vital signs (HR, BP & temp)[2] | Χ | Χ | Day 1 (Pre-Dose) |
| ECG (12-lead)[2] | Χ | X | Day 1 (Pre-Dose) |
| Laboratory (Haematology, clinical chemistry and urinalysis) <sup>[2]</sup> | X | X | Day 1 (Pre-Dose) |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

| Parameter | Study Assessments Considered As Baseline | | Baseline Used in<br>Data Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose) | |
| Pulmonary Assessments <sup>[2]</sup> | X | X | Day 1 (Pre-Dose) |
| Exploratory | | | |
| MRI | X | | Screening |
| PK/PD | | Х | Day 1 (Pre-Dose) |

#### NOTES:

- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- Where both screening and pre-dose are available, the value closest to first dose will be used.
- [1] For all Pain NRS scores averaged over 7 days prior to assessment, the baseline values will be calculated as the average of the 7 days preceding the first dose of study treatment
- [2] For all vital signs, ECG, labs and pulmonary assessments except D<sub>LCO</sub>, the baseline values will be the latest pre-dose assessment. For D<sub>LCO</sub>, a subject's baseline will be taken as the lowest value obtained from the Screening or Day 1(Pre-dose) assessment, or any unscheduled visit in between.

#### 12.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | <ul> <li>Calculate the change from baseline at each given time point<br/>and determine the maximum change.</li> <li>Note that for the ECG outputs this is the maximum increase<br/>from baseline</li> </ul> |
| Ratio to Baseline | = Post-Dose Visit Value / Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 12.5.2.1 Baseline Definitions will be
  used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 12.5.3. Reporting Process & Standards

| <b>Reporting Process</b> | |
|---|---|
| Software | |
| The currently supported versions of SAS software will be used to perform all data analyses, generate tables, figures and listings. | |
| Reporting Area | |
| HARP Server | uk1salx00175 |
| HARP Area | arenv \ arprod \ gsk3196165 \ mid204851 \ final |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ primary |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ internal_01 |

| Reporting Process | |
|---|---|
| | arenv \ arprod \ gsk3196165 \ mid204851 \ internal_02 |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ internal_03 |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ internal_04 |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ internal_05 |
| | arenv \ arprod \ gsk3196165 \ mid204851 \ spotfire |
| QC Spreadsheet | arenv \ arwork \ gsk3196165 \ mid204851 \ final \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ primary \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ internal_01 \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ internal_02 \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ internal_03 \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ internal_04 \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ internal_05 \ documents |
| | arenv \ arwork \ gsk3196165 \ mid204851 \ spotfire \ documents |

#### **Analysis Datasets**

- For the final reporting effort, analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & AdaM IG Version 1.0
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.
- For the purpose of the Administrative Interim Review and Interim analyses, analysis datasets will be generated from SI Datasets.

#### **Generation of RTF Files**

RTF files will be generated for final reporting effort.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL)\* will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.

<sup>\*</sup> website IDSL → supporting documentation → component → stats displays → principles

#### **Reporting Standards**

- The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations)
     will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or contribute to any analyses, unless otherwise stated.
- Unscheduled visits will not be included in figures, unless otherwise stated.
- All unscheduled visits will be included in listings.

| 7 th direction and the term be included in hearinger | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | nacokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Log-Transformed Parameters | |
| Descriptive<br>Summary Statistics | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and geometric coefficient of variation (CV <sub>b</sub> (%)) will be reported. [1] CV <sub>b</sub> (%) = √ (exp(SD²) - 1) * 100 (SD = SD of log transformed data) |
| Figures | Axes will be presented with actual values with an appropriate log-scale (either base 2 or base 10) depending on range of values |
| Graphical Displays | |
| Refer to IDSL St | Refer to IDSL Statistical Principals 7.01 to 7.13. |

## 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used except for ECGs, Blood Pressure and Pulse Rate Measures. If values are the same distance from the target, then the latest assessment value will be taken.
- Triplicate ECG measures will be averaged for each subject and visit prior to generating summary tables.
- Duplicate Blood Pressure and Pulse Rate measures will be averaged for each subject and visit prior to generating summary tables.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from date of first dose of study treatment:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Date of First Dose of Study Treatment → Study Day = Ref Date -Date of First Dose of Study Treatment
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (First Dose of Study Treatment) + 1

#### 12.6.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Calculated as the integer part of (latest of (randomisation date, screening date) date of birth).
- Birth date will be presented in listings as 'YYYY'.
- Age will be categorised into subgroups <18 years, 18-<65 years and >=65 years

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### Race Category

- White: 'White: Arabic/North African Heritage' and 'White: White/Caucasian/European Heritage', or both of these, but no other category checked
- African descent: 'African American/African Heritage', and no other category checked

#### **Demographics**

 Asian: 'Asian – Central/South Asian Heritage', 'Asian – East Asian Heritage', 'Asian – Japanese Heritage', and 'Asian – South East Asian Heritage', or any combination of these, but no other category checked

Other: Any combination that has not been categorized above ('mixed race')

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

#### Duration of Exposure in Days = Treatment Stop Date – (Treatment Start Date) + 14

- Subjects who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Visits x Total Dose at Each Visit)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

#### **Medical History**

#### **Disease Duration**

- OA duration since diagnosis in months will be calculated based on the formula:
  - OA Duration Since Diagnosis in Months = (Date of First Dose of Study Treatment Start date of formal OA diagnosis + 1)/30.25
- OA duration since first symptoms in months will be calculated based on the formula:
  - OA Duration Since First Symptoms in Months = (Date of First Dose of Study Treatment Start date of first symptoms + 1)/30.25

#### 12.6.3. Safety

#### **ECG Parameters**

#### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{OTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value, THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

#### **ECG Parameters**

$$TCB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$
  $QTCF$ 

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Places= '< x ' becomes x 0.01
  - Example 2: 1 Decimal Place= '> x' becomes x + 0.1
  - Example 3: 0 Decimal Places= '< x' becomes x 1

#### **Pulmonary Assessments**

#### **Borg CR10**

- The Borg CR10 Scale is being used to assess patient-reported shortness of breath (difficulty in breathing)
- The Borg CR10 Scale® is graded from:
  - o 0, "Nothing at all", = none, to 10, "Extremely Strong", "Maximal", = the most intense perception or feeling the subject has ever experienced.
  - There is allowance for gradings > 10, which are designated as "Absolute Maximum" or "Highest Possible" and is marked with a "●" in the scale
  - A 3 is designated as being "Moderate" on the scale.
- No imputations will be done for missing data.

#### **Pulse Oximetry**

- Pulse Oximetry will be categorised into subgroups <80%, 80% to 90% and ≥90%.
- Lower values represent a worse result.

#### **12.6.4.** Efficacy

#### **Efficacy**

#### 24h average hand pain NRS score

- Measured by a daily pain Numerical Rating Scale (NRS) based on 24h average hand pain intensity with anchors "0" (no pain) and "10" (worst imaginable pain), which is averaged over the 7 days prior to assessment visit with GSK3196165 or placebo.
- The 7 day average score is calculated by

 $\sum$ (Daily 24h average hand pain NRS scores in the 7 days prior to assess

Total numer of days 24h average hand pain NRS is recorded in 7 days prior to

 \* If a subject records their daily pain NRS scores for less than 4 days out of the 7 days prior to assessment visit, then the average NRS score for the week prior to the assessment visit will be recorded as missing.

#### **Efficacy**

• The 7 day average score will be calculated using the 7 days prior to assessment visit, excluding any values that have been used to calculate previous averages, e.g. if a patient attends a visit on Day 9 (hence 7 day average will be calculated using Days 2 to 8) and attends their next visit on Day 14 (hence 7 day average should be calculated using Days 7 to 13), any overlapping days will be excluded from the calculation of the Day 14 average (i.e. Days 7 and 8).

#### 24h worst hand pain NRS score

- Measured by patients using a daily pain Numerical Rating Scale (NRS) based on 24h worst hand pain intensity with anchors "0" (no pain) and "10" (worst imaginable pain, which is averaged over the 7 days prior to assessment visit with GSK3196165 or placebo.
- The score is calculated by
  - $\Sigma$ (Daily 24h worst hand pain NRS scores in the 7 days prior to assessment visit)
  - Total numer of days 24h worst hand pain NRS is recorded in 7 days prior to assessment visit\*
- \* If a subject records their daily pain NRS scores for less than 4 days out of the 7 days prior to assessment visit, then the average NRS score for the week prior to the assessment visit will be recorded as missing.
- The 7 day average score will be calculated using the 7 days prior to assessment visit, excluding any values that have been used to calculate previous averages, e.g. if a patient attends a visit on Day 9 (hence 7 day average will be calculated using Days 2 to 8) and attends their next visit on Day 14 (hence 7 day average should be calculated using Days 7 to 13), any overlapping days will be excluded from the calculation of the Day 14 average (i.e. Days 7 and 8).

#### **AUSCANTM**

- The AUSCAN™ Index is a self-administered questionnaire consisting of a 15-item scale which measures pain (5 items), stiffness (1 item) and degree of disability/physical function (9 items) during the preceding 48h. All items are rated on an NRS scale with anchors "0" (none) to "10" (extreme).
- The scores for each individual domain (Pain/Stiffness/Physical Function) are calculated using a simple summation of the component item scores relating to that domain, therefore the Pain component ranges from 0-50, Stiffness component 0-10 and Physical Function component (0-90).
- The total AUSCAN™ score is calculated using simple summation of the 15 component item scores and therefore ranges from 0-150.
- If ≥2 pain, the stiffness, >2 physical function items are missing, the patient's response on the affected subscale will be regarded as invalid and the deficient subscale(s) will not be used in any analysis.
- Where 1 pain or 1-2 physical function items are missing, the average value for the subscale will be substituted in lieu of the missing item value(s).

#### **Swollen Hand Joint Count**

- Measured by the total number of swollen joints out of a possible 30 (8 DIP, 8 PIP, 2 IP, 10 MCP, 2 CMC) across both hands.
- If there are missing observations for swollen joints then the remaining observations will be
  assessed and weighted by dividing the number presented by the number of non-missing,
  and by multiplying by 30 for the joint count.

#### **Efficacy**

- No imputations for individual joints will be done.
- If a joint is not evaluable at Baseline, then that joint is set to missing throughout the study.
- If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.

#### Painful/Tender Hand Joint Count

- Measured by the total number of tender joints out of a possible 30 (8 DIP, 8 PIP, 2 IP, 10 MCP, 2 CMC) across both hands.
- Joints can be rated 0=no pain/tenderness, 1=mild pain, 2=moderate pain and 3=severe pain.
- A joint is considered tender if it is scored >0 on the tender joint severity scale.
- If there are missing observations for tender joints then the remaining observations will be assessed and weighted by dividing the number presented by the number of non-missing, and by multiplying by 30 for the joint count.
- No imputations for individual joints will be done.
- If a joint is not evaluable at Baseline, then that joint is set to missing throughout the study.
- If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.

#### Patient Global Assessment (PtGA)

- Measured by patients who will complete a global assessment of disease activity using the
  patient global assessment (PtGA) item, an NRS with anchors "0" (very well) to "10" (very
  poor).
- No imputations for missing data will be done.

#### Physician Global Assessment (PhGA)

- Measured by Physicians who will complete a global assessment of disease activity using the physician global assessment item (PhGA), an NRS with anchors "0" (none) to "10" (extremely active).
- No imputations for missing data will be done.

#### 24h Paracetamol Dose

- Measured by total dose of paracetamol taken in 24 hours, which is averaged over the 7 days prior to assessment visit with GSK3196165 or placebo.
- If paracetamol dose is missing on a particular day but a pain NRS score has been recorded on that day, then paracetamol dose is set to 0mg for that day.
- If paracetamol dose is missing on a particular day and a pain NRS score is also missing on that day, then paracetamol dose is set to missing for that day.
- The 7 day average dose is calculated by  $\sum$  (Daily 24h paracetamol doseage in the 7 days prior to assessment visit)

Total numer of days 24h paracetamol dose is recorded in 7 days prior to assessment visit\*

- \* If a subject is missing more than 3 daily paracetamol doses out of the 7 days prior to assessment visit, then the average paracetamol dose for the week prior to the assessment visit will be recorded as missing.
- The 7 day average dose will be calculated using the 7 days prior to assessment visit, excluding any values that have been used to calculate previous averages, e.g. if a patient attends a visit on Day 9 (hence 7 day average will be calculated using Days 2 to 8) and

#### **Efficacy**

attends their next visit on Day 14 (hence 7 day average should be calculated using Days 7 to 13), any overlapping days will be excluded from the calculation of the Day 14 average (i.e. Days 7 and 8).

## 12.6.5. Imaging

#### **Imaging**

#### **HOAMRIS**

- HOAMRIS measures consist of 7 different parameters (Synovitis, Erosive Damage, Cyst, Osteophytes, Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions) that are semiquantitatively assessed by an independent reviewer on a scale of 0-3/3.5, or can be scored as "Not Visible" or "Surgically Modified".
- Each parameter is evaluated on a total of 8 hand joints (DIP Joints 2-5 and PIP Joints 2-5). For erosive damage, cysts, and bone marrow lesions, the distal and proximal ends of the joint are assessed as sub-regions (i.e. D1, D2, P1, and P2).
- There is one score for each parameter per location, per time point.
- Each parameter is scored as follows:
  - Synovitis Scoring:

| Score | Description |
|---|---|
| 0 | Normal, no synovitis |
| 0.5 | Minimal: >0 but decreased from a timepoint scored 1. |
| 1 | Mild: 1-33% volume enhancement |
| 1.5 | Mild-Moderate: >0 and <2, but increased from a timepoint scored 1 or decreased |
| | from a timepoint scored 2. |
| 2 | Moderate: 34-67% volume enhancement |
| 2.5 | Moderate-Severe: >1 and <3, but increased from a timepoint scored 2 or decreased |
| | from a timepoint scored 3. |
| 3 | Severe: 68-100% volume enhanced |
| 3.5 | Very Severe: Increased from a timepoint scored 3. |
| N | Not Visible |
| S | Surgically Modified |

#### Erosive Damage Scoring:

| | 8 |
|---|---|
| Score | Description |
| 0 | Normal, no erosive damage |
| 0.5 | Minimal: >0 but decreased from a timepoint scored 1. |
| 1 | Mild: ≤10% of bone volume or ≤25% joint surface affected |
| 1.5 | Mild-Moderate: >0 and <2, but increased from a timepoint scored 1 or decreased |
| | from a timepoint scored 2. |
| 2 | Moderate: 11-20% of bone volume and/or 26-50% of joint surface affected |
| 2.5 | Moderate-Severe: >1 and <3, but increased from a timepoint scored 2 or decreased |
| | from a timepoint scored 3. |
| 3 | Severe: >20% of bone volume and/or >50% of joint surface affected |
| 3.5 | Very Severe: Increased from a timepoint scored 3. |

| <b>Imaging</b> | | |
|----------------|---|---------------------|
| | N | Not Visible |
| | S | Surgically Modified |

# Cyst Scoring:

| Score | Description |
|-------|-------------------------------------------|
| 0 | Normal, no cyst development |
| 1 | Mild: cysts are ≤10% of bone volume |
| 2 | Moderate: cysts are 11-20% of bone volume |
| 3 | Severe: cysts are >20% of bone volume |
| N | Not Visible |
| S | Surgically Modified |

# o Osteophyte Scoring:

| Score | Description |
|-------|-----------------------------------------------------------------|
| 0 | Normal, no osteophytes |
| 1 | Mild: 1-3 small osteophytes |
| 2 | Moderate: ≥4 small osteophytes and/or ≥1 moderate osteophyte(s) |
| 3 | Severe: at least 1 large osteophyte |
| N | Not Visible |
| S | Surgically Modified |

# o Cartilage Space Loss Scoring:

| Score | Description |
|---|---|
| 0 Normal, no loss of cartilage Space | |
| 1 | Mild: loss of cartilage space without bone-to-bone contact |
| 2 | Moderate: focal complete loss of cartilage space |
| 3 | Severe: complete cartilage space loss affecting >50% of articulating joint area |
| N | Not Visible |
| S | Surgically Modified |

# o Mal-alignment Scoring:

| Score | Description |
|---|---|
| 0 | Normal, no apparent mal-alignment |
| 1 | Mild: ≤10 degree angulation and/or not congruent joint surfaces |
| 2 Moderate: 11-20 degrees angulation and/or moderate subluxation without | |
| | the midline |
| 3 | Severe: >20 degrees angulation and/or subluxation without crossing the midline |
| N | Not Visible |
| S | Surgically Modified |

# O Bone Marrow Lesions:

| Score | Description |
|-------|------------------------------------------------------|
| 0 | Normal, no bone marrow lesions |
| 0.5 | Minimal: >0 but decreased from a timepoint scored 1. |
| 1 | 1 Mild: Lesions are 1-33% of bone volume |

| Imaging | | |
|---|---|---|
| | 1.5 | Mild-Moderate: >0 and <2, but increased from a timepoint scored 1 or decreased from a timepoint scored 2. |
| | 2 | Moderate: lesions are 34-66% of bone volume |
| | 2.5 | Moderate-Severe: >1 and <3, but increased from a timepoint scored 2 or decreased from a timepoint scored 3. |
| | 3 | Severe: lesions are 67-100% of bone volume |
| | 3.5 | Very Severe: Increased from a timepoint scored 3. |
| | N | Not Visible |
| | S | Surgically Modified |

- If an individual location is scored either "Not Visible" or "Surgically Modified" then the score for that location will be set to missing.
- Each individual Parameter will be presented as a total score for the affected/dominant hand which will be calculated by summing scores of all joints at each time point.

#### **HOAMRIQ**

- HOAMRIQ measures consist of the quantitative measurements from the bones and synovial capsules of the following joints:
  - o DIP Joints 2-5
  - o PIP Joints 2-5
  - o MCP Joints 1-5
  - o CMC-1
- 7 different parameters are quantitatively assessed as follows:
  - Synovitis (Volume of Enhancing Pannus):
    - The total volume (in mm<sup>3</sup>) of contrast-enhanced voxels within the synovial capsule.
    - The following joints will be considered:
      - CMC-1
      - DIP 2-5
      - PIP 2-5
      - MCP 1-5
    - Synovitis will be presented as a total measure which is calculated by summing the individual measure for each joint at each time point.
  - Synovitis (Normalised)
    - Normalised Synovitis will be calculated using the Volume of Enhancing Pannus (VEP):

$$\frac{\sum_{all\ joints} \textit{VEP}}{\sum_{all\ joints} \textit{Joint Volume}}$$

- The following joints will be considered:
  - CMC-1
  - DIP 2-5

#### **Imaging**

- PIP 2-5
- MCP 1-5

#### Erosive Damage (Volume of Bone Erosions):

- The volume (in mm<sup>3</sup>) difference between the segmented bones and modelled healthy bones within the 3D MR Image. The measure is taken at the extremities of the bones (15mm length from the joint) or the whole bone.
- The following bones will be considered:
  - D2-5
  - **12-5**
  - M2-5
  - P2-5
  - Trapezium
- Erosive Damage will be presented as a total measure which is calculated by summing the individual measure for each bone at each time point.

#### Erosive Damage (Normalised)

Normalised Erosive Damage will be calculated using the Volume of Bone:

$$\frac{\sum_{all\ bones} Volume\ of\ Bone\ Erosion}{\sum_{all\ bones} Volume\ of\ Bone}$$

- O Cyst:
- Measured as part of the erosions measurement and is therefore quantified but not differentiated from the quantification of erosions, hence no measure is presented separately for this parameter.

#### Osteophyte:

- Captured by Bone Shape Parameters, hence no measure is presented separately for this parameter.

#### Cartilage Space Loss (Joint Space Width):

- The mean difference (in mm) between corresponded patches on the ends of the phalanges of each joint.
- The following joints will be considered:
  - CMC-1
  - DIP 2-5
  - PIP 2-5
  - MCP 1-5
- Cartilage Space Loss will be presented as a total measure which is calculated by summing the individual measure for each joint at each time point.

#### Mal-alignment (Alignment of Bone):

- The 2D angle (in degrees) between phalanges at the DIP, PIP, MCP and CMC joints in the plane of the wrist bones.
- The following joints will be considered:

#### **Imaging**

- CMC-1
- DIP 2-5
- PIP 2-5
- MCP 1-5
- Mal-alignment will be presented as a total measure which is calculated by summing the absolute value of the individual measure for each joint at each time point.
- Bone Marrow Lesions (Volume of Bone Edema) (Normalised):
  - The total volume (in mm<sup>3</sup>) of enhanced voxels within the segmented bone volumes at each joint. The measure is taken at the extremities of the bones (15mm length from the joint), or the whole bone.
  - The following bones will be considered:
    - D2-5
    - **12-5**
    - M2-5
    - P2-5
    - Trapezium
  - Normalised Bone Marrow Lesions will be calculated using the volume of bone:

$$\frac{\sum_{all\ bones} Volume\ of\ Bone\ Edema}{\sum_{all\ bones} Volume\ of\ Bone}$$

 All parameters will be presented as a total measure for the affected/dominant hand at each time point.

### DCE-MRI

- Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI) parameters are measured at each individual joint (DIP Joints 2-5, PIP Joints 2-5, MCP Joints 1-5 and CMC-1) and consist of:
  - Exchange Rate (K<sup>trans</sup>)
  - Interstitial Volume (v<sub>e</sub>)
  - Plasma Volume (v<sub>p</sub>)
  - Initial Rate of Enhancement (IRE)
  - Maximum signal intensity enhancement (ME).
- All DCE-MRI parameters will be presented as a total measure over all joints at each time point.
- DCE-MRI Parameters will be calculated as:

$$\frac{\sum_{all\ joints} Parameter}{Number\ of\ Joints}$$

- All DCE-MRI Parameters will also be presented normalised by the Volume of Enhancing Pannus (VEP).
- Normalised DCE-MRI parameters will be calculated as:

### **Imaging**

$$\frac{\sum_{all\ joints}(VEP*Parameter)}{\sum_{all\ joints}VEP}$$

 All parameters will be presented as a total measure for the affected/dominant hand at each time point.

### **Bone Shape Parameters**

- Surface Area of the Bone:
  - Measured as the whole bone area (in mm²). At the metacarpals, the joint of interest is the MCP and therefore the distal part (15mm length from the joint) shall be measured.
  - o The following bones will be considered:
    - D2-5
    - 12-5
    - M2-5
    - P2-5
    - Trapezium
- All bone shape parameters will be presented as a total measure for the affected/dominant hand which is calculated by summing the individual measure for each bone at each time point.

# 12.6.6. Biomarker

# 12.6.6.1. Pharmacodynamic Biomarkers

| Test Analyte | LBCAT | LBTESTCD | Units | Derived | Details |
|---|---|---|---|---|---|
| Target Engagement | | | | | |
| Free Soluble GM-CSF | BIOMARKER | GMCSFFS | ng/L | | |
| GM-CSF: drug complex | BIOMARKER | GMCSFC | ng/L | | |
| <b>Predictive Biomarkers</b> | | | | | |
| HSCRP | CHEMISTRY | CRP | mg/L | | |
| MRP8/14 COMPLEX | BIOMARKER | S100A8A9 | mg/L | | |
| CCL17 (TARC) | BIOMARKER | CCL17 | ng/L | | |
| 14-3-3η | BIOMARKER | ETA1433 | mg/L | | |
| MMP-3 | BIOMARKER | MMP3 | μg/L | | |
| CXCL13 (BLC) | BIOMARKER | CXCL13 | ng/L | | |
| SAA | BIOMARKER | AMYLOIDA | ng/L | | |
| YKL-40 | BIOMARKER | CHI3L1 | μg/L | | |
| IL6 | BIOMARKER | INTLK6 | ng/L | | |
| CCL22 | BIOMARKER | MDC | ng/L | | |
| Cartilage Biomarkers | | | | | |
| ARGS Neoepitope | BIOMARKER | ARGSNEOE | | | |
| C1M | BIOMARKER | C1M | | | |
| C2M | BIOMARKER | C2M | | | |
| C3M | BIOMARKER | C3M | | | |
| CRPM | BIOMARKER | CRPM | | | |
| VICM | BIOMARKER | VICM | | | |
| Mechanistic Biomarkers | ; | | | | |
| VEGF | BIOMARKER | VEGF | ng/L | | |
| TNFa | BIOMARKER | TNF | ng/L | | |
| IL-1β | BIOMARKER | INTLK1B | ng/L | | |
| IL-8 | BIOMARKER | INTLK8 | ng/L | | |
| IL-10 | BIOMARKER | INTLK10 | ng/L | | |
| IL-13 | BIOMARKER | INTLK13 | ng/L | | |
| IL-4 | BIOMARKER | INTLK4 | ng/L | | |

| IFN-γ | BIOMARKER | IFNG | ng/L |
|-------|-----------|------|------|

#### 12.6.6.2. Safety Biomarkers

| Test Analyte | LBCAT | LBTESTCD | Units | Derived | Details |
|---------------------|-----------|----------|-------|---------|---------|
| Lung Damage | | | | | |
| Anti-GM-CSF auto AB | BIOMARKER | GMCSFAA | | | |

#### 12.6.6.3. Biomarker Derivations

#### **All Parameters**

# **Below Limit of Quantification**

- If a biomarker value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' (or indicated as less than x in the comment field) is present, the corresponding numeric value will be imputed using one half the lower limit of quantification.
- This value will be used in Summary Tables and Figures, but the original recorded result will be listed.

# 12.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

# 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| <b>Element</b> General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Early withdrawal (EW) visits will be assigned to the respective visit according to the Time and Events table in Section 12.2, using the day of the EW visit relative to Day 1.</li> <li>For the first 4 weeks an EW visit more than ±3 days in comparison to the target visit will be assigned to the closest target visit. Starting at Week 4, an EW visit more than 7 days after target visit day will be assigned to the next visit.</li> <li>If a scheduled visit and an EW visit occur within the same visit window and are both available, the later visit will be used for any summaries/analyses. The earlier visit will appear in listing only.</li> <li>For efficacy analyses, if an EW visit is assigned to a non-standard efficacy</li> </ul> |

# 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered</li> </ul> |
| | to be missing data and should be displayed as such. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 12.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: Missing Start Days First of the greath will be used upleas this is before the |
| | <ul> <li>Missing Start Day: First of the month will be used unless this is before the<br/>start date of study treatment; in this case the study treatment start date will<br/>be used and hence the event is considered On-treatment as per Appendix<br/>4: Treatment States and Phases.</li> </ul> |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the<br/>stop date of study treatment; in this case the study treatment stop date will<br/>be used.</li> </ul> |
| | <ul> <li>Completely missing start or end dates will remain missing, with no imputation<br/>applied. Consequently, time to onset and duration of such events will be<br/>missing.</li> </ul> |
| | <ul> <li>Start or end dates which are completely missing (i.e. no year specified) will<br/>remain missing, with no imputation applied.</li> </ul> |
| Concomitant<br>Medications/ | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| Medical<br>History | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 12.7.2.2. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| NRI | Subjects with missing pain NRS scores will be considered as non-responders for the purpose of analyses on the binary endpoints. |
| Change<br>from<br>Baseline | For any analysis on change from baseline values, if the baseline value is missing then all following assessment values are excluded from the analysis. |

# 12.7.2.3. Handling of Endpoint Specific Missing Data

| Element | Reporting Detail |
|---|---|
| NRS score | <ul> <li>If a subject records their daily pain NRS scores for less than 4 days out of the 7 days prior to assessment visit, then the average NRS score for the week prior to the assessment visit will be recorded as missing.</li> <li>For the purpose of the analyses on the continuous endpoints, no imputations for the missing data will be done.</li> </ul> |
| | For the purpose of the analyses on the binary endpoints, subjects with missing NRS scores will be considered as non-responders. |
| AUSCAN™ | <ul> <li>If ≥2 pain, the stiffness item or &gt;2 physical function items are missing, the subject's response on the affected subscale will be regarded as invalid and the deficient subscale(s) will not be used in any analysis.</li> <li>Where 1 pain or 1-2 physical function items are missing, the average value for the subscale will be substituted in lieu of the missing item value(s).</li> <li>Where any individual component score is missing, total score will be set to missing.</li> <li>No imputation for missing total individual component scores will be done.</li> </ul> |
| Swollen Hand<br>Joint Count | <ul> <li>If there are missing observations for swollen joints then the remaining observations will be assessed and weighted by dividing the number presented by the number of non-missing, and by multiplying by 30 for the joint count.</li> <li>No imputations for individual joints will be done.</li> <li>If a joint is not evaluable at Baseline, then that joint is set to missing throughout the study.</li> <li>If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.</li> </ul> |
| Tender Hand<br>Joint Count | <ul> <li>If there are missing observations for tender joints then the remaining observations will be assessed and weighted by dividing the number presented by the number of non-missing, and by multiplying by 30 for the joint count.</li> <li>No imputations for individual joints will be done.</li> <li>If a joint is not evaluable at Baseline, then that joint is set to missing throughout the study.</li> <li>If data for more than 50% of the joints are missing at the time of a given assessment, then the total count will be set to missing for that visit.</li> </ul> |
| PtGA | No imputations for missing data will be done. |
| PhGA | No imputations for missing data will be done. |

| Element | Reporting Detail |
|---|---|
| HOAMRIS | <ul> <li>If an individual joint has a missing score, then the score will be imputed using the average score across all available evaluable joints for each individual component.</li> <li>If data for more than 50% of locations are missing at the time of a given assessment, then the total individual component score will be set to missing for that visit. This threshold may be altered after review of the actual raw data.</li> </ul> |
| | <ul> <li>No imputation for missing total individual component scores will be done.</li> </ul> |
| HOAMRIQ | <ul> <li>If an individual joint has a missing value, then the value will be imputed using the average score across all available evaluable joints for each individual component.</li> <li>If data for more than 50% of locations are missing at the time of a given assessment, then the total individual component score will be set to missing for that visit. This threshold may be altered after review of the actual raw data.</li> <li>No imputation for missing total individual component values will be done.</li> </ul> |
| DCE-MRI | <ul> <li>If an individual joint has a missing value, then the value will be imputed using the average score across all available evaluable joints for each individual component.</li> <li>If data for more than 50% of locations are missing at the time of a given assessment, then the total individual component score will be set to missing for that visit. This threshold may be altered after review of the actual raw data.</li> <li>No imputation for missing total individual component values will be done.</li> </ul> |

# 12.8. Appendix 8: Values of Potential Clinical Importance

# 12.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) High Flag (>x) | |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) High Flag (>x | |
| Albumin | mmol/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | mmol/L | $\Delta$ from BL | | <b>↑ 44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 8.0 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

# 12.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------|-------|------------------------|-------|
| | | Lower Upper | |
| Absolute | | | |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Increase from Baseline QTc | msec | | >60 |

# 12.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |
### 12.9. Appendix 9: Multicenter Studies

There are no planned adjustments for multiple centres or regions. For all analyses, all sites, countries and regions will be pooled.

### 12.10. Appendix 10: Multiple Comparisons & Multiplicity

### 12.10.1. Handling of Multiple Comparisons & Multiplicity

In this phase IIa study, no adjustments will be made for multiple comparisons or multiplicity.

## 12.11. Appendix 11: Model Checking and Diagnostics for Statistical Analyses

#### 12.11.1. Statistical Analysis Assumptions

#### 12.11.1.1. Continuous Endpoints

| Endpoint(s) | • | Continuous Endpoints as described in Section 8.1.2.1. |
|-------------|---|-------------------------------------------------------|
| Analysis | • | MMRM |

- For the MMRM, model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as spatial power, CS or AR(1).
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### 12.11.1.2. Binary Endpoints

| Endpoint(s) | • | Binary Endpoints as described in Section 8.1.2.2 |
|-------------|---|--------------------------------------------------|
| Analysis | • | Generalised Estimating Equations (GEE) |

- For the GEE analyses, model assumptions will be applied, but appropriate adjustments may be made based on the data.
- An unstructured working correlation structure will be assumed and standard errors will be calculated based on the empirical sandwich covariance estimate (default setting for PROC GENMOD in SAS)
- An unstructured correlation structure will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as Independent, CS or AR(1).
  - Quasilikelihood under the Independence Model Criteria (QIC) will be used to assist with the selection of covariance structure.

### 12.12. Appendix 12: Definitions of some Parameters of Interest

### 12.12.1. Laboratory Parameters of Interest

| Lab parameters of interest | Grade | | | |
|---|---|---|---|---|
| or interest | 1 | 2 | 3 | 4 |
| HEMOGLOBIN decrease | Hemoglobin (Hgb) <lln -="" 10.0="" dl;<br="" g=""><lln -="" 100="" 6.2="" <lln="" g="" l;="" l<="" mmol="" th=""><th>Hgb &lt;10.0 - 8.0 g/dL; &lt;6.2 - 4.9<br/>mmol/L; &lt;100 - 80g/L</th><th>Hgb &lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</th><th>Life-threatening consequences; urgent intervention indicated</th></lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9<br>mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated |
| WHITE CELL<br>COUNT decrease | <lln -="" 3.0="" 3000="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <3000 - 2000/mm3; <3.0 - 2.0 x<br>10e9 /L | <2000 - 1000/mm3; <2.0 - 1.0 x<br>10e9 /L | <1000/mm3; <1.0 x<br>10e9 /L |
| TOTAL NEUTROPHILS ABSOLUTE COUNT | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x<br>10e9 /L |
| LYMPHOCYTES ABSOLUTE COUNT decreased | <lln -="" 0.8="" 10e9="" 800="" <lln="" l<="" mm3;="" td="" x=""><td>&lt;800 - 500/mm3; &lt;0.8 - 0.5 x<br/>10e9 /L</td><td>&lt;500 - 200/mm3; &lt;0.5 - 0.2 x<br/>10e9 /L</td><td>&lt;200/mm3; &lt;0.2 x<br/>10e9 /L</td></lln> | <800 - 500/mm3; <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x<br>10e9 /L |
| LYMPHOCYTES<br>ABSOLUTE<br>increased | | >4000/mm3 - 20,000/mm3 ; >4-20<br>x 10e9 /L | >20,000/mm3; >20 x 10e9 /L | |
| PLATELET<br>COUNT | <lln -="" 75,000="" 75.0="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <75,000 - 50,000/mm3; <75.0 -<br>50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0 - 25.0 x 10e9 /L | <25,000/mm3; <25.0 x<br>10e9 /L |
| CREATININE | >1 - 1.5 x baseline; >ULN - 1.5 x<br>ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN |


#### 

| SODIUM | | | | |
|---|---|---|---|---|
| decrease | <lln -="" 130="" l<="" mmol="" td=""><td></td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L;</td></lln> | | <130 - 120 mmol/L | <120 mmol/L; |
| SODIUM increase | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| POTASSIUM | | | | |
| decrease | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln></td></lln> | <lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | <3.0 - 2.5 mmol/L | <2.5 mmol/L |
| POTASSIUM | | | | |
| increase | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L | >7.0 mmol/L |
| CALCIUM | >ULN - 11.5 mg/dL; >ULN - 2.9 | >11.5 - 12.5 mg/dL; >2.9 - 3.1 | >12.5 - 13.5 mg/dL; >3.1 - 3.4 | >13.5 mg/dL; >3.4 |
| increase | mmol/L | mmol/L | mmol/L; | mmol/L |
| CALCIUM | | | | |
| decrease | <lln -="" 1.0="" l<="" mmol="" td=""><td>&lt;1.0 - 0.9 mmol/L</td><td>&lt;0.9 - 0.8 mmol/L</td><td>&lt;0.8 mmol/L</td></lln> | <1.0 - 0.9 mmol/L | <0.9 - 0.8 mmol/L | <0.8 mmol/L |
| ASAT (SGOT) | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALAT (SGPT) | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALKALINE | | | | |
| PHOSPHATASE | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| BILIRUBIN, | | | | |
| TOTAL | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| ALBUMIN | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL; &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td></td></lln> | <3 - 2 g/dL; <30 - 20 g/L | <2 g/dL; <20 g/L | |
| GLUCOSE | >ULN -160 mg/dL; >ULN - 8.9 mmol/L | >160 -250 mg/dL; >8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8 | >500 mg/dL; >27.8<br>mmol/L |
| EST.CREATININ | - | | | |
| E CLEARANCE | <lln -="" 1.73="" 60="" m2<="" ml="" s="" td=""><td>59 - 30 ml/s/1.73 m2</td><td>29 - 15 ml/s/1.73 m2</td><td>&lt;15 ml/s/1.73 m2</td></lln> | 59 - 30 ml/s/1.73 m2 | 29 - 15 ml/s/1.73 m2 | <15 ml/s/1.73 m2 |

# 12.13. Appendix 13: Opportunistic Infections: MedDRA Preferred Terms

### 12.13.1. Opportunistic Infections: MedDRA Preferred Terms

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| AIDS retinopathy | Herpes pharyngitis |
| Acid fast bacilli infection | Herpes sepsis |
| Acinetobacter bacteraemia | Herpes simplex |
| Acinetobacter infection | Herpes simplex cervicitis |
| Acquired immunodeficiency syndrome | Herpes simplex hepatitis |
| Actinomycosis | Herpes simplex meningoencephalitis |
| Actinomycotic abdominal infection | Herpes simplex otitis externa |
| Actinomycotic pulmonary infection | Herpes simplex test positive |
| Acute HIV infection | Herpes simplex virus conjunctivitis neonatal |
| Acute hepatitis B | Herpes simplex visceral |
| Acute hepatitis C | Herpes virus infection |
| Adrenal gland tuberculosis | Herpes zoster |
| Arthritis fungal | Herpes zoster cutaneous disseminated |
| Arthritis salmonella | Herpes zoster disseminated |
| Aspergilloma | Herpes zoster infection neurological |
| Aspergillosis oral | Herpes zoster meningitis |
| Aspergillus infection | Herpes zoster meningoencephalitis |
| Asymptomatic HIV infection | Herpes zoster meningomyelitis |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Asymptomatic viral hepatitis | Herpes zoster necrotising retinopathy |
| Atypical mycobacterial infection | Herpes zoster oticus |
| Atypical mycobacterial lower respiratory tract infection | Herpes zoster pharyngitis |
| Atypical mycobacterial lymphadenitis | Histoplasmosis |
| Atypical mycobacterial pneumonia | Histoplasmosis cutaneous |
| Atypical mycobacterium pericarditis | Histoplasmosis disseminated |
| Bacterial parotitis | Human T-cell lymphocytic virus type II infection |
| BK virus infection | Human T-cell lymphotropic virus infection |
| Biliary tract infection cryptosporidial | Human T-cell lymphotropic virus type I infection |
| Biliary tract infection fungal | Human polyomavirus infection |
| Blastomycosis | Immune reconstitution inflammatory syndrome associated tuberculosis |
| Bone tuberculosis | Intestinal tuberculosis |
| Brachyspira infection | JC virus granule cell neuronopathy |
| Brain empyema | JC virus infection |
| Bronchitis fungal | Joint tuberculosis |
| Bronchopulmonary aspergillosis | Kaposi's sarcoma |
| Bronchopulmonary aspergillosis allergic | Kaposi's sarcoma AIDS related |
| Brucella sepsis | Kaposi's varicelliform eruption |
| Brucellosis | Leptotrichia infection |
| Candida endophthalmitis | Listeria encephalitis |
| Candida infection | Listeria sepsis |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Candida osteomyelitis | Listeriosis |
| Candida pneumonia | Lower respiratory tract herpes infection |
| Candida retinitis | Lower respiratory tract infection fungal |
| Candida sepsis | Lymph node tuberculosis |
| Cerebral aspergillosis | Lymphadenitis fungal |
| Cerebral fungal infection | Lymphoma AIDS related |
| Cerebral toxoplasmosis | Male genital tract tuberculosis |
| Choroid tubercles | Meningitis aspergillus |
| Chronic hepatitis | Meningitis candida |
| Chronic hepatitis C | Meningitis coccidioides |
| Coccidioides encephalitis | Meningitis cryptococcal |
| Coccidioidomycosis | Meningitis fungal |
| Colitis herpes | Meningitis herpes |
| Congenital HIV infection | Meningitis histoplasma |
| Congenital cytomegalovirus infection | Meningitis listeria |
| Congenital hepatitis B infection | Meningitis salmonella |
| Congenital herpes simplex infection | Meningitis toxoplasmal |
| Congenital toxoplasmosis | Meningitis tuberculous |
| Congenital tuberculosis | Meningoencephalitis herpes simplex neonatal |
| Congenital varicella infection | Meningoencephalitis herpetic |
| Conjunctivitis tuberculous | Minor cognitive motor disorder |
| Corynebacterium infection | Mucocutaneous candidiasis |
| Corynebacterium sepsis | Mycobacterial infection |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Cryptococcal cutaneous infection | Mycobacterium abscessus infection |
| Cryptococcal fungaemia | Mycobacterium avium complex immune restoration disease |
| Cryptococcosis | Mycobacterium avium complex infection |
| Cryptosporidiosis infection | Mycobacterium chelonae infection |
| Cutaneous coccidioidomycosis | Mycobacterium fortuitum infection |
| Cutaneous tuberculosis | Mycobacterium kansasii infection |
| Cytomegalovirus chorioretinitis | Mycobacterium marinum infection |
| Cytomegalovirus colitis | Mycobacterium ulcerans infection |
| Cytomegalovirus duodenitis | Mycotic endophthalmitis |
| Cytomegalovirus enteritis | Mycotoxicosis |
| Cytomegalovirus enterocolitis | Myocarditis mycotic |
| Cytomegalovirus gastritis | Myocarditis toxoplasmal |
| Cytomegalovirus gastroenteritis | Nasal herpes |
| Cytomegalovirus gastrointestinal infection | Necrotising fasciitis fungal |
| Cytomegalovirus gastrointestinal ulcer | Necrotising herpetic retinopathy |
| Cytomegalovirus infection | Neonatal candida infection |
| Cytomegalovirus mononucleosis | Neonatal mucocutaneous herpes simplex |
| Cytomegalovirus mucocutaneous ulcer | Neurocryptococcosis |
| Cytomegalovirus myelomeningoradiculitis | Neutropenic sepsis |
| Cytomegalovirus myocarditis | Nocardia sepsis |
| Cytomegalovirus oesophagitis | Nocardiosis |
| Cytomegalovirus pancreatitis | Oesophageal candidiasis |
| Cytomegalovirus pericarditis | Oesophageal tuberculosis |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Cytomegalovirus syndrome | Ophthalmic herpes simplex |
| Cytomegalovirus urinary tract infection | Ophthalmic herpes zoster |
| Cytomegalovirus viraemia | Oro-pharyngeal aspergillosis |
| Disseminated cryptococcosis | Oropharyngeal candidiasis |
| Disseminated cytomegaloviral infection | Osteomyelitis blastomyces |
| Disseminated tuberculosis | Osteomyelitis fungal |
| Ear tuberculosis | Osteomyelitis salmonella |
| Eczema herpeticum | Overgrowth fungal |
| Encephalitis cytomegalovirus | Pancreatitis fungal |
| Encephalitis fungal | Paratyphoid fever |
| Encephalitis post immunisation | Pericarditis fungal |
| Encephalitis post varicella | Pericarditis histoplasma |
| End stage AIDS | Pericarditis tuberculous |
| Endocarditis candida | Perinatal HIV infection |
| Endocarditis histoplasma | Peritoneal candidiasis |
| Enterocolitis AIDS | Peritoneal tuberculosis |
| Enterocolitis fungal | Persistent generalised lymphadenopathy |
| Epididymitis blastomyces | Pneumocystis jirovecii infection |
| Epididymitis tuberculous | Pneumocystis jirovecii pneumonia |
| Epstein-Barr virus associated lymphoma | Pneumonia blastomyces |
| Erythema induratum | Pneumonia cytomegaloviral |
| Erythrasma | Pneumonia fungal |
| Exanthema subitum | Pneumonia herpes viral |
| Extrapulmonary tuberculosis | Pneumonia salmonella |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Eye infection toxoplasmal | Pneumonia toxoplasmal |
| Female genital tract tuberculosis | Polyomavirus-associated nephropathy |
| Fungaemia | Presumed ocular histoplasmosis syndrome |
| Fungal abscess central nervous system | Proctitis herpes |
| Fungal endocarditis | Proctitis monilial |
| Fungal infection | Progressive multifocal leukoencephalopathy |
| Fungal oesophagitis | Prostatitis tuberculous |
| Fungal peritonitis | Pulmonary mycosis |
| Fungal sepsis | Pulmonary trichosporonosis |
| Fungal tracheitis | Pulmonary tuberculoma |
| Funguria | Pulmonary tuberculosis |
| Gastritis fungal | Pyelonephritis fungal |
| Gastritis herpes | Renal tuberculosis |
| Gastroenteritis cryptococcal | Respiratory moniliasis |
| Gastroenteritis cryptosporidial | Respiratory tract infection fungal |
| Gastrointestinal candidiasis | Retinitis histoplasma |
| Gastrointestinal fungal infection | Retroviral infection |
| Genital blister | Retroviral rebound syndrome |
| Genital herpes | Salmonella bacteraemia |
| Genital herpes zoster | Salmonella sepsis |
| Haemorrhagic pneumonia | Salmonellosis |
| Hepatosplenic abscess | Salpingitis tuberculous |
| HIV associated nephropathy | Silicotuberculosis |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| HIV cardiomyopathy | Sinusitis aspergillus |
| HIV enteropathy | Skin candida |
| HIV infection | Spleen tuberculosis |
| HIV infection CDC Group I | Splenic candidiasis |
| HIV infection CDC Group II | Splenic infection fungal |
| HIV infection CDC Group III | Stoma site candida |
| HIV infection CDC Group IV subgroup A | Stoma site infection |
| HIV infection CDC Group IV subgroup B | Superinfection fungal |
| HIV infection CDC Group IV subgroup C1 | Superinfection mycobacterial |
| HIV infection CDC Group IV subgroup C2 | Systemic candida |
| HIV infection CDC Group IV subgroup D | Systemic mycosis |
| HIV infection CDC Group IV subgroup E | T-cell lymphoma |
| HIV infection CDC category A | T-cell type acute leukaemia |
| HIV infection CDC category B | Thyroid tuberculosis |
| HIV infection CDC category C | Tongue fungal infection |
| HIV infection CDC group IV | Toxoplasmosis |
| HIV infection WHO clinical stage I | Tropical spastic paresis |
| HIV infection WHO clinical stage II | Tuberculoma of central nervous system |
| HIV infection WHO clinical stage III | Tuberculosis |
| HIV infection WHO clinical stage IV | Tuberculosis bladder |
| HIV peripheral neuropathy | Tuberculosis gastrointestinal |
| HIV wasting syndrome | Tuberculosis liver |
| Hepatic candidiasis | Tuberculosis of central nervous system |
| Hepatic infection fungal | Tuberculosis of eye |

| Opportunistic Infections: MedDRA Preferred Terms | |
|---|---|
| Hepatitis B | Tuberculosis of genitourinary system |
| Hepatitis C | Tuberculosis of intrathoracic lymph nodes |
| Hepatitis chronic persistent | Tuberculosis of peripheral lymph nodes |
| Hepatitis fulminant | Tuberculosis ureter |
| Hepatitis toxoplasmal | Tuberculous abscess central nervous system |
| Hepatitis viral | Tuberculous endometritis |
| Hepatitis virus-associated nephropathy | Tuberculous laryngitis |
| Hepatosplenic candidiasis | Tuberculous pleurisy |
| Herpes dermatitis | Tuberculous tenosynovitis |
| Herpes oesophagitis | Typhoid fever |
| Herpes ophthalmic | Varicella keratitis |

### 12.14. Appendix 14 – Abbreviations & Trade Marks

### 12.14.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| AUC | Area under the curve |
| AUSCAN | Australian Canadian Hand Osteoarthritis Index |
| Cave | Average steady state concentration during dosing interval |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL | Clearance |
| CL/F | Total body clearance from plasma after SC administration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRF | Case Report Form |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| D <sub>LCO</sub> | Diffusing capacity of the lung for carbon monoxide |
| DCE-MRI | Dynamic Contrast Enhanced Magnetic Resonance Imaging |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Report Form |
| ECG | Electrocardiogram |
| FEV1 | Forced Expiratory Volume in one Second |
| FVC | Forced Vital Capacity |
| GM-CSF | Granulocyte-macrophage colony stimulating factor |
| GUI | Guidance |
| GSK | GlaxoSmithKline |
| Н | Hour |
| HIV | Human Immunodeficiency Virus |
| HOA | Hand Osteoarthritis |
| HOAMRIS | Hand Osteoarthritis Magnetic Resonance Imaging Scoring System |
| HOAMRIQ | Hand Osteoarthritis Magnetic Resonance Imaging Quantitative score |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| Ig | Immunoglobulin |
| IMMS | International Modules Management System |

| Abbreviation | Description |
|---|---|
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| Ka | Absorption rate constant |
| Kg | Kilogram |
| K <sup>trans</sup> | Exchange rate |
| L | Litre |
| MDL | Medicines Development Lead |
| MDT | Medicines Development Team |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Mg | Milligram |
| mL | Milliliter |
| MMRM | Mixed Model Repeated Measures |
| MRI | Magnetic Resonance Imaging |
| NRI | Non-responder Imputation |
| NRS | Numerical Rating Scale |
| OA | Osteoarthritis |
| OMERACT | Outcome measures in Rheumatology |
| PAP | Pulmonary alveolar proteinosis |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PhGA | Physician's Global Assessment |
| PtGA | Patient's Global Assessment |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PRO | Patient reported outcome |
| QC | Quality Control |
| QTc | Corrected QT interval |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAMOS | Randomization & Medication Ordering System |
| RAMRIS | Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious adverse event |
| SC | Subcutaneous |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| t ½ | Elimination half life |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Ve | Interstitial volume |
| Vp | Plasma volume |
| V <sub>ss</sub> /F | Total volume of distribution after SC administration |

### 12.14.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| NONE | WinNonlin |
| | SAS |
| | AUSCAN |

#### 12.15. Appendix 15: List of Data Displays

### 12.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|--------------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic | 4.1 to 4.n | 4.1 to 4.n |
| Pharmacodynamic and / or Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Pharmacokinetic / Pharmacodynamic | 6.1 to 6.n | 6.1 to 6.n |
| Section | List | ings |
| ICH Listings | CH Listings 1 to x | |
| Other Listings | y t | 0 Z |

#### 12.15.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------------|---------|---------|----------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and / or Biomarker | PD_Fn | PD_Tn | PD_Ln |
| Pharmacokinetic / Pharmacodynamic | PKPD_Fn | PKPD_Tn | PK/PD_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 12.15.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|----------------------------------------------|
| PK IA [X] | PK Interim Statistical Analysis Complete |
| Wk6 IA [X] | Week 6 Interim Statistical Analysis Complete |
| AIR [X] | Administrative Interim Review Complete |
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

### 12.15.4. Study Population Tables

| Study Po | pulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject I | Disposition | | | | |
| 1.1. | ITT | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | Journal Requirements Add footnote: For rescreened subjects, the earlier screening is not included. Subjects who got rescreened successfully are not seen as subjects with screening failures. | SAC |
| 1.4. | Enrolled | NS1 | Summary of Number of Subjects by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protocol | Deviation | | | | |
| 1.5. | ITT | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Population | on Analysed | | | | |
| 1.6. | Screened | SP1 | Summary of Study Populations | IDSL | SAC |
| Demogra | aphic and Bas | seline Characteris | tics | | |
| 1.7. | ITT | DM1 | Summary of Demographic Characteristics | ICH E3, GSK CTR, FDAAA, EudraCT Programming note: Include smoking history | Wk6 IA, SAC |
| 1.8. | ITT | Non Standard<br>POP_T1 | Summary of Baseline Efficacy Parameters | Include all Efficacy Parameters | SAC |
| 1.9. | ITT | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, , GSK CTR, FDAAA,<br>EudraCT | SAC |

| Study Po | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.10. | ITT | Non Standard<br>POP_T2 | Summary of Hand OA Disease History | | SAC |
| Medical | condition & C | oncomitant Medi | cations | | |
| 1.11. | ITT | Non Standard<br>POP_T3 | Summary of Current Medical Conditions | ICH E3 | SAC |
| 1.12. | ITT | CM1 | Summary of Concomitant Medication | ICH E3 | SAC |
| 1.13. | ITT | CM1 | Summary of Concomitant OA Medication | | SAC |
| 1.14. | ITT | CM1 | Summary of Prior Medication | | SAC |
| 1.15. | ITT | CM1 | Summary of Prior OA Medication | | SAC |
| Exposur | e and Treatm | ent Compliance | | | |
| 1.16. | Safety | EX1 | Summary of Exposure to Study Treatment | ICH E3 Rows include: - Duration of Drug Exposure (Days) - Number of Injections - Volume of Doses Received (ml) Footnote 'Note: Exposure includes 13 days after the last injection.' | SAC |

### 12.15.5. Efficacy Tables

| Efficacy: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24h avera | age hand pain N | IRS score | | | <u>.</u> |
| 2.1. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in 24h average hand pain NRS Averaged over 7 days Prior to Each Visit | | AIR, Wk6 IA,<br>SAC |
| 2.2. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in 24h average hand pain NRS Averaged over 7 days Prior to Each Visit | | AIR, Wk6 IA,<br>SAC |
| 24h wors | t hand pain NR | S score | | | · |
| 2.3. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in 24h worst hand pain NRS Averaged over 7 days Prior to Each Visit | | AIR, Wk6 IA,<br>SAC |
| 2.4. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in 24h worst hand pain NRS Averaged over 7 days Prior to Each Visit | | AIR, Wk6 IA,<br>SAC |
| Proportio | on of subjects w | vith percentage re | duction in 24h average hand pain NRS | | <u>.</u> |
| 2.5. | ITT | Non Standard<br>EFF_T3 | Summary and Analysis of the Proportion of Subjects Achieving a 30% or More Reduction in 24h average hand pain NRS Averaged over 7 days Prior to Each Visit | | SAC |
| 2.6. | ITT | Non Standard<br>EFF_T3 | Summary and Analysis of the Proportion of Subjects Achieving a 50% or More Reduction in 24h average hand pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | | SAC |
| Proportio | on of subjects w | vith percentage re | duction in 24h worst hand pain NRS | | |
| 2.7. | ITT | Non Standard<br>EFF_T3 | Summary and Analysis of the Proportion of Subjects Achieving a 30% or More Reduction in 24h worst hand pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | | SAC |

| Efficacy: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | ITT | Non Standard<br>EFF_T3 | Summary and Analysis of the Proportion of Subjects Achieving a 50% or More Reduction in 24h worst hand pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | | SAC |
| AUSCAN | 3.1 NRS | | | | |
| 2.9. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in AUSCAN 3.1 NRS Individual Components Scores, at Each Visit | Include: AUSCAN Pain, AUSCAN Physical Function, AUSCAN Stiffness, AUSCAN Total Note: Page by Component. | Wk6 IA, SAC |
| 2.10. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in AUSCAN 3.1 NRS Individual Components Scores | Include: AUSCAN Pain, AUSCAN Physical Function, AUSCAN Stiffness, AUSCAN Total Note: Page by Component. | Wk6 IA, SAC |
| Joint Ass | essments | | | , | |
| 2.11. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in the Number of Soft Tissue Swollen Hand Joints, at Each Visit | | SAC |
| 2.12. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in the Number of Soft Tissue Swollen Hand Joints | | SAC |
| 2.13. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in the Number of Tender Hand Joints, at Each Visit | | SAC |
| 2.14. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in the Number of Tender Hand Joints | | SAC |
| Disease G | Slobal Assessn | nent | | | |
| 2.16. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in the Physician's Global Assessment (NRS 0-10), at Each Visit | | SAC |

| Efficacy: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.17. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in the Physician's Global Assessment (NRS 0-10) | | SAC |
| 2.18. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in the Patients' Global Assessment (NRS 0-10), at Each Visit | | SAC |
| 2.19. | ITT | Non Standard<br>EFF_T2 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in the Patients' Global Assessment (NRS 0-10) | | SAC |
| Imaging | | | | | |
| 2.20. | ITT | Non Standard<br>EFF_T4 | Summary of Observed Result and Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS | Individual Components Include: Synovitis, Erosive damage, Cyst, Osteophyte Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions | SAC |
| 2.21. | ITT | Non Standard<br>EFF_T5 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS | Individual Components Include: Synovitis, Erosive damage, Cyst, Osteophyte Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions | SAC |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 2.22. | ITT | Non Standard<br>EFF_T4 | Summary of Observed Result and Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIQ | <ul> <li>Individual Components Include synovitis, normalised synovitis, normalised erosive damage, cartilage space loss, malalignment and normalised bone marrow lesions.</li> <li>Add footnote 'Note: Synovitis is normalised by the total joint volume, erosive damage and bone marrow lesions are normalised by volume of bone.'</li> </ul> | SAC |
| 2.23. | ІТТ | Non Standard<br>EFF_T5 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIQ | <ul> <li>Individual Components Include synovitis, normalised synovitis, normalised erosive damage, cartilage space loss, malalignment and normalised bone marrow lesions.</li> <li>Add footnote 'Note: Synovitis is normalised by the total joint volume, erosive damage and bone marrow lesions are normalised by volume of bone.'</li> </ul> | SAC |

| Efficacy: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.24. | ITT | Non Standard<br>EFF_T4 | Summary of Observed Result and Change from Baseline in Joint Inflammation: DCE-MRI | <ul> <li>Includes ktrans, normalised Ktrans, VE, normalised VE, VP, normalised VP, IRE, normalised IRE, ME, normalised ME.</li> <li>Add Footnote: 'Note: All normalised parameters have been normalised using the Volume of Enhancing Pannus (VEP).'</li> <li>Add units to parameter line.</li> </ul> | SAC |
| 2.25. | ITT | Non Standard<br>EFF_T5 | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Joint Inflammation: DCE-MRI | Includes ktrans, normalised Ktrans, VE, normalised VE, VP, normalised VP, IRE, normalised IRE, ME, normalised ME. Add Footnote: 'Note: All normalised parameters have been normalised using the Volume of Enhancing Pannus (VEP).' Add units to parameter line. | SAC |
| 2.26. | ITT | Non Standard<br>EFF_T4 | Summary of Observed Result and Change from Baseline in Bone Shape Parameters | Includes Surface Area of Bone | SAC |
| Paraceta | mol | | | <u> </u> | |
| 2.27. | ITT | Non Standard<br>EFF_T1 | Summary of Observed Result and Change from Baseline in 24h Total Dosage of Paracetamol Averaged over 7 days Prior to Each Visit | | SAC |
| 2.28. | ITT | Non Standard<br>EFF_T6 | Summary of the Proportion of Subjects Reporting Paracetamol Use in the 7 days Prior to Each Visit | | AIR, SAC |

### 12.15.6. Efficacy Figures

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 24h ave | erage hand pai | n NRS score | | | |
| 2.1. | ITT | Non Standard<br>EFF_F1 | Individual Subject Profile Plots of 24h Average Hand Pain NRS Averaged Over 7 Days Prior to Each Visit, by Treatment Group | X-Axis : Visit : Continuous Scale<br>Y-Axis : Parameter (Unit) scaled<br>accordingly<br>Legend: no legend to be displayed | SAC |
| 2.3 | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in 24h<br>Average Hand Pain NRS Averaged over 7 days Prior to Each<br>Visit | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly | AIR, Wk6 IA,<br>SAC |
| 2.4. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in 24h Average Hand Pain NRS Averaged over 7 days Prior to Each Visit (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | AIR, Wk6 IA,<br>SAC |
| 24h wo | rst hand pain I | NRS score | | | |
| 2.5. | ITT | Non Standard<br>EFF_F1 | Individual Subject Profile Plots of 24h Worst Hand Pain NRS<br>Averaged over 7 days Prior to Each Visit, by Treatment Group | X-Axis : Visit : Continuous Scale<br>Y-Axis : Parameter (Unit) scaled<br>accordingly<br>Legend: no legend to be displayed | SAC |
| 2.6. | ITT | Non Standard<br>EFF_F1 | Individual Subject Profile Plots of Daily 24h Worst Hand Pain NRS, by Treatment Group | X-Axis: Day: Continuous Scale Y-Axis: Parameter (Unit) scaled accordingly Legend: no legend to be displayed | SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.7. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in 24h Worst Hand Pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | X-Axis : Visit<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | AIR, Wk6 IA,<br>SAC |
| 2.8. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in 24h worst hand pain NRS Averaged over 7 days Prior to Each Visit (from Repeated Measures Analysis), at Each Visit | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | AIR, Wk6 IA,<br>SAC |
| Propor | tion of subject | s with percentage | reduction in 24h average hand pain NRS | | |
| 2.9. | ІТТ | Non Standard<br>EFF_F2 | Proportion of Subjects in Each Treatment Group Achieving a 30% Reduction in 24h Average Hand Pain NRS Averaged over 7 days Prior to Each Visit | X-Axis: Visit Y-Axis: Proportion of Subjects (%) Note: Do not incude Cl's | SAC |
| 2.10. | ITT | Non Standard<br>EFF_F3 | Proportion of Subjects in Each Treatment Group Achieving a 50% Reduction in 24h Average Hand Pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | X-Axis: Visit Y-Axis: Proportion of Subjects (%) Note: Do not incude Cl's | SAC |
| Propor | tion of subject | s with percentage | reduction in 24h worst hand pain NRS | | |
| 2.11. | ITT | Non Standard<br>EFF_F3 | Proportion of Subjects in Each Treatment Group Achieving a 30% Reduction in 24h Worst Hand Pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | X-Axis: Visit Y-Axis: Proportion of Subjects (%) Note: Do not incude CI's | SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12. | ITT | Non Standard<br>EFF_F3 | Proportion of Subjects in Each Treatment Group Achieving a 50% Reduction in 24h Worst Hand Pain NRS Averaged over 7 days Prior to Each Visit, at Each Visit | X-Axis: Visit Y-Axis: Proportion of Subjects (%) Note: Do not incude Cl's | SAC |
| AUSCA | N 3.1 NRS | | | | l |
| 2.13. | ITT | Non Standard<br>EFF_F1 | Individual Subject Profile Plots of AUSCAN 3.1 NRS Individual Component Scores, by Treatment Group | X-Axis: Visit Y-Axis: Parameter (Unit) scaled accordingly Individual Components include: AUSCAN Pain, AUSCAN Physical Function, AUSCAN Stiffness, AUSCAN Total | SAC |
| 2.14. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in AUSCAN 3.1 NRS Individual Component Scores, at Each Visit | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Individual Components include: AUSCAN Pain, AUSCAN Physical Function, AUSCAN Stiffness, AUSCAN Total | Wk6 IA, SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | X-Axis : Visit<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | |
| 2.15. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in AUSCAN 3.1 NRS Individual Component Scores (from Repeated Measures Analysis) | Add footnote: 'Note: Repeated<br>Measures Analysis adjusted for<br>Baseline Value, Treatment Group,<br>Visit, Treatment Group by Visit<br>Interaction [and Baseline Value by Visit<br>Interaction]' | Wk6 IA, SAC |
| | | | | Individual Components include:<br>AUSCAN Pain, AUSCAN Physical<br>Function, AUSCAN Stiffness,<br>AUSCAN Total | |
| Joint A | ssessments | | | | |
| 2.16. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Number of Soft Tissue Swollen Hand Joints, at Each Visit | X-Axis : Visit Y-Axis : Change from Baseline in Parameter (Unit) scaled accordingly | SAC |
| 2.17. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in the Number of Soft Tissue Swollen Hand Joints (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Number of Tender Hand Joints, at Each Visit | X-Axis : Visit<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC |
| | | | | X-Axis : Visit Y-Axis : Change from Baseline in Parameter (Unit) scaled accordingly | |
| 2.19. | ІТТ | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in the Number of Tender Hand Joints (from Repeated Measures Analysis) | Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | SAC |
| Diseas | e Global Asses | sment | | | |
| 2.20. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Physician's Global Assessment (NRS 0-10), at Each Visit | X-Axis : Visit Y-Axis : Change from Baseline in Parameter (Unit) scaled accordingly | SAC |
| | | Non Standard EFF_F2 Plot of Least Squares Means and 95% CI of Change from Baseline in Physician's Global Assessment (NRS 0-10) (from Repeated Measures Analysis) | | X-Axis : Visit<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | |
| 2.21. | ITT | | Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | SAC | |
| 2.22. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Patients' Global Assessment, at Each Visit | X-Axis : Visit<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.23. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in Patients' Global Assessment (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | SAC |
| Imagin | g | | | | |
| 2.24. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Individual Components Include: Synovitis, Erosive damage, Cyst, Osteophyte Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.25. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Individual Components Include: Synovitis, Erosive damage, Cyst, Osteophyte Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | |
| 2.26. | ΙΤΤ | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIQ | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Individual Components Include: synovitis, normalised synovitis, normalised erosive damage, cartilage space loss, mal-alignment and normalised bone marrow lesions. Add footnote 'Note: Synovitis is normalised by the total joint volume, erosive damage and bone marrow lesions are normalised by volume of bone.' | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.27. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIQ (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Individual Components Include: synovitis, normalised synovitis, normalised erosive damage, cartilage space loss, mal-alignment and normalised bone marrow lesions. Add footnote 'Note: Synovitis is normalised by the total joint volume, erosive damage and bone marrow lesions are normalised by volume of bone.' Add footnote: 'Note: Repeated | [Priority] |
| | | | | bone.' | |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.28. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Joint Inflammation: DCE-MRI | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Includes ktrans, normalised Ktrans, VE, normalised VE, VP, normalised VP, IRE, normalised IRE, ME, normalised ME. Add Footnote: 'Note: All normalised parameters have been normalised using the Volume of Enhancing Pannus (VEP).' Add units to parameter line. | SAC |

| NI - | Damidati. | IDSL / TST ID / | T'd. | D Notes | Deliverable |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | [Priority] |
| 2.29. | ITT | Non Standard<br>EFF_F2 | Plot of Least Squares Means and 95% CI of Change from Baseline in Joint Inflammation: DCE-MRI (from Repeated Measures Analysis) | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Includes ktrans, normalised Ktrans, VE, normalised VE, VP, normalised VP, IRE, normalised IRE, ME, normalised ME. Add Footnote: 'Note: All normalised parameters have been normalised using the Volume of Enhancing Pannus (VEP).' Add units to parameter line. Add footnote: 'Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit, Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]' | SAC |
| 2.30. | ІТТ | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in Bone Shape Parameters | X-Axis: Visit Y-Axis: Change from Baseline in Parameter (Unit) scaled accordingly Includes Surface Area of Bone Add units to parameter line. | SAC |
| Efficac | Efficacy: Figures | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] | | | |
| 2.31. | ITT | Non Standard<br>EFF_F2 | Plot of Mean and 95% CI of Change from Baseline in 24h Total Dosage of Paracetamol Averaged over 7 days Prior to Each Visit | | AIR, SAC | | | |
| Additio | nal MRI | | | | | | | |
| 2.32. | ІТТ | Non Standard | Ordered Scatter Plot of Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS | X-Axis : Percentile<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC | | | |
| 2.33. | ІТТ | Non Standard | Ordered Scatter Plot of Change from Baseline in Inflammatory<br>Structural Joint Damage: HOAMRIQ | X-Axis : Percentile<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC | | | |
| 2.34. | ІТТ | Non Standard | Ordered Scatter Plot of Change from Baseline in Joint Inflammation: DEC-MRI | X-Axis : Percentile<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC | | | |
| 2.35. | ІТТ | Non Standard | Ordered Scatter Plot of Change from Baseline in Bone Shape Parameters | X-Axis : Percentile<br>Y-Axis : Change from Baseline in<br>Parameter (Unit) scaled accordingly | SAC | | | |

# 12.15.7. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | • |
| 3.1. | Safety | Non Standard<br>SAFE_T1 | Overall Summary of Adverse Events | | SAC |
| 3.2. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | Wk6 IA, SAC |
| 3.3. | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 | SAC |
| 3.4. | Safety | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | GSK CTR | Wk6 IA, SAC |
| 3.5. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC |
| Serious | s and Other Sig | gnificant Adverse | Events | | |
| 3.6. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | Wk 6 IA, SAC |
| 3.7. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL | Wk6 IA, SAC |
| 3.8. | Safety | Non Standard<br>SAFE_T2 | Summary of Adverse Events of Special Interest | Include any AESI, Serious Infections with subgroup of serious respiratory infections, Opportunistic Infections, PAP, Neutropenia, Hypersensitivity Reactions | SAC |
| 3.9. | Safety | Non Standard<br>SAFE_T3 | Summary of Adverse Events of Special Interest – Injection Site Reactions | | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | Safety | Non Standard<br>SAFE_T4 | Summary of Adverse Events of Special Interest – Systemic Hypersensitivity Reactions related to GSK3196165 | | SAC |
| Labora | tory | | | | |
| 3.11. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | ICH E3 | SAC |
| 3.12. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
| 3.13. | Safety | LB1 | Summary of Urinalysis Changes from Baseline | ICH E3 | SAC |
| 3.14. | Safety | Non Standard<br>SAFE_T6 | Summary of the Proportion of Subjects with Urinalysis Findings | | SAC |
| 3.15. | Safety | Non Standard<br>SAFE_T7 | Summary of Laboratory Parameters of Interest by CTCAE Grade | Note: Definitions of Grades can be found in and Laboratory Parameters of Interest can be found in Section 12.12.1. If multiple values are mapped to one visit: the value with the worst CTCAE grade will be considered. If there are more than one value of this grade, the later value will be considered. | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.16. | Safety | LB18 | Shift Table of Laboratory Parameters of Interest from Baseline to Worst CTCAE Grade | Note: Definitions of Grades can be found in and Laboratory Parameters of Interest can be found in Section 12.12.1. Add footnotes: Note: Just parameters which can be classified in CTCAE grades are displayed. Note: Laboratory parameters of interest that have no results with a CTCAE grade were not included. | SAC |
| ECG | | | | | |
| 3.17. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| 3.18. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| 3.19. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC |
| Vital Si | gns | | | | |
| 3.20. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC |
| lmmun | ogenicity | | | | |
| 3.21. | Safety | Non Standard<br>SAFE_T8 | Summary of Immunogenicity Results | | SAC |
| Pulmor | nary Assessme | ents | | | |
| 3.22. | Safety | Non Standard<br>SAFE_T9 | Summary of Subjects with Pulmonary Findings | | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.23. | Safety | Non Standard<br>SAFE_T5 | Summary of Persistent Cough, Dyspnea and D <sub>LCO</sub> Decrease | | SAC |
| 3.24. | Safety | Non Standard<br>SAFE_T10 | Summary of Pulse Oximetry | | SAC |
| 3.25. | Safety | Non Standard<br>SAFE_T11 | Summary of Change from Baseline in Pulse Oximetry (%) | | SAC |
| 3.26. | Safety | Non Standard<br>SAFE_T11 | Summary of Change from Baseline in D <sub>LCO</sub> | Note: Baseline is defined as the lowest value during the screening period prior to the first study drug administration. | SAC |
| 3.27. | Safety | Non Standard<br>SAFE_T12 | Proportion of Subjects with a 15% Relative Decrease from Baseline in D <sub>LCO</sub> | | SAC |
| 3.28. | Safety | Non Standard<br>SAFE_T11 | Summary of Change from Baseline in Spirometry Data | Please add a parameter information above the table for the two separate parameters FEV1 and FVC | SAC |
| 3.29. | Safety | Non Standard<br>SAFE_T13 | Summary of Cough Data | | SAC |
| 3.30. | Safety | Non Standard<br>SAFE_T11 | Summary of Change from Baseline in Borg Dyspnea Score | | SAC |
| 3.31. | Safety | Non Standard<br>SAFE_T14 | Summary of Borg Dyspnea Questionnaire Data | | SAC |

# 12.15.8. Safety Figures

| Safety | Safety : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 3.1. | Safety | AE10 | Plot of Common (>=5%) Adverse Events and Relative Risks | Sorted by decreasing relative risk | SAC |
| Labora | tory Values | | | | |
| 3.2. | Safety | LB9 | Distribution of Laboratory Parameters of Interest by Visit and Treatment with Maximum over Time | Generate plots for the following parameters Hemoglobin, Total WBCs, Neutrophil Counts, Platelet Counts, ALT, AST and Total Bilirubin. | SAC |
| ECGs | | | | | |
| 3.3. | Safety | EG8 | Distribution of QTc Change by Time and Treatment | | SAC |
| Pulmor | Pulmonary Assessments | | | | |
| 3.4. | Safety | Non Standard<br>SAFE_F1 | D <sub>LCO</sub> Patient Profiles Over Time by Treatment | | SAC |

## 12.15.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 4.1. | PK | Non Standard<br>EFF_T1 | Summary of GSK3196165 serum concentrations by visit | | PK IA, Wk6<br>IA, SAC |
| 4.2. | PK | Non Standard | Summary of derived steady state exposure parameters | | PK IA, Wk6 IA |
| PK para | PK parameters | | | | |
| 4.3. | PK | Non Standard | Summary of derived PK parameters | | PK IA, Wk6 IA |

# 12.15.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK con | centration | | | | |
| 4.1. | PK | Non Standard | Plot of GSK3196165 concentration by visit | | PK IA, Wk6 IA |
| 4.2. | PK | Non Standard | Comparison of GSK3196165 concentration by visit in HOA and RA population | | PK IA, Wk6 IA |
| 4.3. | PK | Non Standard | Comparison of derived GSK3196165 steady state exposure in HOA, RA, healthy volunteers and multiple sclerosis population | | PK IA, Wk6 IA |
| PK para | PK parameters | | | | |
| 4.4. | PK | Non Standard | Plot of distribution of the derived PK parameters in HOA, RA, healthy volunteers and multiple sclerosis population | | PK IA, Wk6 IA |

# 12.15.11. Pharmacodynamic and / or Biomarker Tables

| Pharma | codynamic an | d/or Biomarker : | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Target | Engagement B | iomarkers | | | |
| 5.1. | Safety | Non Standard<br>PD_T1a or<br>PD_T1b | Summary of Observed Result and Change from Baseline in<br>Target Engagement Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |
| Predict | ive Biomarkers | 3 | | | |
| 5.2. | Safety | Non Standard<br>PD_T1a or<br>PD_T1b | Summary of Observed Result and Change from Baseline in Predictive Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |
| 5.3. | Safety | Non Standard<br>PD_T2a or<br>PD_T2b | Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Predictive Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |
| Cartilag | je Biomarkers | | | | |
| 5.4. | Safety | Non Standard<br>PD_T1a or<br>PD_T1b | Summary of Observed Result and Change from Baseline in Cartilage Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |
| Mechar | nistic Biomarke | ers | | · | |

| Pharma | acodynamic ar | d/or Biomarker : | Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.5. | Safety | Non Standard<br>PD_T1a or<br>PD_T1b | Summary of Observed Result and Change from Baseline in Mechanistic Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |
| Safety | Biomarkers | | | | |
| 5.6. | Safety | Non Standard<br>PD_T1a or<br>PD_T1b | Summary of Observed Result and Change from Baseline in Safety Biomarkers | Use appropriate table shell depending on whether or not log transformation has been performed. If there are both log transformed and not log transformed biomarkers, then display in two separate outputs. | SAC |

204851

# 12.15.12. Pharmacodynamic and / or Biomarker Figures

| Pharma | acodynamic an | d or Biomarker : | Figures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Target | Engagement B | iomarkers | | | |
| 5.1. | Safety | Non Standard<br>PD_F2 | Plot of Distribution of Target Engagement Biomarkers | | SAC |
| 5.2. | Safety | Non Standard<br>PD_F1 | Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Target Engagement Biomarkers, at Each Visit | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |
| Predict | ive Biomarkers | 5 | | | |
| 5.3. | Safety | Non Standard<br>PD_F2 | Plot of Distribution of Predictive Biomarkers | | SAC |
| 5.4. | Safety | Non Standard<br>PD_F1 | Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Predictive Biomarkers, at Each Visit | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |
| 5.5. | Safety | Non Standard<br>PD_F1 | Plot of Least Squares Means and 95% CI of Change from Baseline in Predictive Biomarkers (from Repeated Measures Analysis) | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |
| Cartila | ge Biomarkers | | | | |
| 5.6. | Safety | Non Standard<br>PD_F2 | Plot of Distribution of Cartilage Biomarkers | | SAC |

| Pharma | acodynamic an | d or Biomarker : | Figures | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.7. | Safety | Non Standard<br>PD_F1 | Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Cartilage Biomarkers, at Each Visit | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |
| Mechai | nistic Biomark | ers | | | |
| 5.8. | Safety | Non Standard<br>PD_F2 | Plot of Distribution of Mechanistic Biomarkers | | SAC |
| 5.9. | Safety | Non Standard<br>PD_F1 | Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Mechanistic Biomarkers, at Each Visit | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |
| Safety | Biomarkers | | | | |
| 5.10. | Safety | Non Standard<br>PD_F2 | Plot of Distribution of Safety Biomarkers | | SAC |
| 5.11. | Safety | Non Standard<br>PD_F1 | Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Safety Biomarkers, at Each Visit | X-Axis: Visit Y-axis: "Change from Baseline in <biomarker>" or "Ratio to Baseline in <biomarker>" if log-transformation is required</biomarker></biomarker> | SAC |

# 12.15.13. Pharmacokinetic / Pharmacodynamic Figures

| Pharmacokinetic / Pharmacodynamic : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1. | PK | Non Standard | Plot of change from baseline in 24h average hand pain intensity at week 4 versus pre-dose concentration at week 4 | | SAC |
| 6.2. | PK | Non Standard | Plot of change from baseline in 24h average hand pain intensity at week 6versus pre-dose concentration at week 6 | | SAC |

204851

# 12.15.14. ICH Listings

| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screening Failure | Journal guidelines | SAC |
| 2. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 4. | Enrolled | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | Enrolled | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoco | ol Deviations | | | | |
| 6. | Enrolled | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | Enrolled | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | l | | | |
| 8. | Enrolled | SA3 | Listing of Subjects Excluded from Any Population | ICH E3 | SAC |
| Demog | raphy | | | 1 | 1 |
| 9. | ITT | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | ITT | DM9 | Listing of Race | ICH E3 | SAC |
| Medica | l condition & c | oncomitant medi | cations | | |
| 11. | ITT | MH2 | Listing of Current/Past Medical Conditions | | SAC |
| 12. | ITT | CM3 | Listing of Prior and Concomitant Medications (Non-OA) | IDSL | SAC |
| 13. | ITT | CM3 | Listing of Prior and Concomitant OA Medications | | SAC |
| 16. | ITT | Non Standard POP_L1 | Listing of OA Disease History | | SAC |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposu | ıre | | | | |
| 17. | Safety | EX1 | Listing of Exposure to Study Treatment Data | ICH E3 | SAC |
| Advers | e Events | | | | |
| 18. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 19. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 20. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 21. | Safety | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | Wk6 IA, SAC |
| 22. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC |
| 23. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 24. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| 25. | Safety | AE7 | Listing of Subject Numbers for Adverse Events of Special Interest (AESIs) | ICH E3 | SAC |
| Labs | 1 | | | | • |
| 26. | Safety | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 27. | Safety | LB5 | Listing of Laboratory Values of Potential Clinical Importance | | SAC |
| 28. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 29. | Safety | UR2a | Listing of Urinalysis Data for Subjects with Abnormalities of Potential Clinical Importance | ICH E3 | SAC |
| Vital si | gns | | | <u></u> | 1 |

| ICH : Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 30. | Safety | VS4 | Listing of Vital Signs Data | | SAC |
| ECG | | | | | 1 |
| 31. | Safety | EG3 | Listing of ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 32. | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | IDSL | SAC |
| 33. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | IDSL | SAC |
| 34. | Safety | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC |
| Vital sig | gns | | | | |
| 35. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | IDSL Include Systolic BP, Diastolic BP, Pulse and Oxygen Saturation. | SAC |
| 36. | Safety | VS4 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| Immun | ogenicity | | | | |
| 37. | Safety | IMM2 | Listing of Immunogenicity Results | | SAC |
| Pulmor | nary Assessme | ents | | | |
| 38. | Safety | Non Standard POP_L2 | Listing of Subjects with Persistent Cough, Dyspnea or D <sub>LCO</sub> Decrease | | SAC |
| 39. | Safety | Non Standard<br>POP_L3 | Listing of Pulmonary Assessments | | SAC |
| 40. | Safety | Non Standard<br>POP_L4 | Listing of Pulmonary Function Tests | | SAC |

204851

# 12.15.15. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Efficac | y | | | | • |
| 41. | ITT | Non Standard<br>EFF_L1 | Listing of Individual Subject Hand Pain NRS Averaged over 7 Days Prior to Each Visit | | SAC |
| 42. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Average Hand Pain NRS Averaged over 7 Days Prior to Each Visit | | SAC |
| 43. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of GEE Analysis on Proportion of Subjects<br>Achieving 30% Reduction in Average Hand Pain NRS<br>Averaged over 7 Days Prior to Each Visit | | SAC |
| 44. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of GEE Analysis on Proportion of Subjects<br>Achieving 50% Reduction in Average Hand Pain NRS<br>Averaged over 7 Days Prior to Each Visit | | SAC |
| 45. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Worst Hand Pain NRS Averaged over 7 Days Prior to Each Visit, by Visit | | SAC |
| 46. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of GEE Analysis on Proportion of Subjects<br>Achieving 30% Reduction in Worst Hand Pain NRS Averaged<br>over 7 Days Prior to Each Visit | | SAC |
| 47. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of GEE Analysis on Proportion of Subjects<br>Achieving 50% Reduction in Worst Hand Pain NRS Averaged<br>over 7 Days Prior to Each Visit | | SAC |
| 48. | ITT | Non-Standard<br>EFF_L3 | Listing of Individual Subject AUSCAN 3.1 NRS Individual Component Scores | | SAC |
| 49. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in AUSCAN 3.1 NRS Individual Component Scores, by Visit | | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 50. | ITT | Non-Standard<br>EFF_L4 | Listing of Individual Subject Number of Soft Tissue Swollen or Tender Hand Joints, by Visit | | SAC |
| 51. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Number of Soft Tissue Swollen Hand Joints, by Visit | | SAC |
| 52. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Number of Tender Hand Joints, by Visit | | SAC |
| 53. | ITT | Non Standard<br>EFF_L5 | Listing of Individual Subject Pain/Tenderness Hand Joint Assessment, by Visit | | SAC |
| 54. | ITT | GA4 | Listing of Individual Subject Patient's and Physician's Global Assessments, by Visit | List both the Patients and Physicians<br>Global Assessments in the same<br>output with separate columns for each | SAC |
| 55. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Physician's Global Assessment, by Visit | | SAC |
| 56. | ITT | Non-Standard<br>EFF_L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Patient's Global Assessment, by Visit | | SAC |
| lmagin | g | | | | |
| 57. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Inflammatory Structural Joint Damage: HOAMRIS | Individual Components Include:<br>Synovitis, Erosive damage, Cyst,<br>Osteophyte Cartilage Space Loss,<br>Mal-alignment and Bone Marrow<br>Lesions | SAC |
| 58. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Inflammatory Structural Joint Damage: HOAMRIQ | Individual Components Include:<br>synovitis, normalised synovitis,<br>normalised erosive damage, cartilage<br>space loss, mal-alignment and<br>normalised bone marrow lesions | SAC |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 59. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Joint Inflammation: DCE-MRI | Includes ktrans, normalised Ktrans,<br>VE, normalised VE, VP, normalised<br>VP, IRE, normalised IRE, ME,<br>normalised ME. | SAC |
| 60. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Bone Shape Parameter | Includes Surface Area of Bone | SAC |
| PK | | | | | |
| 61. | PK | Non Standard<br>PK_L1 | Listing of Individual Subject Pharmacokinetic Data | | SAC |
| Biomai | rker | | | | |
| 62. | Safety | Non Standard<br>PD_L1 | Listing of Individual Subject Target Engagement | | SAC |
| 63. | Safety | Non Standard<br>PD_L1 | Listing of Individual Subject Predictive Biomarkers | | SAC |
| 64. | Safety | Non Standard<br>PD_L1 | Listing of Individual Subject Cartilage Biomarkers | | SAC |
| 65. | Safety | Non Standard<br>PD_L1 | Listing of Individual Subject Mechanistic Biomarkers | | SAC |
| 66. | Safety | Non Standard<br>PD_L1 | Listing of Individual Subject Safety Biomarkers | | SAC |
| 67. | Safety | Non Standard<br>EFF_ L2 | Statistical Listing of Repeated Measures Analysis of Change from Baseline in Predictive Biomarkers | | SAC |
| Additio | nal | | | | |

| Non-IC | Non-ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 68. | ITT | GA4 | Listing of Individual Subject Daily Hand Pain NRS Scores | List both the 24h Average and 24h Worst Hand Pain Score in the same output with separate columns for each. Only display absolute values | SAC |
| 69. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIS | Individual Components Include: Synovitis, Erosive damage, Cyst, Osteophyte Cartilage Space Loss, Mal-alignment and Bone Marrow Lesions | SAC |
| 70. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Change from Baseline in Inflammatory Structural Joint Damage: HOAMRIQ | Individual Components Include:<br>synovitis, normalised synovitis,<br>normalised erosive damage, cartilage<br>space loss, mal-alignment and<br>normalised bone marrow lesions | SAC |
| 71. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Change from Baseline in Joint Inflammation: DCE-MRI | Includes ktrans, normalised Ktrans,<br>VE, normalised VE, VP, normalised<br>VP, IRE, normalised IRE, ME,<br>normalised ME. | SAC |
| 72. | ITT | Non Standard<br>EFF_L6 | Listing of Individual Subject Change from Baseline in Bone Shape Parameter | Includes Surface Area of Bone | SAC |

## 12.16. Appendix 17: Example Mock Shells for Data Displays

Example: POP T1

Protocol: 204851 Confidential Population: Intent-to-Treat


Table 1.x Summary of Baseline Efficacy Parameters

| | | Placebo | GSK3196165 180mg | Total |
|---|---|---|---|---|
| | Statistic | N=XX | N=xx | N=xx |
| 24h average hand pain<br>NRS score averaged over<br>7 days prior to BL | n | xx | xx | xx |
| | Mean | XX.XX | XX.XX | XX.XX |
| | SD | xx.xxx | xx.xxx | xx.xxx |
| | Median | xx.xx | XX.XX | xx.xx |
| | Min | XX.X | XX.X | XX.X |
| | Max | XX.X | XX.X | XX.X |
| | n | XX | XX | XX |
| 24h worst hand pain NRS score averaged over 7 days prior to BL | n | xx | xx | xx |
| AUSCAN 3.1 NRS Total<br>Score | n | xx | xx | XX |
| AUSCAN 3.1 NRS Pain<br>Score | n | xx | xx | xx |
| AUSCAN 3.1 NRS Physical Function Score | n | XX | XX | XX |
| | ••• | | | <b></b> |

| | | Placebo | GSK3196165 180mg | Total |
|---|---|---|---|---|
| | Statistic | N=xx | N=xx | N=xx |
| AUSCAN 3.1 NRS<br>Stiffness Score | n | xx | xx | xx |
| | | | <del></del> | |
| Number of Soft Tissue<br>Swollen Hand Joints | n | xx | xx | xx |
| Number of Tender Hand<br>Joints | n | XX | xx | XX |
| | | ••• | | |
| PhGA | n | XX | xx | xx |
| PtGA | n | XX | xx | xx |
| CRP (mg/L) | n | XX | XX | xx |
| | | | ••• | ••• |

Note: PtGA= Patient's Global Assessment of Disease Activity, PhGA= Physician's Global Assessment of Disease Activity, CRP= C-Reactive Protein

Programming Note: Make sure to use the correct number of decimal places for each of the variables. Programming Note: show for all variables all descriptive statistics

204851

Example: POP T2


Population: Intent-to-Treat

Table 1.x Summary of OA Disease History

| | | Placebo | GSK3196165 180mg | Total |
|---|---|---|---|---|
| | Statistic | N=xx | N=xx | N=xx |
| Time since OA diagnosis (months) | n | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X |
| | SD | xx.xx | XX.XX | XX.XX |
| | Min | xxx | xxx | XXX |
| | Median | xxx | xxx | XXX |
| | Max | XXX | xxx | XXX |
| Time since start of OA symptoms (months) | n | xx | xx | XX |
| | Mean | XXX.X | XXX.X | XXX.X |
| | SD | XX.XX | xx.xx | XX.XX |
| | Min | XXX | xxx | XXX |
| | Median | XXX | xxx | XXX |
| | Max | XXX | xxx | xxx |

Note: Time since OA diagnosis and start of OA symptoms is calculated up to date of first study drug administration.

Example: POP T3


Population: Intent-to-Treat

| MedDRA vX.X<br>System Organ Class<br>Preferred Term | Placebo<br>N=xx<br>n (%) | GSK3196165 180mg<br>N=xx<br>n (%) | Total |
|---|---|---|---|
| Number of subjects with at least one medical history condition | xx (xx) | xx (xx) | xx (xx) |
| Cardiovascular Risk Factors | xx (xx) | xx (xx) | xx (xx) |
| Coronary Artery Disease | xx (xx) | xx (xx) | xx (xx) |
| Myocardial Infarction | xx (xx) | xx (xx) | xx (xx) |
| ••• | xx (xx) | xx (xx) | xx (xx) |
| System Organ Class 1 | xx (xx) | xx (xx) | xx (xx) |
| Preferred Term 1 | xx (xx) | xx (xx) | xx (xx) |
| Preferred Term 2 | xx (xx) | xx (xx) | xx (xx) |
| ••• | xx (xx) | xx (xx) | xx (xx) |

#### Notes to Programming Team:

• Cardiac Disorders to be taken from CRF.

204851

Example: EFF T1


Population: Intent-to-Treat

Table 2.x

Summary of Observed Result and Change from Baseline in [Parameter]

[Component: AUSCAN Pain/AUSCAN Physical Function/AUSCAN Stiffness/AUSCAN Total]

| | | Observed Results | | | Change from Baseline Results | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Visit | n | Mean<br>(95% CI) | SD | Median<br>(Min,Max) | n | BL<br>Mean | Mean<br>(95% CI) | SD | Median<br>(Min,Max) |
| GIOUP | ATSIC | | | | | | | | | |
| Placebo | Baselin | Х | x.xx | x.xxx | X.XX | | | | | |
| (N=XX) | е | Х | (x.xx, x.xx) | | (x.x, x.x) | | | | | |
| | Week 1 | Х | X.XX | X.XXX | X.XX | XX | x.xx | X • X | x.xx | X.X |
| | | Х | (x.xx, x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| | Week 2 | Х | X.XX | X.XXX | X.XX | XX | X.XX | X • X | X.XX | X • X |
| | | Х | (x.xx, x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| GSK319616 | Baselin | Х | X.XXX | x.xxx | X.XX | | | | | |
| 5 180mg<br>(N=XX) | е | Х | (x.xx, x.xx) | | (x.xx, x.xx) | | | | | |
| | Week 1 | Х | x.xxx | X.XXX | X.XX | XX | x.xx | x.x | x.xx | x.x |
| | | Х | (x.xx, x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| | | | | | | | | | | ••• |

Note: BL Mean for Week X is the mean of the Baseline values of all subjects with a non-missing value at Week X.

204851

Example: EFF T2


Population: Intent-to-Treat

Table 2.x

Mixed Model Repeated Measures Analysis (MMRM) of the Change from Baseline in [Parameter]

#### [Component: AUSCAN Pain/AUSCAN Physical Function/AUSCAN Stiffness/AUSCAN Total]

| | | | GSK3196165 |
|--------|-------------------------|---------|--------------|
| | | Placebo | 180mg |
| Visit | Statistic | N=xx | N=xx |
| E7 1 1 | | | |
| Week 1 | n | XX | XX |
| | LS Mean | X.XX | X.XX |
| | LS Mean Change | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% Confidence Interval | | (x.xx, x.xx) |
| | p-value | | 0.xxx |
| Week 2 | n | | |
| | LS Mean | X.XX | X.XX |
| | LS Mean Change | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% CI for Difference | | (x.xx, x.xx) |
| | | | (, |

Note: Repeated Measures Analysis adjusted for Baseline Value, Treatment Group, Visit and Treatment Group by Visit Interaction [and Baseline Value by Visit Interaction]

Note: n is the number of subjects with non-missing data at that visit.

204851

Example: EFF T3


Population: Intent-to-Treat

Table 2.x

Summary and Analysis of the Proportion of Subjects Achieving a [30/50]% or More Reduction in [Parameter] at Each Visit

| Visit | Statistic | Placebo<br>N=xx | GSK3196165 180mg<br>N=xx |
|--------|---------------|-----------------|--------------------------|
| Week 1 | n (%) | xx (xx) | xx (xx) |
| | Difference to | () | () |
| | Placebo (%) | | XX |
| | 95% CI (%) | | (xx.x, xx.x) |
| | Odds Ratio | | XX.X |
| | 95% CI (%) | | (xx.xx, xx.xx) |
| Week 2 | n (%) | xx (xx) | xx (xx) |
| | Difference to | . , | |
| | Placebo (%) | | XX |
| | 95% CI (%) | | (xx.x, xx.x) |
| | Odds Ratio | | XX.X |
| | 95% CI (%) | | (xx.xx, xx.xx) |

Note: Missing subjects have been assumed to be non-responders.

Note: Positive differences and Odds Ratios >1 indicate an improvement of treatment over placebo.

Note: 95% confidence intervals for the difference to placebo are constructed using asymptotic Wald confidence limits without correction.

Note: 95% confidence intervals for odds ratios are constructed using exact confidence limits.

Note: Generalised Estimating Equations Analysis adjusted for Baseline Score, Treatment Group, Visit and Treatment Group by Visit Interaction

204851

Example: EFF T4

Population: Intent-to-Treat

Table 2.x

Summary of Observed Result and Change from Baseline in [Inflammatory Structural Joint Damage/Joint Inflammation/Bone Shape Parameters]: [HOAMRIS/HOAMRIQ/DCE-MRI]

Parameter (Unit): <Synovitis/ Erosive Damage/ Cysts/ Osteophyte/ Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions> <Synovitis/ Synovitis (Normalised)/ Erosive Damage/ Erosive Damage (Normalised)/ Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions (Normalised)>

< Exchange rate, Interstitial volume, Plasma volume, Initial rate of enhancement, Maximal signal intensity enhancement>
<Surface Area of Bone>

| | | Observed Results | | | | Change from Baseline Results | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Visit | n | Mean<br>(95% CI) | SD | Median<br>(Min,Max) | n | BL Mean | Mean<br>(95% CI) | SD | Median<br>(Min,Max) |
| Placebo<br>(N=XX) | Baseline | xx | x.xx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.x, x.x) | | | | | |
| (=: ====, | Week 1 | XX | (x.xx, x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | XX | X.XX | x.x<br>(x.x,x.x) | X.XX | x.x<br>(x.x, x.x) |
| | Week 2 | XX | x.xx<br>(x.xx,x.xx) | X.XXX | x.xx<br>(x.xx, x.xx) | XX | X.XX | x.x<br>(x.x,x.x) | X.XX | (x.x, x.x) |
| | Week 4 | XX | x.xx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | XX | X.XX | x.x<br>(x.x,x.x) | x.xx | x.x<br>(x.x, x.x) |
| GSK3196165<br>180mg<br>(N=XX) | Baseline | xx | x.xxx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | | | | | |
| . , | Week 1 | XX | x.xxx<br>(x.xx,x.xx) | X.XXX | x.xx<br>(x.xx, x.xx) | XX | x.xx | x.x<br>(x.x,x.x) | x.xx | x.x<br>(x.x, x.x) |
| | | | <del></del> | | <del></del> | | | | | |

<Note: Synovitis is normalized by the total joint volume, erosive damage and bone marrow lesions are normalized by volume of bone.>

< Note: All parameters have been normalized by the Volume of Enhancing Pannus (VEP).>

Example: EFF T5


Population: Intent-to-Treat

#### Table 2.x

Repeated Measures Analysis of Observed Result and Change from Baseline in [Inflammatory Structural Joint Damage/Joint Inflammation]: [HOAMRIS/HOAMRIQ/DCE-MRI]

Parameter (Unit): <Synovitis/ Erosive Damage/ Cyst/ Osteophyte Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions> <Synovitis/ Synovitis (Normalised)/ Erosive Damage (Normalised)/ Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions (Normalised)>

< Exchange Rate, Interstitial Volume, Plasma Volume, Initial Rate of Enhancement, Maximal Signal Intensity Enhancement>

| | | | GSK3196165 |
|-----------|-------------------------|---------|-------------|
| | | Placebo | 180mg |
| Visit | Statistic | N=xx | N=xx |
| r.r 1 - 1 | | | |
| Week 1 | n | XX | XX |
| | LS Mean | X.XX | X.XX |
| | LS Mean Change | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% Confidence Interval | | x.xx - x.xx |
| | p-value | | 0.xxx |
| Week 2 | n | | |
| | LS Mean | X.XX | X.XX |
| | LS Mean Change | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% CI for Difference | | x.xx - x.xx |
| | p-value | | 0.xxx |

Note: Repeated measures analysis adjusted for <Parameter> baseline value, treatment group, visit, treatment group by visit interaction and baseline value by visit interaction.

Note: n is the number of subjects with non-missing data at that visit.

<Note: Synovitis is normalized by the total joint volume, erosive damage and bone marrow lesions are normalized by volume of bone.>

< Note: All parameters have been normalized by the Volume of Enhancing Pannus (VEP).>

204851

Example: EFF T6


Population: Intent-to-Treat

2.x Summary of the Proportion of Subjects Reporting Paracetamol Use in the 7 Days Prior to Each Visit

| Baseline n<br>No P | | | |
|--------------------|-------------------------|---------|---------|
| No P | | XX | xx |
| | aracetamol (%) | xx (xx) | xx (xx) |
| Para | cetamol for >=1 day (%) | xx (xx) | xx (xx) |
| Week 1 n | | xx | xx |
| No P | aracetamol (%) | xx (xx) | xx (xx) |
| Para | cetamol for >=1 day (%) | xx (xx) | xx (xx) |

•••
Example: EFF F1 Page 1 of x

Protocol: 204851 Confidential Population: Intent-to-Treat

Figure 2.x Individual Subject Profile Plots of [Parameter], by Treatment Group

Component: <AUSCAN Pain/AUSCAN Physical Function/AUSCAN Stiffness/ AUSCAN Total>



Note: Each of the lines represents one subject.

Note: B=Baseline


Population: Intent-to-Treat

Figure 2.x

Plot of Mean and 95% CI of Change from Baseline in [Parameter], at Each Visit

[Component/Parameter(Unit)]: <AUSCAN Pain/AUSCAN Physical Function/AUSCAN Stiffness/ AUSCAN Total>
<Synovitis/ Erosive Damage/ Cyst/ Osteophyte Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions>
<Synovitis/ Synovitis (Normalised)/ Erosive Damage (Normalised)/ Cartilage Space Loss/ Mal-alignment/ Bone Marrow Lesions
(Normalised)>

< Exchange Rate, Interstitial Volume, Plasma Volume, Initial Rate of Enhancement, Maximal Signal Intensity Enhancement>



Programming Note: Legend to be centered.

Example: SAFE T1


Population: Safety

Table 3.x
Overall Summary of Adverse Events

| Category | Placebo<br>N=xx<br>n (%) [#] | GSK3196165 180mg<br>N=xx<br>n (%) [#] |
|---|---|---|
| Any AEs | xx (xx) [x] | xx (xx) [x] |
| Serious AEs | xx (xx) [x] | xx (xx) [x] |
| AEs leading to permanent discontinuation of study treatment | xx (xx) [x] | xx (xx) [x] |
| Drug-related AEs | xx (xx) [x] | xx (xx) [x] |
| AEs leading to Death | xx (xx) [x] | xx (xx) [x] |

Note: n=number of subjects with at least one event. #=number of individual occurrences

Programming note: Include Withdrawals due to AE to "permanent discontinuation of study drug".

Example: SAFE T2


Population: Safety

| Category | Placebo (N=xx) n (%) [: | <b>#</b> ] | | GSK3<br>(N=x<br>n | 196165 180m<br>x)<br>(%) [#] | ng |
|---|---|---|---|---|---|---|
| | . , . | | | | | |
| Any AESI | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Serious Infections | xx | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Serious Respiratory Infections | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Opportunistic Infections | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Neutropenia | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Pulmonary Alveolar Proteinosis | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Hypersensitivity Reactions | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |
| Injection Site Reactions | XX | (xx%) | [xx] | XX | (xx%) [x | xx] |

AESI = Adverse Event of Special Interest.

Note: n=number of subjects reporting at least one event. [#] is the number of individual occurrences.

Example: SAFE T3


Population: Safety

 $\label{eq:Table 3.x} \textbf{Summary of Adverse Events of Special Interest - Injection Site Reactions}$ 

| | Placebo<br>N=xx | GSK3196165 180mg<br>N=xx |
|---|---|---|
| Number of Subjects with an | n (%) [#] | n (%) [#] |
| Injection Site Reaction | xx (xx) [xx] | xx (xx) [xx] |
| <= 1 Day Post Injection | xx (xx) [xx] | xx (xx) [xx] |
| > 1 Day Post Injection (\$) | xx (xx) [xx] | xx (xx) [xx] |
| Reported as AE | xx (xx) [xx] | xx (xx) [xx] |
| Reported as SAE | xx (xx) [xx] | xx (xx) [xx] |
| Itching/pruritis occurrence | xx (xx) [xx] | xx (xx) [xx] |
| Redness/erythema occurrence | xx (xx) [xx] | xx (xx) [xx] |
| Pain occurrence | xx (xx) [xx] | xx (xx) [xx] |
| Bruising occurrence | xx (xx) [xx] | xx (xx) [xx] |
| Swelling/edema | xx (xx) [xx] | xx (xx) [xx] |
| Warm to touch | xx (xx) [xx] | xx (xx) [xx] |

Note: n=number of subjects with at least one event. #=number of individual occurrences Note: (\$) until 1 day before next injection.

Example: SAFE T4


Population: Safety

Table 3.x Summary of Adverse Events of Special Interest - Systemic Hypersensitivity Reactions Related to GSK3196165

| | Placebo<br>N=xx | GSK3196165 180mg<br>N=xx |
|---|---|---|
| Type of Systemic Reaction | n (%) [#] | n=xx<br>n (%) [#] |
| Control - Nonconstitution Brooking | () | () [] |
| Systemic Hypersensitivity Reaction <= 1 Day Post Injection | xx (xx) [xx]<br>xx (xx) [xx] | xx (xx) [xx]<br>xx (xx) [xx] |
| > 1 Day Post Injection (\$) | xx (xx) [xx] | xx (xx) [xx] |
| Reported as an AE | xx (xx) [xx] | xx (xx) [xx] |
| Reported as an SAE | xx (xx) [xx] | xx (xx) [xx] |
| Headache | xx (xx) [xx] | xx (xx) [xx] |
| Pruritis | xx (xx) [xx] | xx (xx) [xx] |
| Urticaria | xx (xx) [xx] | xx (xx) [xx] |
| Rash | xx (xx) [xx] | xx (xx) [xx] |
| Angioedema | xx (xx) [xx] | xx (xx) [xx] |
| Met an Anaphylaxis Criterion | xx (xx) [xx] | xx (xx) [xx] |
| Anaphylactic Criterion 1 | xx (xx) [xx] | xx (xx) [xx] |
| Anaphylactic Criterion 2 | xx (xx) [xx] | xx (xx) [xx] |
| Anaphylactic Criterion 3 | | |

Note: n=number of subjects with at least one event. #=number of individual occurrences Note: (\$) until 1 day before next injection.

Example: SAFE T5


Population: Safety

 $\label{eq:table 3.x} \textbf{Summary of Persistent Cough, Dyspnea and } D_{\text{LCO}} \, \textbf{Decrease}$ 

| | Placebo | GSK3196165 180mg |
|---|---|---|
| | N=xx | N=xx |
| | n (%) | n (응) |
| Persistent Cough | xx (xx) | xx (xx) |
| Persistent Dyspnea | xx (xx) | xx (xx) |
| Persistent $D_{LCO}$ decrease >15% from baseline | xx (xx) | xx (xx) |

Note: n=number of subjects reporting at least one event in that category.

Note: Persistent is defined as any event with duration >=15 days. Cough must be grade 2 or 3. Dyspnea is determined from Borg scores >=3. Events were confirmed by the Safety Review Team.

Example: SAFE T6


Population: Safety

Table 3.x

Laboratory Evaluation: Summary of Proportion of Subjects with Urinalysis Findings

(Intent-to-Treat Population)

Laboratory Parameter: Protein

| | Placebo<br>N=xx | GSK3196165 180mg |
|----------|-----------------|------------------|
| | n (%) | N=xx<br>n (%) |
| Paraller | | |
| Baseline | | |
| n | XX | XX |
| 1+ | xx (xx) | xx (xx) |
| 2+ | xx (xx) | xx (xx) |
| 3+ | xx (xx) | xx (xx) |
| Negative | xx (xx) | xx (xx) |
| Trace | xx (xx) | xx (xx) |
| Week xx | | |
| n | XX | XX |
| 1+ | xx (xx) | xx (xx) |
| 2+ | xx (xx) | xx (xx) |
| 3+ | xx (xx) | xx (xx) |
| Negative | xx (xx) | xx (xx) |
| Trace | xx (xx) | xx (xx) |
| Week xx | | |
| | XX | XX |

Note: Percentages calculated based on the number of subjects with a valid assessment at the respective visit (n/M\*100%).

Programming Note: If multiple values are mapped to one visit: the value with the worst CTCAE grade will be considered. If there are more than one value of this grade, the later value will be considered.

Programming Note: Use this shell for all categorical parameters of Urinalysis, in case there are more than only Protein.

204851

Example: SAFE T7


Population: Safety

| Parameter | Visit | CTCAE Version 4.0 | Placebo<br>N=xx<br>n(%) | GSK3196165 180mg<br>N=xx<br>n(%) |
|---|---|---|---|---|
| Parameter 1 | Baseline | n | XX | XX |
| | | Grade 1 | xx(xx) | xx(xx) |
| | | Grade 2 | xx(xx) | xx(xx) |
| | | Grade 3 | xx(xx) | xx(xx) |
| | | Grade 4 | xx(xx) | xx(xx) |
| | Week x | n | xx | xx |
| | | Grade 1 | xx(xx) | xx(xx) |
| | | Grade 2 | xx(xx) | xx(xx) |
| | | Grade 3 | xx (xx) | xx (xx) |
| | | Grade 4 | xx (xx) | xx (xx) |
| Parameter 2 | | | | |

Note: Just parameters which can be classified in CTCAE grades are displayed.

Note: Laboratory parameters of interest that have no results with a CTCAE grade were not included.

Note: Percentages calculated based on the number of subjects with a valid assessment at the respective visit.

Programming Note: Laboratory Parameters of Interest and according CTCAE Grades can be found in the RAP Appendix 12. Programming Note: If multiple values are mapped to one visit: the value with the worst CTCAE grade will be considered. If there are more than one value of this grade, the later value will be considered.

Example: SAFE T8


Population: Safety

Table 3.x Summary of Immunogenicity Results

Assay: [Anti-GSK3196165 Binding AB Detection]

| | | Placebo | GSK3196165 180mg |
|-----------------------|----------|----------|------------------|
| | | N=xx | N=xx |
| Visit | | n (%) | n (%) |
| Baseline | n | xx | xx |
| | Positive | xx (xx%) | xx (xx%) |
| | Negative | xx (xx%) | xx (xx%) |
| Anytime Post-Baseline | n | xx | xx |
| _ | Positive | xx (xx%) | xx (xx%) |
| | - to + | xx (xx%) | xx (xx%) |
| | + to + | xx (xx%) | xx (xx%) |
| | Negative | xx (xx%) | xx (xx%) |
| | + to - | xx (xx%) | xx (xx%) |
| | - to - | xx (xx%) | xx (xx%) |
| Week 1 | n | xx | xx |
| | Positive | xx (xx%) | xx (xx%) |
| | Negative | xx (xx%) | xx (xx%) |
| Week X | n | xx | xx |

Note: Change refers to change from Baseline. Percentages for change are based on the number at risk at baseline, e.g. "- to +" and "- to -" are based on "Negative" at baseline.

Note: Percentages for Positive/Negative are based on the number of subjects at each visit.

Programming Note: Positive here refers to confirmed positive results, this should be evident from the dataset. Programming Note: "Anti-GSK3196165 Binding AB Detection" might have a slightly different naming convention in the dataset. Use the term from the dataset.

Programming Note: Include all relevant assessments.

Example: SAFE T9


Population: Safety

Table 3.x Summary of Subjects with Pulmonary Findings

| Subjects with at least one event of | Placebo<br>N=xx<br>n (%) | GSK3196165 180mg<br>N=xx<br>n (%) |
|---|---|---|
| 15% relative decrease from Baseline in $D_{\text{\tiny LCO}}$ | xx (xx) | xx (xx) |
| 15% relative decrease from Baseline in $D_{\text{LCO}}$ to $<\!70\%$ | xx (xx) | xx (xx) |
| Cough | xx (xx) | xx (xx) |
| Abnormal Lung Auscultation | xx (xx) | xx (xx) |

Note: Subjects with at least one event of 15% relative decrease from baseline in DLCO includes any subject with at least one decrease >15%. Cough includes subjects who reported cough of any grade. Abnormal lung auscultation includes subjects with any abnormality reported.

Example: SAFE\_T10

Population: Safety

Table 3.x Summary of Pulse Oximetry

| | Placebo | GSK3196165 180mg |
|----------------------------|---------|------------------|
| Visit | N=xx | N=xx |
| Blood Oxygen | n (%) | n (%) |
| Baseline | | |
| n | XX | xx |
| < 80% | xx (xx) | xx (xx) |
| 80% to 90% | xx (xx) | xx (xx) |
| >=90% | xx (xx) | xx (xx) |
| Worst Post-Baseline Result | | |
| n | XX | XX |
| < 80% | xx (xx) | xx (xx) |
| 80% to 90% | xx (xx) | xx (xx) |
| >=90% | xx (xx) | xx (xx) |

Note: Post-baseline percentages calculated based on the number of subjects in the relevant subgroup (n/M\*100%).

204851

Example: SAFE T11


Population: Safety

| | | | | Observe | d Result: | 3 | | | Cha | nge fro | om Basel | ine Resu | lts | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | Visit | n | Mean | SD | Median | Min | Max | n | BL Mean | Mean | SD | Median | Min | Max |
| Placebo (N=XX) | Baseline | XX | X.XX | x.xxx | X.XX | X.X | x.x | | | | | | | |
| | Week 1 | XX | X.XX | X.XXX | X.XX | X.X | X . X | XX | X.XX | X.XX | X.XXX | X.XX | X.X | х.х |
| | Week 2 | XX | X.XX | X.XXX | X.XX | X.X | X . X | XX | X.XX | X.XX | X.XXX | X.XX | X.X | х.х |
| | Week 3 | XX | X.XX | X.XXX | X.XX | X . X | X . X | XX | X.XX | X.XX | X.XXX | X.XX | X.X | X . X |
| | Week 4 | XX | X.XX | X.XXX | X.XX | X.X | X . X | XX | X.XX | X.XX | X.XXX | X.XX | $X \cdot X$ | X . X |
| | • • • | | | | | | | | | | | | | |
| GSK3196165 180mg<br>(N=XX) | Baseline | XX | x.xx | x.xxx | X.XX | X • X | x.x | | | | | | | |
| , | | XX | X.XX | x.xxx | X.XX | х.х | X . X | XX | | x.xx | x.xxx | X.XX | х.х | х.х |

Note: Baseline is defined as the lowest value during the screening period prior to the first study drug administration. Note: BL Mean for Week X is the mean of the Baseline values of all subjects with a non-missing value at Week X.

Programming note: First footnote only applies to DLCO outputs.

204851

Example: SAFE T12


Population: Safety

 $\mbox{Table 3.x} \\ \mbox{Summary of Proportion of Subjects with a 15% Relative Decrease from Baseline in $D_{LCO}$}$ 

| Visit | Placebo<br>N=xx | GSK3196165 180mg<br>N=xx |
|----------|-----------------|--------------------------|
| Decrease | n (%) | n (%) |
| Week 12 | | |
| n | XX | XX |
| ≥15% | xx (xx) | xx (xx) |
| <15% | xx (xx) | xx (xx) |
| Missing | xx (xx) | xx (xx) |

Note: Percentages calculated based on the number of subjects attending the respective visit. Notes to Programming Team:

• Compare Baseline value with value from Visit X. Count all subjects with a decrease of at least 15%.

Example: SAFE\_T13

Population: Safety

Table 3.x Summary of Cough Data

| Visit | Category | Placebo<br>N=xx<br>n(%) | GSK3196165 180mg<br>N=xx<br>n(%) |
|---|---|---|---|
| Baseline | n | XX | XX |
| | Had a Cough | xx (xx) | xx (xx) |
| | New | xx (xx) | xx (xx) |
| | Stable | xx (xx) | xx (xx) |
| | Worsening | xx (xx) | xx (xx) |
| | No Cough | xx (xx) | xx (xx) |
| | Missing | xx (xx) | xx (xx) |
| Week <1,, X> | n | xx | xx |
| | Had a Cough Since last Visit | xx (xx) | xx (xx) |
| | New | xx (xx) | xx (xx) |
| | Stable | xx (xx) | xx (xx) |
| | Worsening | xx (xx) | xx (xx) |
| | No Cough | xx (xx) | xx (xx) |
| | Missing | xx (xx) | xx (xx) |

Note: Percentages calculated based on the number of subjects attending the respective visit.

Example: SAFE T14


Population: Safety

Table 3.x Summary of Borg Dyspnea Questionnaire Data

| | Placebo<br>N=xx | GSK3196165 180mg<br>N=xx |
|---|---|---|
| visit Result | n (%) | n−xx<br>n (%) |
| 1010 | 11 (0) | 11 (0) |
| Baseline n | XX | xx |
| 0 Nothing at all | xx (xx) | xx (xx) |
| 0.3 | xx (xx) | xx (xx) |
| 0.5 Extremely weak | xx (xx) | xx (xx) |
| (Just noticeable) | | |
| 0.7 | xx (xx) | xx (xx) |
| 1 Very weak | xx (xx) | xx (xx) |
| 1.5 | xx (xx) | xx (xx) |
| 2 Weak (Light) | xx (xx) | xx (xx) |
| 2.5 | xx (xx) | xx (xx) |
| 3 Moderate | xx (xx) | xx (xx) |
| 4 | xx (xx) | xx (xx) |
| 5 Strong (Heavy) | xx (xx) | xx (xx) |
| | xx (xx) | xx (xx) |
| Missing | xx (xx) | xx (xx) |
| Week <1,, X> n | xx | xx |
| 0 Nothing at all | xx (xx) | xx (xx) |
| 0.3 | xx (xx) | xx (xx) |
| <pre>0.5 Extremely weak (Just noticeable)</pre> | xx (xx) | xx (xx) |

Note: Percentages calculated based on the number of subjects with a valid assessment at the respective visit.


Example: SAFE\_F1
Protocol: 204851 Confidential

Population: Safety

Figure 3.x D<sub>LCO</sub> Patient Profiles over Time by Treatment



Example: PD T1a


Population: Safety

Table 5.x

Summary of Observed Result and Change from Baseline in Target Engagement Biomarkers ##For Not Log Transformed Biomarkers##

Biomarker (Unit): <Name of Biomarker>

| | | | Obser | ved Result | S | | Cha | ange from Base | line Resul | ts |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | 771 - 1 - | n | Mean | SD | Median | n | BL Mean | Mean | SD | Median |
| Group | Visit | | (95% CI) | | (Min,Max) | | | (95% CI) | | (Min, Max) |
| Placebo | Baseline | XX | X.XX | x.xxx | x.xx | | | | | |
| (N=XX) | | | (x.xx,x.xx) | | (x.x, x.x) | | | | | |
| | Week 1 | XX | X.XX | X.XXX | X.XX | XX | X.XX | X • X | X.XX | X.X |
| | | | (x.xx,x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| | Week 2 | XX | X.XX | X.XXX | X.XX | XX | X.XX | X • X | X.XX | X . X |
| | | | (x.xx,x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| | Week 4 | XX | X.XX | X.XXX | X.XX | XX | X.XX | X • X | X.XX | X . X |
| | | | (x.xx,x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |
| | | ••• | | ••• | | | | | | |
| GSK3196165 | Baseline | XX | X.XXX | X.XXX | X.XX | | | | | |
| 180mg<br>(N=XX) | | | (x.xx,x.xx) | | (x.xx, x.xx) | | | | | |
| | Week 1 | XX | X.XXX | x.xxx | X.XX | XX | X.XX | X • X | X.XX | X.X |
| | | | (x.xx,x.xx) | | (x.xx, x.xx) | | | (x.x,x.x) | | (x.x, x.x) |

Note: The baseline value is the latest pre-dose assessment.

Note: BL Mean for Week X is the mean of the Baseline values of all subjects with a non-missing value at Week X.

Note: Values below LLQ are imputed to 0.5\*LLQ

Programming Note: The number of displayed decimal digits in the table can be different for each Biomarker.

Example: PD T1b


Population: Safety

Biomarker (Unit): <Name of Biomarker>

| | | | Observ | red Result | .S | | Ra | tio to Baseli: | ne Results | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | Geometric Mean<br>(95% CI) | CV <sub>b</sub> (%) | Median<br>(Min,Max) | n | BL<br>Geometric | Geometric<br>Mean Ratio | CV <sub>b</sub> (%) | Median<br>(Min,Max) |
| Treatment<br>Group | Visit | | | | | | Mean | (95% CI) | | |
| Placebo<br>(N=XX) | Baseline | XX | x.xx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.x, x.x) | | | | | |
| | Week 1 | XX | x.xx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | XX | X.XX | x.x<br>(x.x,x.x) | x.xx | x.x<br>(x.x, x.x) |
| | Week 2 | XX | x.xx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | XX | X.XX | x.x $(x.x,x.x)$ | x.xx | x.x<br>(x.x, x.x) |
| | Week 4 | XX | x.xx<br>(x.xx,x.xx) | X.XXX | x.xx<br>(x.xx, x.xx) | XX | X.XX | $x \cdot x$ $(x \cdot x, x \cdot x)$ | X.XX | x.x<br>(x.x, x.x) |
| | | | | ••• | | | <b></b> | | ••• | |
| GSK3196165<br>180mg<br>(N=XX) | Baseline | XX | x.xxx<br>(x.xx,x.xx) | x.xxx | x.xx<br>(x.xx, x.xx) | | | | | |
| | Week 1 | XX | x.xxx $(x.xx,x.xx)$ | x.xxx | x.xx<br>(x.xx, x.xx) | XX | x.xx | x.x $(x.x,x.x)$ | X.XX | x.x<br>(x.x, x.x) |

Note:  $CV_b$  = geometric coefficient of variation.

Note: The baseline value is the latest pre-dose assessment. BL Geometric Mean for Week X is the geometric mean of the

Baseline values of all subjects with a non-missing value at Week X.

Note: Values below LLQ are imputed to 0.5\*LLQ

Programming Note: The number of displayed decimal digits in the table can be different for each Biomarker.

Example: PD T2a


Population: Safety

Table 5.x

Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Target Engagement Biomarkers ## for not-log transformed biomarkers ##

Biomarker (Unit): <Biomarker>

| | | | GSK3196165 |
|--------|-------------------------|---------|-------------|
| | | Placebo | 180mg |
| Visit | Statistic | N=xx | N=xx |
| Week 1 | n | XX | XX |
| | LS Mean | X.XX | X.XX |
| | LS Mean Change | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% Confidence Interval | | x.xx - x.xx |
| | p-value | | 0.xxx |
| Week 2 | n | | |
| | LS Mean | x.xx | x.xx |
| | LS Mean Change | X.XX | x.xx |
| | Standard Error | X.XXX | X.XXX |
| | Difference from Placebo | | X.XX |
| | 95% CI for Difference | | x.xx - x.xx |

•••

Note: Repeated measures analysis adjusted for <Biomarker> baseline value, treatment group, visit, treatment group by visit and baseline by visit interactions.

Note: n is the number of subjects with non-missing data at that visit.

Example: PD T2b


Table 5.x

Mixed Model Repeated Measures Analysis (MMRM) of Change from Baseline in Target Engagement Biomarkers ## for log transformed biomarkers ##

Biomarker (Unit): <Biomarker>

| | | | GSK3196165 |
|--------|-------------------------------------|---------|-------------|
| | | Placebo | 180mg |
| Visit | Statistic | N=xx | N=xx |
| Week 1 | n | xx | xx |
| | LS Geometric Mean | X.XX | X • XX |
| | LS Geometric Mean Ratio to Baseline | X.XX | X.XX |
| | Standard Error | x.xxx | X.XXX |
| | Ratio to Placebo | | X.XX |
| | 95% Confidence Interval | | x.xx - x.xx |
| | p-value | | 0.xxx |
| Week 2 | n | | |
| | LS Geometric Mean | X.XX | X.XX |
| | LS Geometric Mean Ratio | X.XX | X.XX |
| | Standard Error | X.XXX | X.XXX |
| | Ratio to Placebo | | X.XX |
| | 95% Confidence Interval | | x.xx - x.xx |
| | p-value | | 0.xxx |

Note: Repeated measures analysis adjusted for <Biomarker> baseline value, treatment group, visit, treatment group by visit and baseline by visit interactions.

Note: n is the number of subjects with non-missing data at that visit.

Example: PD F1


Population: Intent-to-Treat

#### Figure 5.x

Plot of Mean/Geometric Mean and 95% CI of Change from Baseline in Target Engagement Biomarkers, at Each Visit

#### Biomarker(Unit): <Biomarker>



Note: Values below LLQ are imputed to 0.5\*LLQ.

Note: The baseline value is the latest pre-dose assessment.

<Note: Repeated measures analysis adjusted for <Biomarker> baseline value, treatment group, visit and treatment group by visit and baseline by visit interactions.>

Programming Note: Legend to be centered.

Programming Note: Y-axis label is "Change from Baseline in <Biomarker>" or "Ratio to Baseline in <Biomarker>" if log-

transformation is required

Example: PD F2


Population: Intent-to-Treat

Figure 5.x Plot of Distribution of <Biomarkers>

Biomarker(Unit): <Biomarker>

Treatment: <Overall/Placebo/GSK3196165 180mg>



Note: Values below LLQ are imputed to 0.5\*LLQ.

Note: The baseline value is the latest pre-dose assessment.

204851

Example: POP\_L1

Population: Intent-to-Treat

Listing x

Listing of OA Disease History

Treatment Group: <Placebo, GSK3196165 180mg>

| Site ID/<br>Subject ID | Date of OA Diagnosis | Time since OA Diagnosis (months) [a] | Start Date of OA<br>Symptoms | Time since Start of OA<br>Symptoms (months) [a] |
|---|---|---|---|---|
| XX/XXXXX | DD-MMM-YYYY | XX.X | DD-MMM-YYYY | XX.X |
| XX/XXXXX | | | | |
| XX/XXXXX | | | | |

[a] Up to date of first study medication administration.

204851

Example: POP L2


Population: Intent-to-Treat

Listing x

Subjects with Persistent Cough, Dyspnea or D<sub>LCO</sub> Decrease

| Site ID/ Subject ID | <pre>Gender/Age(years)/Race/Weight(kg):</pre> | Treatment<br>at Event<br>Onset | Type of<br>Event | Start of Event (Relative Day) |
|---|---|---|---|---|
| XXXX/XXXXXX | F/XX/XXXX/XX | Placebo | DLCO<br>Cough | DD-MMM-YYYY (XX) |

Programming Note: Just show subjects who experienced at least one of the events during the study.

204851

Example: POP L3


Population: Intent-to-Treat

Listing x

Listing of Pulmonary Assessments

Treatment Group: <Placebo, GSK3196165 180mg>

Site ID/ Subject ID: XXXX/XXXXXX Gender/Age(years)/Race/Weight(kg): F/XX/XXXX/XX

| Visit | Date of<br>Assessment<br>DD-MMM-YYYY<br>(Relative Day) | Chest X-Ray | Blood<br>Oxygen<br>(%) | Cough/<br>Grade | Borg<br>Dyspnea<br>Result | Chest Auscultation<br>abnormal/<br>Classification of<br>Chest Auscultation<br>abnormal |
|---|---|---|---|---|---|---|
| Screening | DD-MMM-YYYY (XX) | <pre><normal, -="" abnormal="" clinically="" not="" significant="" significant,=""></normal,></pre> | XX | Yes/ x | XXXX | Yes/ Stable |
| Baseline | DD-MMM-YYYY (XX) | | XX | No | XXXX | No |
| Week 1 | | | | | | |
| Etc. | | | | | | |
| 200. | | | | | | |

Example: POP L4


Population: Intent-to-Treat

Listing x

Listing of Pulmonary Function Tests

Treatment Group: <Placebo, GSK3196165 180 mg>

Site ID/ Subject ID: XXXX/XXXXXX Gender/Age(years)/Race/Weight(kg): F/XX/XXXX/XX

| | Date of<br>Assessment | Spirom | etry | _ | Gas | | |
|---|---|---|---|---|---|---|---|
| Visit | DD-MMM-YYYY<br>(Relative Day) | FEV1<br>(L) | FVC<br>(L) | Reason of Missed<br>Spirometry | Transfer (D <sub>LCO</sub> ) (%) | Reason of Missed $D_{\text{LCO}}$ | $D_{	ext{LCO}}$ Lower than 85% of Baseline Value |
| Screening | DD-MMM-YYYY<br>(XX) | xx.x | XX.X | XXXXXXX | xx.x | XXXXXXX | Yes |
| Baseline | DD-MMM-YYYY<br>(XX) | XX.X | XX.X | XXXXXXX | XX.X | XXXXXXX | No |

Week 1 Etc.

Note: Baseline is the visit recording the lowest DLCO value obtained from the Screening or Day 1 assessment, or any unscheduled visit in between.

Protocol: 204851 Confidential Page 1 of x Population: Intent-to-Treat

#### Treatment Group: <Placebo, GSK3196165 180mg>

| | | 24h Average Hand<br>Days | d Pain NRS Avera<br>Prior to Visit | aged over 7 | | Pain NRS Averaged<br>Prior to Visit | d over 7 Days |
|---|---|---|---|---|---|---|---|
| Site ID/<br>Subject ID | Visit | Observed/CfB | 30%<br>Reduction<br>from<br>Baseline | 50%<br>Reduction<br>from<br>Baseline | Observed/ CfB | 30%<br>Reduction<br>from<br>Baseline | 50%<br>Reduction<br>from<br>Baseline |
| XXXX/ XXXXX | Baseline | X.XX | | | X.XX | | |
| | Week X | x.xx/-x.xx | Yes | No | x.xx/ x.xx | No | No |
| | Etc. | Etc. | | | Etc. | | |
| XXXX/ XXXXX | Baseline | x.xx | | | x.xx | | |
| | Week X | x.xx/ x.xx | No | No | x.xx/ -x.xx | Yes | Yes |
| | Etc. | Etc. | | | Etc. | | |

Note: CfB= Change from Baseline.

Notes to Programming Team:

• This listing will be sorted by Site ID, Subject ID, Visit Date

204851


Example: EFF\_L2
Protocol: 204851 Confidential

Population: Intent-to-Treat

Listing x

Statistical Listing of [...]

Display all SAS Output from Analysis


Population: Intent-to-Treat

Listing x

Listing of Individual Subject AUSCAN 3.1 NRS Individual Component Scores

Treatment Group: <Placebo, GSK3196165 180mg>

| Site ID/ | | Pain Subscale | Physical Function | Stiffness Subscale | Total Score |
|---|---|---|---|---|---|
| Subject ID | Visit | Score | Subscale Score | Score | |
| XXXX/ XXXX | Baseline | Xx | Xx | Xx | Xxx |
| | Week X | Xx | Xx | Xx | Xxx |
| | Etc. | | | | |
| XXXX/ XXXX | Baseline | Xx | Xx | Xx | Xxx |
| | Week X | Xx | Xx | Xx | Xxx |
| | Etc. | | ••• | | |

Notes to Programming Team:

• This listing will be sorted by Site ID, Subject ID, Visit Date


Population: Intent-to-Treat

Listing x

Listing of Individual Subject Number of Tender or Swollen Hand Joints, by Visit

Treatment Group: <Placebo, GSK3196165 180mg>

Site ID/Subject ID: XXXXX/ XXXXXXX

| Visit | | Right Hand Joints | Left Hand Joints | Total Number of Joints |
|---|---|---|---|---|
| Baseline | Tender | PIP 2, PIP3, PIP4,<br>MCP1 | PIP2, PIP3 | 6 |
| | Swollen | PIP2, PIP4 | | 2 |
| Week 1 | Tender | PIP 2, PIP3, PIP4,<br>MCP1 | PIP2, PIP3 | 6 |
| | Swollen | PIP2, PIP4 | | 2 |

Notes to Programming Team:

<sup>•</sup> This listing will be sorted by Site ID, Subject ID, Visit Date


Population: Intent-to-Treat

Listing x

Listing of Individual Subject Pain/Tenderness Hand Joint Assessment, by Visit

Treatment Group: <Placebo, GSK3196165 180mg>

Site ID/Subject ID: XXXXX/ XXXXXXX

| Visit | Pain/Tenderness | Right Hand Joints | Left Hand Joints | Total Number of Joints |
|---|---|---|---|---|
| | Severity | | | |
| Baseline | Mild | PIP 2, PIP3, PIP4,<br>MCP1 | PIP2, PIP3 | 6 |
| | Moderate | PIP2, PIP4 | | 2 |
| | Severe | PIP5 | | 1 |
| \ 4 | | | P-P0 P-P0 | |
| Week 1 | Mild | PIP 2, PIP3, PIP4,<br>MCP1 | PIP2, PIP3 | 6 |
| | Moderate | PIP2, PIP4 | | 2 |
| | Severe | PIP5 | | 1 |

Notes to Programming Team:

<sup>•</sup> This listing will be sorted by Site ID, Subject ID, Visit


Population: Intent-to-Treat

Listing x

Listing of Individual Subject Inflammatory Structural Joint Damage: HOAMRIS

Treatment Group: <Placebo, GSK3196165 180mg>

| Site ID/<br>Subject ID | Visit | Number of<br>Available<br>Joints | Synovitis | Erosive<br>Damage | Cyst | Osteophyte | Cartilage<br>Space Loss | Mal-<br>alignment | Bone<br>Marrow<br>Lesions |
|---|---|---|---|---|---|---|---|---|---|
| XXXX/ XXXXX | Baseline | Xx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |
| | Week X | Xx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |
| | ••• | | | | | | | | |
| XXXX/ XXXXX | Baseline | Xx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |
| | Week X | Xx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |

Notes to Programming Team:

• This listing will be sorted by Site ID, Subject ID, Visit

204851

Example: PK\_L1


Population: Intent-to-Treat

Listing x

Listing of Individual Subject Pharmacokinetic Data

Treatment Group: <Placebo, GSK3196165 180mg>

Site ID/ Subject ID: XXXX/XXXXXX Gender/Age(years)/Race/Weight(kg): F/XX/XXXX/XX

| Visit | Date and Time Sample<br>Taken (Relative Day) | Dose Volume administered (mL) | PLASMA GSK3196165 ng/mL | Reason Test not Done |
|---|---|---|---|---|
| Screening | DDMMMYYY/ HH:MM (XX) | x.x | XXX | |
| Baseline | DDMMMYYY/ HH:MM (XX) | x.x | ΑΛΑ | XXXXX |
| Week X | | x.x | xxx | |

Example: PD L1


Population: Intent-to-Treat

Listing x

Listing of Individual Subject <Target Engagement/Predictive/...> Biomarkers

Treatment Group: <Placebo, GSK3196165 180mg >

Site ID/ Subject ID: XXXX/XXXXXX Gender/Age(years)/Race/Weight(kg): F/XX/XXXX/XX

| Biomarker (Unit) | Visit | Date and Time Sample Taken (Relative Day) | Result | Change from<br>Baseline | Ratio from<br>Baseline (%) |
|---|---|---|---|---|---|
| XXXXX (XX) | Screening<br>Baseline<br>Week X<br>Etc. | DD-MMM-YYYY / HH:MM (xx) DD-MMM-YYYY / HH:MM (xx) | xx.x<br>xx.x | xx.x<br>xx.x | xx.x<br>xx.x |
| XXXXX (XX) | Baseline<br>Week X<br>Etc. | DD-MMM-YYYY / HH:MM (xx) | xx.x | xx.x | xx.x |

Note: Values below LLQ are imputed to 0.5\*LLQ.